



# An Open-Label, Randomized, Non-Comparative Phase 2 Study of ARV-471 or Anastrozole in Post-Menopausal Women With ER+/HER2- Breast Cancer in the Neoadjuvant Setting

**Statistical Analysis Plan** 

Version: Draft 3.0

Date: 15 November 2024



Version: Final 3.0
Date: 15Nov2024
Statistical Analysis Plan

# SIGNATURE PAGE





Date: 15Nov2024
Statistical Analysis Plan

# **Table of Contents**

| SIGN | ATURE PAGE | 2 |
|-------|--------------------------------------------|----|
| | of Contents | |
| | REVIATIONS | |
| | ntroduction | |
| | tudy Design. | |
| 2.1 | Study Objectives, Endpoints, and Estimands | |
| 2.1.1 | Study Objectives and Endpoints | |
| 2.1.2 | Estimands | |
| 2.2 | Sample Size Considerations. | |
| | nalysis Sets | |
| | eneral Considerations | |
| 4.1 | Programming Environment | |
| 4.2 | General Statistical Methods | |
| 4.2.1 | Analysis Groups | |
| 4.2.2 | Descriptive Summaries | |
| 4.2.3 | Presentation Conventions | |
| 4.3 | Covariates and Strata | |
| 4.4 | Subgroups | 15 |
| 4.5 | Multiple Comparison/Multiplicity | |
| 5 D | Definitions & Data Handling Conventions | |
| 5.1 | Study Day, Duration, and Study Periods | |
| 5.1.1 | Study Day | |
| 5.1.2 | Duration | 16 |
| 5.2 | Analysis Visit Windows | 16 |
| 5.3 | Baseline and Change from Baseline | 16 |
| 5.4 | Missing Data | |
| 5.4.1 | Partial or Missing Dates and Time | 16 |
| 5.4.2 | Other Missing Values | |
| | TUDY POPULATION AND DISPOSITION | |
| 6.1 | Analysis Sets | |
| 6.2 | Participant Disposition | |



Date: 15Nov2024
Statistical Analysis Plan

| 6.3 | Protocol Deviations | 17 |
|---|---|---|
| 7 | Demographics And Disease Characteristics | 18 |
| 7.1 | Demographics and Baseline Characteristics | 18 |
| 7.2 | Disease Staging and Disease Characteristics | 18 |
| 7.3 | Disease Staging at Post-Surgery | 19 |
| 7.4 | Molecular Biology of Disease at Baseline | 20 |
| 7.5 | Prior Cancer Related Surgery/Biopsy | 20 |
| 7.6 | Medical History | 21 |
| 8 | Protocol-Required Drug Exposure And Compliance | 21 |
| 9 | Prior and Concomitant Therapies | 22 |
| 9.1 | Prior and Concomitant Medications | 22 |
| 10 | Efficacy Analyses | 22 |
| 10.1 | Assessment | 22 |
| 10.1 | .1 Tumor Biopsies | 22 |
| 10.1 | .2 Radiographic Imaging | 22 |
| 10.1 | .3 Physical Exam | 22 |
| 10.1 | .4 Local Pathological Assessments | 23 |
| 10.2 | Definitions of Efficacy Endpoints | 23 |
| 10.2 | 2.1 Ki-67 Percentage at C1D15 (Primary) | 23 |
| 10.2 | ER Percentage at C1D15 | 23 |
| 10.2 | 2.3 pCR Rate | 23 |
| 10.2 | mPEPI Score and mPEPI0 Rate | 23 |
| 10.2 | 2.5 Breast Conserving Surgery (BCS) Rate | 24 |
| 10.2 | 2.6 Radiographic Response per mRECIST in Primary Tumor during Cycle 6 | 24 |
| 10.2 | 2.7 Caliper-Based Response | 24 |
| 10.2 | 2.8 CCCA Rate | 24 |
| 10.3 | Analysis of Efficacy Variables | 24 |
| 10.3 | Ki-67 Percentage at C1D15 (Primary) | 24 |
| 10.3 | 3.2 Binary or Categorical Endpoints | 25 |
| 10.3 | Primary Tumor Assessments | 25 |
| 10.3 | ER AQUA Score Percentage at C1D15 and Surgery | 25 |
| 10.3 | PR H-score Percentage at C1D15 and Surgery | 26 |



Date: 15Nov2024
Statistical Analysis Plan

| 10.3.6 | Subgroup Analyses | 26 |
|--------|--------------------------------------------------------------|----|
| 11 Sa | ıfety Analyses | 26 |
| 11.1 | Adverse Events | 27 |
| 11.2 | Deaths | 28 |
| 11.3 | Vital Signs | 28 |
| 11.4 | Clinical Laboratory | 28 |
| 11.5 | 12-Lead Electrocardiogram | 29 |
| 11.6 | Eastern Cooperative Oncology Group (ECOG) Performance Status | 29 |
| | ther Analyses | |
| 12.1 | Pharmacokinetics | 29 |
| | Pharmacodynamics | |
| | hedule of Analyses | |
| 14 Re | eferences | 30 |



Date: 15Nov2024
Statistical Analysis Plan

# MODIFICATION HISTORY

| DRAFT VERSION HISTORY | | |
|---|---|---|
| Draft 0.1 | 09Jan2023 | The first draft based on Original Protocol dated on 27 May 2022 |
| Draft 0.1 | 27Jan2023 | Update based on Amendment #1 dated on 09 Jan 2023 and comments from internal reviewer |
| Draft 0.2 | 10Mar2023 | Update based on Arvinas comments |
| Draft 0.3 | 17Apr2023 | * Accept Arvinas updates and Caidya updates in draft 0.2 |
| | | * Remove the summary for BOR and ORR, add summary for radiographic response per mRECIST in primary tumor during Cycle 6 |
| | | * Update based on Arvinas comments on TFL shells |
| Draft 0.4 | 24Apr2023 | Correct Typo |
| Final 1.0 | 25Apr2023 | N/A |
| Draft 1.1 | 16Jan2024 | Update based on Arvinas comments on dryrun TFLs |
| Draft 1.2 | 24May2024 | Update based on Arvinas comments and new requests |
| Final 2.0 | 03June2024 | Accept the updates in version 1.2 and make minor updates based on Arvinas comments |
| Draft 2.1 | 06Sep2024 | Update CI round rules and baseline definition |
| | | Add Estimands in the document |
| Draft 2.2 | 11Oct2024 | Update based on the comments on dryrun #2 draft: |
| | | * Update the definition of subgroups — derivation will be from primary target lesion(s) and laboratory data instead of IRT |
| | | * Add summary for participants with Tumor<br>Biopsies at each visit, medical history,<br>absolute dose intensity, relative dose intensity,<br>subgroup analysis for change of tumor size by<br>baseline tumor size category |



Date: 15Nov2024
Statistical Analysis Plan

| | | | * Add additional plots for KI-67 at surgery,<br>ER AQUA Score, PR H-score |
|---|---|---|---|
| | | | * Update Concomitant Medications and<br>TEAE definition |
| Draft 2.3 | 14Nov2024 | Accept the updates in version 2.2 and the edite by Arvinas in version 2.2 | |
| | | | Update based on the comments on dryrun #2 final: |
| | | | * update 'MedDRA 24.0' to 'MedDRA 27.0 or higher' |
| | | | * Tornado plot for treatment emergent adverse<br>events with Grade 3 or higher by Preferred<br>Term |
| | | | * Add imputation for PR H-score post-baseline value of 0 for the derivation of log transform analysis |
| Final 3.0 | 15Nov2024 | | Accept update in 2.3 |



Date: 15Nov2024
Statistical Analysis Plan

# **ABBREVIATIONS**

| | 1 |
|----------|-------------------------------------------------------|
| AE | adverse event |
| ALT | alanine aminotransferase |
| Alk Phos | alkaline phosphatase |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BCS | breast conserving surgery |
| BID | twice daily |
| BP | blood pressure |
| CBR | clinical benefit response |
| CCCA | complete cycle cell arrest |
| CI | confidence interval |
| Cmax | maximum observed concentration |
| Cmin | minimum observed concentration |
| CRF | case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| Ctrough | trough concentration |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EDC | electronic data capture |
| ER | estrogen receptor |
| HER2 | human epidermal growth factor receptor 2 |
| IHC | immunohistochemistry |
| ISH | in situ hybridization |
| LSM | least square means |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mPEPI | modified Pre-Operative Endocrine Prognostic Index |
| MRI | magnetic resonance imaging |
| NA | not applicable |
| NCI | National Cancer Institute |
| NET | neoadjuvant endocrine therapy |
| ORR | objective response rate |
| pCR | pathologic complete response |
| PD | pharmacodynamics(s) |
| PK | pharmacokinetic(s) |
| PR | partial response |
| PT | preferred term |
| QTc | corrected QT |
| QTcF | corrected QT (Fridericia method) |
| mRECIST | modified Response Evaluation Criteria in Solid Tumors |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | Stable Disease |
| SOC | standard of care |
| _~~~ | 5.001.001.001.001.001.001.001.001.001.00 |



Date: 15Nov2024
Statistical Analysis Plan

| t1/2 | terminal elimination half-life |
|-------|----------------------------------|
| Tbili | total bilirubin |
| TEAE | treatment-emergent adverse event |
| Tmax | time to maximum concentration |
| TRAE | treatment-related adverse event |
| ULN | upper limit of normal |



 Date: 15Nov2024
Statistical Analysis Plan

#### 1 INTRODUCTION

The objective of this document is to detail the statistical methodology to be used in the summary and the final statistical analysis of clinical study protocol ARV-471-BC-201: "An Open-Label, Randomized, Non-Comparative Phase 2 Study of ARV-471 or Anastrozole in Post-Menopausal Women With ER+/HER2- Breast Cancer in the Neoadjuvant Setting".

This SAP is based on Protocol dated on 09 Jan 2023 and Case Report Forms (CRFs) dated on 23 Aug 2023.

#### 2 STUDY DESIGN

This is a Phase 2, open-label, randomized, non-comparative, proof of concept study of ARV-471 or anastrozole in participants with ER+/HER2- breast cancer amenable to definitive surgical resection. The main goal of this study is to evaluate the biological activity of ARV-471 and anastrozole, respectively.

Participants will be randomized in a 2:1 manner to receive treatment on one of two treatment arms for approximately 5.5 months:

- Arm A: ARV-471 200 mg orally, daily and continuously until day before surgical resection (no later than C6D18 + 14 days)
- Arm B: anastrozole 1 mg orally, daily and continuously until day before surgical resection (no later than C6D18 + 14 days)

Stratification will occur based on the following features of the participant's breast cancer:

- Size of primary breast tumor (T-stage):  $\leq 2$  cm,  $\geq 2$  to  $\leq 5$  cm, or  $\geq 5$  cm.
- Ki-67 score (assessed locally): < 20% or  $\ge 20\%$

Participants will have a screening biopsy, an on-treatment biopsy on C1D15 ( $\pm$  5 days), and surgical resection approximately 5.5 months after starting treatment (C6D18  $\pm$  14 days). Participants will return for follow up 30 days ( $\pm$  7 days) after definitive surgical resection. After surgery, participants will receive SOC radiation and systemic therapy (chemotherapy, endocrine therapy, etc.) in accordance with local practice guidelines per the treating physician's discretion. No participant should take study drug dispensed for the trial after surgical resection, and no study drug should be dispensed after surgical resection.

#### 2.1 Study Objectives, Endpoints, and Estimands

#### 2.1.1 Study Objectives and Endpoints

| Objective | Endpoints |
|---|---|
| Primary | |
| Evaluate the effects of ARV-471 and anastrozole, respectively, on Ki-67 expression in tumors after 2 weeks of treatment | Percent change in Ki-67 expression between baseline and C1D15 tumor biopsies |
| Secondary | |



 Date: 15Nov2024
Statistical Analysis Plan

| Evaluate the safety and tolerability of ARV-471 and anastrozole, respectively | Incidence of all adverse events, serious adverse events, and adverse events leading to study drug discontinuation |
|---|---|
| Evaluate the clinical and pathological response of ARV-471 and anastrozole, respectively | Pathologic stage, pathologic complete response (pCR)rate, and modified Preoperative Endocrine Prognostic Index (mPEPI) score at the time of surgical resection (C6D18 ± 14 days); rates of breast conserving surgery (BCS); radiographic response of the primary tumor based on breast imaging during cycle 6; caliper-based response on C6D1 |
| Exploratory | |
| Evaluate the effects of ARV-471 and anastrozole, respectively, on CCCA after 2 weeks of treatment | CCCA (Ki67 ≤2.7%) rates at C1D15 |
| Evaluate ER degradation of ARV-471 | Percent change in estrogen receptor (ER) protein levels between baseline and C1D15 |
| Evaluate the effects of ARV-471 and anastrozole, respectively, on Ki-67, and ER degradation by ARV-471 in tumors at the time of surgical resection. Explore additional biomarkers that may be | Changes in ER and Ki-67 expression between baseline and Cycle 6 surgical tumor samples; Rates of CCCA in the Cycle 6 surgical samples. Additional biomarkers may include, but are |
| associated with the effects of ARV-471 in tumor tissue | not limited to, PgR expression, |
| Correlate exposure of ARV-471 with ER reduction | Correlate population PK model-derived PK parameters (AUC, Cmin, Cmax) with ER reduction or other response parameters |

#### 2.1.2 Estimands

# 2.1.2.1 Primary Estimands

The primary estimand of this study is defined as the percent change in Ki-67 expression between baseline and C1D15 tumor biopsies observed from each Arm, respectively. Descriptive statistics will be provided to evaluate the effects of ARV-471 and anastrozole, respectively, on Ki-67 expression in tumors after two weeks of treatment. No comparisons between the treatment arms are planned.

Treatments: ARV-471 (Arm A) and anastrozole (Arm B)

Population: post-menopausal women with newly diagnosed and treatment naïve ER+/HER2-breast cancer that is amenable to definitive surgical resection. Participants must also have tumor that is at least 1.5 cm by imaging due to biopsy requirements for this study. The primary analysis regarding Ki-67 expression will be performed in all enrolled participants who received at least one dose of study treatment and had evaluable Ki-67 measurements from baseline and C1D15 visits.



Date: 15Nov2024
Statistical Analysis Plan

Variable: the log-transformed Ki-67 after approximately two weeks of treatment as a percentage of the baseline value, ie, the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline.

Intercurrent events: only participants with evaluable Ki-67 results from baseline and C1D15 visits will be included in the primary analysis. No participants will be censored or excluded due to any reasons other than missing Ki-67 data.

Population-level summary: the log-transformed percentage Ki-67 will be modelled using a GLM. Refer to Protocol Section 9.3.2 and the SAP for more details.

#### 2.1.2.2 Secondary Estimands

There are no key secondary endpoints defined for this study. No estimands are defined for any of the secondary or exploratory endpoints.

# 2.2 Sample Size Considerations

There are no plans for formal comparisons between ARV-471 and anastrozole. No power calculations are needed. Approximately 150 participants will be randomized to the two treatment arms in 2:1 ratio (100 participants to the ARV-471 arm and 50 participants to the anastrozole arm). These numbers were chosen to provide meaningful information about the primary endpoint, ie, changes (on-treatment C1D15 vs baseline) in Ki-67 expression levels after approximately 2 weeks of treatment with ARV-471 and anastrozole, respectively.

Table 1 and Table 2 provide a list of probable scenarios demonstrating the width of the CIs for the primary endpoint under the assumption that 80% (ie, n=120) of the randomized participants will provide valid Ki-67 measurements from both their baseline and C1D15 visits. Table 2 indicates that the width of the 80% CIs of the mean percentage Ki-67 after 2 weeks of treatment by ARV-471 will not exceed 14% and the width of the 95% CIs will not exceed 21.6% if the mean percentage of the corresponding baseline values after 2 weeks of treatment ranges from approximately 20% to 40%. The planned sample size will provide estimates for the treatment effect in terms of the reduction of Ki-67 with reasonable precision.

Table 1 Confidence Intervals for Mean Percentage of Baseline Value in Ki-67 After Two Weeks

| Number of participants/arm <sup>a</sup> | Mean<br>percentage<br>Ki-67 in<br>two weeks <sup>b</sup> | SD of log-<br>transformed<br>percent<br>change in Ki-<br>67 <sup>c</sup> | 80% CI <sup>d</sup> | 95% CI <sup>d</sup> |
|---|---|---|---|---|
| 100 (80 evaluable) | 20% | | (17.3%, 23.1%) | (16.0%, 25.0%) |
| | 30% | 1.0 | (26.0%, 34.7%) | (24.0%, 37.5%) |
| | 40% | | (34.6%, 46.2%) | (32.0%, 50.0%) |
| | 20% | | (16.8%, 23.8%) | (15.3%, 26.1%) |
| | 30% | 1.2 | (25.2%, 35.7%) | (23.0%, 39.2%) |
| | 40% | | (33.6%, 47.6%) | (30.6%, 52.2%) |
| 50 (40 evaluable) | 20% | | (16.3%, 24.6%) | (14.5%, 27.5%) |
| | 30% | 1.0 | (24.4%, 36.9%) | (21.8%, 41.3%) |
| | 40% | | (32.5%, 49.2%) | (29.1%, 55.1%) |



 Date: 15Nov2024
Statistical Analysis Plan

| Number of participants/arm <sup>a</sup> | Mean<br>percentage<br>Ki-67 in<br>two weeks <sup>b</sup> | SD of log-<br>transformed<br>percent<br>change in Ki-<br>67 <sup>c</sup> | 80% CI <sup>d</sup> | 95% CI <sup>d</sup> |
|---|---|---|---|---|
| | 20% | | (15.6%, 25.6%) | (13.6%, 29.4%) |
| | 30% | 1.2 | (23.4%, 38.4%) | (20.4%, 44.0%) |
| | 40% | | (31.2%, 51.2%) | (27.3% 58.7%) |

a. Approximately 100 participants will be enrolled to the ARV-471 arm with 80 participants providing valid Ki-67 data. Approximately 50 participants will be enrolled to the anastrozole arm with 40 participants providing valid Ki-67 data.

Table 2 Confidence Intervals for the Ratio Between the Mean Percentage of Baseline Values for Ki-67 Observed from ARV-471 and Anastrozole Arms (Ki-67 Evaluable Participants N=120)

| Mean<br>percentage<br>Ki-67 with<br>ARV-471 <sup>a</sup> | Mean<br>percentage<br>Ki-67 with<br>anastrozole <sup>a</sup> | SD of log-<br>transformed<br>percentage<br>Ki-67 b | Difference of mean<br>percentage Ki-67<br>(anastrozole –<br>ARV-471) | 80% CI for the ratio<br>of mean percentage<br>Ki-67 ° | 95% CI for the ratio of mean percentage Ki-67 ° |
|---|---|---|---|---|---|
| 20% | 30% | 1.0 | | (1.17, 1.93) | (1.02, 2.20) |
| 30% | 40% | 1.0 | 1.0 | (1.71, 1.04) | (0.91, 1.96) |
| 20% | 30% | 1.2 | | (1.11, 2.02) | (0.95, 2.38) |
| 30% | 40% | 1.2 | | (0.99, 1.80) | (0.84, 2,11) |
| 20% | 28% | 1.0 | | (1.09, 1.80) | (0.95, 2.05) |
| 30% | 38% | 1.0 | 8% | (0.99, 1.63) | (0.86, 1.86) |
| 20% | 28% | 1.2 | 0 / 0 | (1.04, 1.89) | (0.88, 2.22) |
| 30% | 38% | 1.2 | .4 | (0.94, 1.71) | (0.80, 2.01) |
| 20% | 25% | 1.0 | | (0.97, 1.60) | (0.85, 1.83) |
| 30% | 35% | 1.0 | 50/ | (0.91, 1.50) | (0.80, 1.71) |
| 20% | 25% | 1.2 | 5% | (0.93, 1.69) | (0.79, 1.98) |
| 30% | 35% | 1.2 | 1.2 | (0.86, 1.57) | (0.74, 1.85) |

a. Assume the relative reduction in Ki-67 attributed to ARV-471 exceeds the reduction attributed to anastrozole by 5%, 8% and 10% respectively in various scenarios.

#### 3 ANALYSIS SETS

For purposes of analysis, the following analysis sets are defined.

| <b>Analysis Set</b> | Description |
|---|---|
| Full Analysis Set | All enrolled participants who were randomized. Participants are analyzed according to the treatment they have been randomized to. |

b. Percentage Ki-67 in two weeks is defined as the ratio between Ki-67 reported from C1D15 visit and baseline respectively.

c. Ki-67 measurements are assumed to follow a log-normal distribution. The CIs are generated using the quantiles of the standard normal distribution on the log scale. Various values for the SD of the log-transformed Ki-67 percent change are provided to mimic the variability reported in the coopERA study (Hurvitz 2022). d. The CIs are presented in the original percentage scale through exponential-transformation of the CIs generated using the log-transformed Ki-67 data.

b. Assume the same SD for the log-transformed percent change in Ki-67 in either arm.

c. The ratio is defined as the mean percentage Ki-67 with anastrozole divided by the mean percentage Ki-67 with ARV-471. A ratio above unity (1) is in favor of ARV-471.



 Date: 15Nov2024
Statistical Analysis Plan

| Safety Analysis Set | All enrolled participants who receive at least 1 dose of study |
|---|---|
| | intervention. |
| Ki-67 Evaluable Set | All enrolled participants who were randomized and received at |
| | least one dose of study treatment and had evaluable Ki-67 |
| | measurements other than '0' or '< 1' from baseline and evaluable |
| | Ki-67 measurements from C1D15 visits. |
| Pharmacodynamic/ | The Pharmacodynamic/Biomarker analysis population is defined as |
| Biomarker Analysis | all enrolled participants with at least 1 of the Pharmacodynamic/ |
| Set(s) | Biomarkers evaluated at pre and/or post dose. |
| PK Concentration | The PK Concentration Analysis Set includes all participants in the |
| Analysis Set | Safety Analysis Set who have at least one plasma concentration |
| | (including those below the limit of quantification) for ARV-471, or |
| | ARV-473. |

#### 4 GENERAL CONSIDERATIONS

# 4.1 Programming Environment

All analyses will be conducted using SAS<sup>©</sup> version 9.4 or later.

#### 4.2 General Statistical Methods

The statistical analyses will be presented for the different analysis sets as defined in Section 3.

#### 4.2.1 Analysis Groups

The summary will be presented as ARV-471 200 mg, anastrozole 1 mg, and overall.

#### 4.2.2 Descriptive Summaries

In general, numerical variables will be summarized using descriptive statistics, displaying the number of participants in the respective analysis group, the number of participants with data, mean, standard deviation, median, minimum (min) and maximum (max).

Categorical variables will be summarized by using frequency counts and percentages. In addition, the number of participants with missing values will be displayed. Unless otherwise specified, the denominators used for calculating sample proportions will be the number of participants for each level of the analysis group defined above in the specified statistical analysis set (or a subset of the statistical analysis set under use).

Statistical methods for efficacy endpoints are described in section 10.2.

#### 4.2.3 Presentation Conventions

Means and medians will be presented by 1 additional decimal place and standard deviation will be presented by 2 additional decimal places than the standard presentation level of the respective data. Minimum and maximum values will be presented using the same number of decimal places as the original data. Confidence limits will be presented by 1 additional decimal place than corresponding point estimates.



 Date: 15Nov2024
Statistical Analysis Plan

If not otherwise stated, percentages will be presented to 1 decimal place. However, when the percentage (or estimated proportion) is 100% exactly, no decimal place will be shown, whereas a presented 100.0% implies that the percentage is in the half-open interval [99.95%, 100%). The number of decimal places may be adjusted, e.g., if the above default choices may lead to misinterpretation of the presented data.

If the number of participants in a category is 0, then percentage will not be displayed, and only a count of 0 will be shown. However, structural zeros (e.g., when the count is deemed to be 0 before obtaining actual data), missing data or inapplicable/unevaluable summaries will be presented as –, NA or NE.

In listings, data will be sorted by study part, arm, and participant. When appropriate by visit, scheduled timepoint or other identifiers for sequence or type of observation.

#### 4.3 Covariates and Strata

The stratification factors include Size of primary breast tumor ( $\leq 2$  cm,  $\geq 2$  to  $\leq 5$  cm, or  $\geq 5$  cm) and Baseline Ki-67 local score ( $\leq 20\%$  vs  $\geq 20\%$ ).

# 4.4 Subgroups

The primary endpoint will be presented for subgroups defined by the following criteria that will be derived from primary target lesion(s) and laboratory data instead of IRT:

- Size of primary breast tumor (T-stage):  $\leq 2$  cm,  $\geq 2$  to  $\leq 5$  cm, or  $\geq 5$  cm
- Baseline Ki-67 score (assessed locally):  $< 20\% \text{ vs} \ge 20\%$
- Baseline Ki-67 score (assessed centrally): < 20% vs > 20%

Other factors will be considered if the observed data imply potential findings of clinical interest.

# 4.5 Multiple Comparison/Multiplicity

This is a Phase 2 proof of concept study designed to generate data informing future studies about ARV-471. There are no plans for formal comparisons or hypotheses testing. There is no need for Type I error control. Descriptive statistics (including point estimates and two-sided CIs) will be provided for all parameters of interest. For information purposes, all the 2-sided CIs will be reported on both 80% and 95% confidence levels.

#### 5 DEFINITIONS & DATA HANDLING CONVENTIONS

# 5.1 Study Day, Duration, and Study Periods

#### 5.1.1 Study Day

Day 1 will be the date corresponding to the date of first ARV-471/anastrozole dose. Study Day = Assessment Date – Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date – Date of Day 1 for assessment prior to Day 1.

Unless otherwise specified, day is the primary time unit for derived time and durations. Derived time units include week=7 days, month=30.436875 days, and (Gregorian) year=365.2425 days=12 months. Thus, 1 month and 4 weeks are considered different.



Date: 15Nov2024
Statistical Analysis Plan

#### 5.1.2 Duration

Unless otherwise specified, duration of time is defined from the starting day through the ending day, inclusive of both boundary days.

#### 5.2 Analysis Visit Windows

Participant visits will be presented according to the nominal visit as obtained upon the eCRF. All values will be included in the participant data listings.

# 5.3 Baseline and Change from Baseline

The baseline value is defined to be the last non-missing assessment on/before the date of the first ARV-471/anastrozole dose. In case the randomized subject does not receive any treatment, the baseline will be the last assessment on/before the date of randomization. Change from baseline (CFB) calculations for a treatment window assessment will be the applicable treatment window assessment minus the baseline assessment. If either the treatment window assessment value or the baseline value is/are missing, then CFB will be set to missing for descriptive analysis purposes, unless otherwise specified.

# 5.4 Missing Data

# 5.4.1 Partial or Missing Dates and Time

The incomplete dates (e.g., start and/or stop dates of AE, concomitant medication) will be assumed as the most conservative value possible. In general, unless the available parts of the partial date preclude an AE to be treatment-emergent, the AE will be considered treatment-emergent; similarly, unless the available parts of the partial date exclude a medication to be concomitant, the medication will be considered as a concomitant medication.

For example, if the start date has a missing day value, the first day of the month will be imputed for study day computations, etc. If day is missing for an end date, the last day of the month will be imputed. If the start date has a missing month value, the first month of the year will be imputed for study day computations, etc. If month is missing for an end date, the last month of the year will be imputed. For determination of treatment-emergent status, the start date will be imputed as the date of the first dose of study drug, unless there is clear evidence (through comparison of partial dates/times) to suggest otherwise.

Date imputation will only be used for computational purposes such as treatment-emergent status, etc. Actual data values, as they appear in the original eCRFs, will be presented in the participant data listings. Non-monotone partial dates (e.g., day and month are non-missing but year is missing) need to be queried and resolved before DBL.

#### 5.4.2 Other Missing Values

Every effort will be made to obtain the required data at each scheduled evaluation from all participants who have been enrolled. In general, missing data will not be imputed and the data will be analyzed as they are recorded.



Date: 15Nov2024
Statistical Analysis Plan

#### 6 STUDY POPULATION AND DISPOSITION

# 6.1 Analysis Sets

The number and percentage of participants in each analysis set as defined in Section 3 will be summarized using the Full Analysis Set as described in Section 4.2.1.

Corresponding data listing will be provided using the Full Analysis Set.

# 6.2 Participant Disposition

The number and percentage of the following will be summarized using the Enrolled Participants /Ki-67 Evaluable Set as described in Section 4.2.1, including:

- Completed Treatment per Protocol
- ARV-471/Anastrozole early discontinuation
- Reason for ARV-471/Anastrozole early discontinuation
  - o Disease Progression per Response Criteria
  - o Clinical Progression
  - o Withdrawal of Consent
  - o Significant non-compliance
  - o Pregnancy
  - o Death
  - o Adverse Event
  - Study Terminated by Sponsor
  - o Lost to Follow-up
  - Other
- Completed study per Protocol
- Study early discontinuation
- Reason for study early discontinuation
  - o Withdrawal of Consent
  - Study Terminated by
  - o Sponsor
  - o Lost to Follow-up
  - o Death
  - o Other

Disposition of participants will be provided in a data listing using the Full Analysis Set.

Additionally, the number of participants with Tumor Biopsies (including Ki-67 and PgR636, etc.) at Screen/Cycle 1 day 15/ Cycle 6 day 18/Unscheduled will be summarized. The number and percentage of participants with the tested result or uninterpretable per test per visit will be summarized.

#### **6.3** Protocol Deviations

Protocol Deviation Management version: 1.0 dated 04 Jan 2023 (by Translational Research In Oncology) defined the study specific procedures and responsibilities for managing Protocol Deviations. Protocol Deviation severity includes minor, major or critical. The deviations will be categorized as:

- Informed Consent
- IMP/NIMP



 Date: 15Nov2024
Statistical Analysis Plan

- Protocol Compliance
- Safety
- ICH/GCP

All protocol deviations in each arm will be summarized by severity and categories. Protocol Deviation will also be listed in the Full Analysis Set.

#### 7 DEMOGRAPHICS AND DISEASE CHARACTERISTICS

# 7.1 Demographics and Baseline Characteristics

The following demographic characteristics will be summarized using Full Analysis Set and Ki-67 Evaluable Set as described in Section 4.2.1:

- Age (as reported in EDC) (n, mean, SD, minimum, maximum)
- Sex (female)
- Age group (age  $\geq 60$ , or age < 60)
- Race (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or other Pacific Islander, White, Other, Unknown)
- Ethnicity (Hispanic or Latino, not Hispanic or Latino, not reported)
- Weight (kg) at baseline (n, mean, SD, minimum, maximum)
- Height (cm) at baseline (n, mean, SD, minimum, maximum)
- ECOG Status (0, 1)
- Size of primary breast tumor (T-stage) ( $\leq 2$  cm,  $\geq 2$  to  $\leq 5$  cm, or  $\geq 5$  cm)
- Post-menopausal reason (Prior bilateral oophorectomy, Age >= 60 years, Age < 60 and amenorrheic for at least 12 months and FSH/estradiol in the postmenopausal range)

Demographic characteristics will also be provided in a data listing using the Full Analysis Set.

# 7.2 Disease Staging and Disease Characteristics

The following disease staging and disease characteristics will be summarized using the Full Analysis Set and Ki-67 Evaluable Set described in Section 4.2.1:

- Time since initial diagnosis (months), defined as time from the date of initial diagnosis to the date of first ARV-471/anastrozole dose (n, mean, SD, minimum, maximum)
- Time since current staging (months), defined as time from the date of current staging to the date of first ARV-471/anastrozole dose (n, mean, SD, minimum, maximum)
- Primary diagnosis (ER+ HER2- Breast Cancer)
- Stage at initial diagnosis (Stage 0, Stage IA, Stage IB, Stage IIA, Stage IIIB, Stage IIIA, Stage IIIB, Stage IIIC, Stage IV, Unknown)
- Disease stage at screening (Stage 0, Stage IA, Stage IB, Stage IIA, Stage IIIA, Stage IIIB, Stage IIIC, Stage IV, Unknown)
- Primary tumor at initial diagnosis (TX, T0, Tis, T1mi, T1a, T1b, T1c, T2, T3, T4a, T4b, T4c)
- Primary tumor at screening (TX, T0, Tis, T1mi, T1a, T1b, T1c, T2, T3, T4a, T4b, T4c)



 Date: 15Nov2024
Statistical Analysis Plan

- Imaging modality for primary tumor at screening (CT, MRI, Ultrasound, Mammogram)
- Regional lymph node at initial diagnosis (cNX, cN0, cN1, cN2a, cN2b, cN3a, cN3b, cN3c)
- Regional lymph node at screening (cNX, cN0, cN1, cN2a, cN2b, cN3a, cN3b, cN3c)
- Distant metastasis at initial diagnosis (M0, M1, Unknown)
- Distant metastasis at screening (M0, M1, Unknown)
- Histopathological classification at initial diagnosis (In-Situ Carcinoma, Invasive Ductal Carcinoma, Invasive Lobular Carcinoma, Invasive Mixed Ductal and Lobular Breast Carcinoma, Invasive Carcinoma NOS, Invasive Adenocarcinoma NOS, Tubular Carcinoma, Invasive Mucinous Adenocarcinoma, Other)
- Histopathological classification at screening (In-Situ Carcinoma, Invasive Ductal Carcinoma, Invasive Lobular Carcinoma, Invasive Mixed Ductal and Lobular Breast Carcinoma, Invasive Carcinoma NOS, Invasive Adenocarcinoma NOS, Tubular Carcinoma, Invasive Mucinous Adenocarcinoma, Other)
- Histopathological grade at initial diagnosis (Grade 1, Grade 2, Grade 3, Grade X)
- Histopathological grade at screening (Grade 1, Grade 2, Grade 3, Grade X)
- Planned type of breast surgery (Breast conserving surgery, Mastectomy)

The disease staging and disease characteristics will be listed using Full Analysis Set.

## 7.3 Disease Staging at Post-Surgery

The number and percentage of subjects with the following disease staging at post-surgery will be summarized using the Full Analysis Set and Ki-67 Evaluable Set described in Section 4.2.1:

Pathologic Tumor - ypT, n(%)

- ypTx
- ypT0
- ypTis
- ypT1mi
- ypT1a
- ypT1b
- ypT1c
- vpT2
- ypT3
- ypT4a
- ypT4b
- vpT4c

Multiple Foci of Residual Tumor?, n(%)

- Yes
- No

Pathologic Lymph Nodes - ypN, n(%)

- ypNX
- ypN0
- ypN0(i+)
- ypN0(mol+)



Date: 15Nov2024
Statistical Analysis Plan

- ypN1
- ypN1mi
- ypN1a
- ypN1b
- ypN1c
- ypN2
- ypN2a
- ypN2b
- ypN3
- ypN3a
- ypN3b
- ypN3c

Distant Metastasis (M), n(%)

- M0
- pM1
- Unknown

Lymphatic Vascular Invasion Classification, n(%)

- Present
- Not Present
- Unknown

The disease staging at post-surgery will be listed using Full Analysis Set.

# 7.4 Molecular Biology of Disease at Baseline

The molecular biology of disease - HER2 status, Ki67, Estrogen receptor, Progesterone receptor at baseline will be summarized using the Full Analysis Set and Ki-67 Evaluable Set:

- Perform of HER2 status, Ki67, Estrogen receptor, Progesterone receptor (Yes, No)
- Sample site of HER2 status, Ki67, Estrogen receptor, Progesterone receptor (Breast, Lymph Node, Other)
- HER2 analytical method (IHC, ISH)
- HER2 analytical result (0, 1+, 2+, 3+, Positive, Negative, Unknown)
- % of Tumor cells with Ki67 (assessed locally) (n, mean, SD, minimum, maximum, < 20% vs  $\geq 20\%$ )
- % of Tumor cells with Ki67 (assessed centrally) (n, mean, SD, minimum, maximum,  $< 20\% \text{ vs} \ge 20\%$ )
- % of Tumor cells with Estrogen receptor (n, mean, SD, minimum, maximum, < 10% vs  $\geq$  10%)
- % of Tumor cells with Progesterone receptor (n, mean, SD, minimum, maximum, < 1% vs  $\geq$  1%)

The molecular biology of disease will be listed using Full Analysis Set.

#### 7.5 Prior Cancer Related Surgery/Biopsy

The following prior cancer related surgery/biopsy characteristics will be summarized descriptively using Full Analysis Set as described in Section 4.2.1:

• Any prior surgery/biopsy related to the disease under trial (Yes)



Date: 15Nov2024
Statistical Analysis Plan

- Procedure (Sentinel node biopsy, Axillary sampling, Fine needle aspiration, Core needle biopsy, Other)
- Procedure location (Breast, Lymph node, Other)
- Laterality (Left, Right, Bilateral, Not applicable)
- Time since most recent surgery/biopsy (months), defined as time from the most recent date of surgery to the date of first ARV-471/Anastrozole dose (n, mean, SD, minimum, maximum)

#### 7.6 Medical History

Medical histories are coded according to Medical Dictionary for Regulatory Activities (MedDRA version 27.0 or higher) and will be classified as system organ class and preferred terms.

The number and percentage of participants will be summarized according to system organ class and preferred terms. If a participant has more than one disease within a system organ class and/or preferred terms the participant will be counted only once per system organ class or preferred terms.

The medical history will be listed using the Full Analysis Set.

#### 8 PROTOCOL-REQUIRED DRUG EXPOSURE AND COMPLIANCE

The dosing data for ARV-471 and Anastrozole be summarized descriptively using the Safety Analysis Set as described in Section 4.2.1.

The follow exposure parameters for ARV-471 and Anastrozole will be derived separately and will be summarized with n. mean, sd, median, min, max:

- **Duration of treatment** (week) is defined as the time from the date of first dose to the date of last dose
- **Cumulative dose** (mg) is the sum of 'Actual total daily dose' × (End date- Start date+1) per record
- **Absolute Dose Intensity** (mg/week) is defined as (Cumulative Dose (mg)/(Duration of Treatment (week).
- Relative Dose Intensity (%) is defined as (Absolute Dose Intensity (mg/week))/ (Initial Planned Weekly Dose (mg/week). ARV-471 Initial Planned Weekly Dose (mg/week) is 1400 mg/week (200\*7). Anastrozole Initial Planned Weekly Dose (mg/week) is 7 mg/week (1\*7).
- **Total planned dose** (mg) is the sum of 'Planned total daily dose' × (End date- Start date+1) per record
- **Compliance** is 100\*(Cumulative dose/Total planned dose)
- Number of compliant patients (with compliance  $\geq 80\%$   $\leq 120\%$ ).

The number and percentage of participants with dose discontinued, dose interrupted, dose reduced, dose increased, reasons for the action taken (Adverse event, Participant missed/Skipped dose, Medication error, Other) will be presented. All dosing data (including



 Date: 15Nov2024
Statistical Analysis Plan

the above derived dosing parameters) will also be presented in a data listing using the Safety Analysis Set.

#### 9 PRIOR AND CONCOMITANT THERAPIES

Full Analysis Set will be used to list diagnostic and medical procedures.

# 9.1 Prior and Concomitant Medications

Prior and concomitant medications and on-study anti-cancer therapy will be coded according to WHO-Drug B3 Global version September 2024 or most current version with Anatomical Therapeutic Chemical (ATC) Classification System and preferred names (PN). Prior medications include the medications that are ended before Day 1. Concomitant medications include the medications that are used/started on/after Day 1 and within 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

The number and percentage of participants with prior medication or concomitant medications will be summarized by ATC level 2 category and preferred name will be summarized using the Full Analysis Set as described in Section 4.2.1. If a participant received more than 1 drug within an ATC2 or PN, the participant will be counted only once for this ATC2 and PN.

Prior and concomitant medications and on-study anti-cancer therapy will also be provided in a data listing using the Full Analysis Set.

#### 10 EFFICACY ANALYSES

#### 10.1 Assessment

#### 10.1.1 Tumor Biopsies

Tumor samples for Ki67, estrogen receptor (ER), and PD endpoints will be collected at screening, C1D15 (+ 5 days), surgical resection (after approximately 5.5 months of treatment). Ki-67 expression will be measured by IHC. ER expression will be measured by quantitative immunofluorescence. These analyses will be done in a blind manner at the **central laboratories**.

#### 10.1.2 Radiographic Imaging

Radiographic imaging (eg, breast ultrasound, breast MRI with contrast, and/or mammogram) will be performed at screening, C4D1 (± 7 days), and within 7 days prior to surgical resection. Tumor responses are assessed based on mRECIST criteria by Investigator. The overall tumor response per visit includes Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Not Evaluable (NE).

#### 10.1.3 Physical Exam

Caliper based measurements of the primary breast tumor will be performed during physical exam at screening, day 1 of cycle 1~cycle 6, and C6D18 prior to the surgery.



 Date: 15Nov2024
Statistical Analysis Plan

#### 10.1.4 Local Pathological Assessments

Local pathological assessments of the tissue include surgical resection (performed after approximately 5.5 months of treatment) for surgical procedure (Breast Conserving Surgery (BCS), Mastectomy), post-surgery pathologic stage (ypT and ypN stage), and post-surgery pathologic response (Pathological Complete Response (pCR), Pathological Partial Response (pPR), No Response (NR)).

# 10.2 Definitions of Efficacy Endpoints

# 10.2.1 Ki-67 Percentage at C1D15 (Primary)

The tumor biopsies Ki-67 expression (%) at baseline and C1D15 will be collected. The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\log(\text{Ki-67} \text{ at C1D15}) - \log(\text{Ki-67} \text{ at baseline})$  and the treatment effects will be back transformed. The percentage change of Ki67 from baseline at C1D15 will be derived as =  $100 \times (\% \text{ Ki67} \text{ at C1D15} - \% \text{ Ki67} \text{ at baseline})/\% \text{ Ki67}$  at baseline.

If the value at C1D15/surgery is reported as "0", "<1", or other special characters will be imputed as '0.1" with % as unit.

## 10.2.2 ER Percentage at C1D15

The tumor biopsies ER expression will be reported with AQUA score (absolute quantification score in arbitrary units) at baseline and C1D15. The endpoint is the percentage change of ER expression obtained from C1D15 visit and baseline, which will be derived as =  $100 \times (ER AQUA score at C1D15 - ER AQUA score at baseline)/ ER AQUA score at baseline.$ 

# **10.2.3 pCR Rate**

Post-Surgery Pathological Response will be reported as Pathological Complete Response (pCR), Pathological Partial Response (pPR), No Response (NR). Additionally, pCR will also be programmatically derived according to the definition in the protocol using Disease Staging – Post-Surgery data: pCR is defined as no invasive cancer in the breast and sampled axillary lymph nodes following completion of neoadjuvant systemic therapy (ie, Pathologic Tumor - ypT = ypT0 or ypTis, and Pathologic Lymph Nodes – ypN = ypN0 in the current AJCC staging system). pCR rate is the proportion of participants with pCR, which are either determined by site pathologist or derived based on EDC data.

#### 10.2.4 mPEPI Score and mPEPI0 Rate

Modified Pre-operative Endocrine Prognostic Index (mPEPI) score will be derived from factors assigned a numerical score following Neoadjuvant endocrine treatment (NET) according to the following table (Ellis 2008, Sanati 2015). The factors include Ki67 expression in the surgical specimen, pathologic tumor size, and lymph node status. Total mPEPI score (mPEPI\_T) per participant is the sum of mPEPI score of each factor. mPEPI0 rate is the proportion of participants achieving mPEPI T 0 after treatment (before surgery).

| Pathology, biomarker status | mPEPI Score |
|-----------------------------|-------------|
| Pathological tumor size | |
| T1/2 | 0 |
| T3/4 | 3 |
| Node status | |



 Date: 15Nov2024
Statistical Analysis Plan

| Pathology, biomarker status | mPEPI Score |
|-----------------------------|-------------|
| Negative | 0 |
| Positive | 3 |
| Ki67 level (centrally) | |
| 0%-2.7% | 0 |
| >2.7%-7.3% | 1 |
| >7.3%–19.7% | 1 |
| >19.7%-53.1% | 2 |
| >53.1% | 3 |

# 10.2.5 Breast Conserving Surgery (BCS) Rate

Breast conserving surgery (BCS) Rate is the proportion of participants receiving breast conserving surgery.

# 10.2.6 Radiographic Response per mRECIST in Primary Tumor during Cycle 6

The percentage of subjects with Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Not Evaluable (NE) per mRECIST at Cycle 6 (before surgery) will be calculated.

Percentage change of target lesions and target lesion (primary tumor) from baseline at each visit and the best percentage change of target lesions and target lesion (primary tumor) from baseline will be summarized.

#### 10.2.7 Caliper-Based Response

The percentage change from the baseline of the primary breast tumor in physical exam will be calculated by visit. The best percentage change from baseline, Caliper-based response, which is maximum percentage decrease or minimum percentage increase if there is no decrease per participant.

#### **10.2.8 CCCA Rate**

Complete cycle cell arrest (CCCA) at Week 2/surgery is defined as Ki67 score  $\leq$  2.7%. CCCA rate is the proportion of participants achieving CCCA at Week 2 (or C1D15)/surgery.

#### 10.3 Analysis of Efficacy Variables

All efficacy data and the derived endpoints will be listed. The endpoints will be analyzed below.

# 10.3.1 Ki-67 Percentage at C1D15 (Primary)

Analysis of Ki-67 reduction will be based on Ki-67 Analysis Set.

The log-transformed Ki-67 after approximately 2 weeks of treatment as a percentage of the baseline value, ie, the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, will be modelled using a GLM, with both derived stratification factors (ie, baseline Ki-67 score (local laboratory and central laboratory) and the tumor size) and treatment as covariates, or with treatment as only covariate Treatment effects for each arm will be summarized using the LSM and their two-sided 80% CI and 95% CI on the log scale. In addition, for easier interpretation of the data, the treatment effects will be back transformed



 Date: 15Nov2024
Statistical Analysis Plan

and expressed as the geometric means and their CIs on the original percentage scale by treatment arm.

LSM difference between two arms and its two-sided 80% CI and 95% CI will be calculated on the log scale. The treatment effects will be back transformed and expressed as the geometric means and their CIs on the ratio of original percentage scale.

The calculation will use Ki-67 score from central laboratory.

Same analysis will be performed for the Ki-67 Percentage at surgery using Full Analysis Set.

Spider plot for individual Ki-67 value at C1D15 and Surgery, Box plot for Ki-67 percentage change from baseline at C1D15 and Surgery will be presented.

#### 10.3.2 Binary or Categorical Endpoints

Analysis of these parameters will be based on Full Analysis Set. The participants without post baseline assessment will be considered as Not Evaluable in Post-Surgery Pathological Response and Radiographic Response per mRECIST and counted in denominator.

The number and percentage of participants with Post-Surgery Pathological Response and Radiographic Response per mRECIST during Cycle 6 will be summarized. pCR rate, mPEPI rate, BCS rate, and CCCA rate will be computed by treatment arm along with the 80% CI and 95% CI using Wilson method.

Odds ratios of CCCA rate and mPEPI rate between the treatments adjusted for the stratification factors through the Cochran-Mantel-Haenszel method will be provided along with their 80% CIs and 95% CIs.

The number and percentage of participants with Post-Surgery Disease Staging will be summarized using both Full Analysis Set and Ki-67 Analysis Set.

#### 10.3.3 Primary Tumor Assessments

Caliper-based primary breast tumor size in physical exam and its percentage change from baseline at each visit will be summarized with n, mean, sd, median, min, max using Full Analysis Set. Caliper-based response is the best percentage change from baseline (maximum percentage decrease or minimum percentage increase if there is no decrease per participant), which will be presented with n. mean, sd, median, min, max and Waterfall Plot.

Sum of target lesion and primary target lesion at each visit will be calculated separately. The size and its percentage change from baseline at each visit will be summarized with n. mean, sd, median, min, max using Full Analysis Set. The best percentage change from baseline (maximum percentage decrease or minimum percentage increase if there is no decrease per participant) will be presented in with n. mean, sd, median, min, max and Waterfall Plot.

A spider plot for the percentage change of target lesion from baseline will be presented.

# 10.3.4 ER AQUA Score Percentage at C1D15 and Surgery

ER AQUA score reduction will be analyzed using Full Analysis Set with Normalized AQUA score from Navigate transfer at screen and C1D15/Surgery. The percentage change of ER AQUA score from baseline will be analyzed using a GLM, with both derived stratification factors (ie, baseline Ki-67 score (from central lab only) and the tumor size) and treatment as covariates, or with treatment as only covariate. Treatment effects for each arm and difference



Date: 15Nov2024
Statistical Analysis Plan

between two arms will be summarized using the LSM and their two-sided 80% CI and 95% CI. Additionally, the percentage change of log-transformed ER AQUA score from baseline will be analyzed using a GLM with treatment as only covariate. Treatment effects for each arm and difference between two arms will be summarized using the LSM and their two-sided 80% CI and 95% CI. The treatment effects will be back transformed and expressed as the geometric means and their CIs on the ratio of original scale. Baseline values of 0 are not imputed and the participants will be excluded in the summary. Post-baseline value of 0 will be imputed as 0.1 for the derivation of log transform analysis.

#### 10.3.5 PR H-score Percentage at C1D15 and Surgery

PR (progesterone receptor) H-score (H-score = (SCORE\_1)\*1 + (SCORE\_2)\*2 + (SCORE\_3)\*3) reduction will be analyzed using Full Analysis Set with PgR636 assessment at screen and C1D15/Surgery. If a value includes a special character such as "<" or ">", the value after the special character will be used for the derivation of H-score. Baseline values of 0 are not imputed and the participants will be excluded in the summary. Post-baseline value of 0 will be imputed as 0.1 for the derivation of log transform analysis.

The percentage change of PR H-score from baseline will be analyzed using a GLM with treatment as only covariate. Treatment effects for each arm and difference between two arms will be summarized using the LSM and their two-sided 80% CI and 95% CI. Additionally, the percentage change of log-transformed PR H-score from baseline will be analyzed using a GLM with treatment as only covariate. Treatment effects for each arm and difference between two arms will be summarized using the LSM and their two-sided 80% CI and 95% CI. The treatment effects will be back transformed and expressed as the geometric means and their CIs on the ratio of original scale. For the log transformation, observed 0 will be converted to 0.1 for calculation.

Spider plot for individual PR H-score at C1D15 and Surgery, Box plot for PR H-score percentage change from baseline at C1D15 and Surgery will be presented.

#### 10.3.6 Subgroup Analyses

Summaries of the primary endpoint will be presented for subgroups defined by the following criteria:

- Size of primary breast tumor (T-stage):  $\leq 2$  cm,  $\geq 2$  to  $\leq 5$  cm, or  $\geq 5$  cm
- Baseline Ki-67 score (assessed locally):  $< 20\% \text{ vs} \ge 20\%$
- Baseline Ki-67 score (assessed centrally):  $< 20\% \text{ vs} \ge 20\%$

Other factors will be considered if the observed data imply potential findings of clinical interest. Results of the primary analysis will be reported within each subgroup.

# 11 SAFETY ANALYSES

All safety analyses will be performed on the Safety Analysis Set.



 Date: 15Nov2024
Statistical Analysis Plan

#### 11.1 Adverse Events

Adverse events (AE) will be coded using MedDRA 27.0 or higher and graded according to the NCI-CTCAE 5.0.

Summaries of AEs will be based on treatment-emergent AEs (TEAEs). A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV-471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last). TEAE summaries will be presented by System Organ Class (SOC) and Preferred Term (PT). Although AEs may be reported more than once for a PT or SOC in a participant, each participant will only be counted once per SOC and PT.

An overview of Treatment Emergent Adverse Events (TEAEs), including number and percent of participants who had any TEAE, TEAE related to study drug, serious TEAEs, serious TEAEs related to study drug, TEAE leading to drug withdrawn, TEAEs leading to drug interrupted, TEAEs leading to dose reduced, TEAE related to study drug leading to drug withdrawn, TEAEs related to study drug leading to drug interrupted, TEAEs related to study drug leading to dose reduced, TEAEs ≥ grade 3 in severity, TEAEs related to study drug ≥ grade 3 in severity, TEAE leading to death.

Number and percentages of participants with TEAEs will be presented by SOC and PT in the following summaries:

- TEAEs
- TEAEs related to study drug
- TEAEs with grade 3 or higher
- TEAEs with grade 3 or higher related to study drug
- Serious TEAEs
- Serious TEAEs to study drug
- TEAEs leading to drug withdrawn
- TEAEs related to study drug leading to drug withdrawn
- TEAEs leading to drug interrupted
- TEAEs related to study drug leading to drug interrupted
- TEAEs leading to dose reduced
- TEAEs related to study drug leading to dose reduced
- TEAEs leading to death

Number and percentages of participants with TEAEs will be presented by PT in the following summaries:

- TEAEs
- TEAEs related to study drug
- Serious TEAEs
- Serious TEAEs to study drug

Tornado plots for treatment emergent adverse events in  $\geq$  5% subjects of any arm by Preferred Term and with Grade 3 or higher by Preferred Term will be presented.



 Date: 15Nov2024
Statistical Analysis Plan

Number and percentages of participants with TEAEs will be presented by SOC, PT and maximum CTCAE grade in the following summaries:

- TEAEs
- TEAEs related to study drug
- Serious TEAEs
- Serious TEAEs to study drug

Number and percentages of participants with MedDRA SMQ for Torsade de Pointes will be presented by PT and maximum CTCAE grade. PTs include Electrocardiogram QT interval abnormal, Electrocardiogram QT prolonged, Long QT syndrome, Long QT syndrome congenital, Torsade de pointes, Ventricular tachycardia, Arrhythmic storm, Cardiac arrest, Cardiac death, Cardiac fibrillation, Cardio-respiratory arrest, Electrocardiogram repolarization abnormality, Electrocardiogram U wave inversion, Electrocardiogram U wave present, Electrocardiogram U-wave abnormality, Loss of consciousness, Seizure, Sudden cardiac death, Sudden death, Syncope, Ventricular arrhythmia, Ventricular fibrillation, Ventricular flutter, Ventricular tachyarrhythmia.

Participant listings will be provided for participants with all AEs.

#### 11.2 Deaths

The reason of subject death will be summarized using Safety Analysis Set. Death information will be provided in a listing.

# 11.3 Vital Signs

Vital signs parameters with abnormal clinically significant will be provided in a data listing.

#### 11.4 Clinical Laboratory

For lab values in the form of  $\langle x, \leq x \rangle$ , below lower quantification limit, etc., the value will be imputed as x/2 or half of the lower quantification limit for the purpose of numerical descriptive summary. For lab values in the form of  $\geq x, \geq x$ , above upper quantification limit, etc., the value will be imputed as x or upper quantification limit for the purpose of numerical descriptive summary. When such imputation occurs, footnotes will be presented to clarify the imputation rule. The original lab values will be presented in data listings.

The Laboratory test value and change from baseline for continuous parameters over hematology tests, chemistry tests, coagulation tests will be summarized using descriptive statistics (n, mean, SD, median, minimum, maximum) by visit.

The value of hematology tests, coagulation tests, and chemistry tests will be graded with CTCAE 5.0. Shift of hematology tests, coagulation tests, and chemistry tests from baseline CTCAE grade to the worst postbaseline CTCAE grade will be presented. If a parameter includes both hypo- and hyper- CTCAE grade derivation, hypo- and hyper- will be tabulated separately. If the baseline is not CTCAE gradable (e.g., AST increase), the baseline measurement will be categorized as low/normal/high according to reference ranges.

Laboratory hematology, chemistry, coagulation, and urinalysis will be provided in data listings.



Date: 15Nov2024
Statistical Analysis Plan

# 11.5 12-Lead Electrocardiogram

Triplicate 12-lead ECGs include Heart Rate, PR Interval, QRS Duration, QT Interval, QTcB Interval (Bazette's), QTcF Interval (Fridericia's). The mean of each parameter per visit will be used to summary. The value and change from baseline at each visit/timepoint will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum). If a parameter is tested only one time, the value will be used for summary directly.

The number and percentage of participants in the following QTcB and QTcF categories will also be summarized:

- QTcB/QTcF at Baseline
  - o QTcB/QTcF >450 msec
  - o QTcB/QTcF >480 msec
  - o QTcB/QTcF >500 msec
- QTcB/QTcF Worst Post-Baseline
  - o QTcB/QTcF >450 msec
  - o QTcB/QTcF >480 msec
  - o QTcB/QTcF >500 msec
- QTcB/QTcF Worst Change from Baseline
  - $\circ$  >30 msec
  - o >60 msec

All ECG data (scheduled or unscheduled) will be displayed in a data listing.

# 11.6 Eastern Cooperative Oncology Group (ECOG) Performance Status

All ECOG scores will be provided in a data listing.

#### 12 OTHER ANALYSES

#### 12.1 Pharmacokinetics

Pharmacokinetic blood samples from participants receiving ARV-471 may be collected at pre-dose, 1 hour ( $\pm$  15 min) post-dose, 2 hours ( $\pm$  15 min) post-dose, 4 hours ( $\pm$  30 min) post-dose on Cycle 2 Day 1, pre-biopsy on Cycle 1 Day 15, and pre-surgery on Cycle 6 Day 18. The plasma concentrations of ARV-471 and ARV-473 of individual participants will be presented by listings and summarized.

The plasma concentrations of ARV-471 and ARV-473 on Cycle 2 Day 1 will be summarized by time-point using PK analysis set. The following concentration data on Cycle 2 Day 1 should be flagged and excluded from summary.

- a. Pre-dose samples are collected after dosing time.
- b. Post-dose samples are collected out of time window.
- c. Received ARV-471 dose is different from the planned dose

Correlation of population PK model-derived PK parameters (AUC, Cmin, Cmax) with ER reduction or other response parameters may be explored. The analysis plan and report may be provided separately.



 Date: 15Nov2024
Statistical Analysis Plan

#### 12.2 Pharmacodynamics

Exploratory analyses include evaluation of the effects of ARV-471 and anastrozole, respectively, on Ki-67, and ER degradation by ARV-471 in tumors at the time of surgical resection. Changes in ER and Ki-67 expression between baseline and Cycle 6 surgical tumor samples as well as rates of CCCA in the cycle 6 surgical samples will be summarized for the full analysis set. The ER changes will be reported as a percentage change from baseline and derived as: 100 x (ER AQUA at surgery – ER AQUA at baseline)/ER AQUA at baseline. The Ki67 changes will be reported as a percentage change from baseline and derived as: 100 x (% Ki67 at surgery - % Ki67 at baseline)/% Ki67 at baseline. Treatment effects for each arm will be summarized using the LSM and their two-sided 80% CI and 95% CI.

Complete cycle cell arrest (CCCA) at surgical resection is defined as Ki67 score  $\leq$  2.7%. CCCA rate is the proportion of participants achieving CCCA at surgical resection.

Any additional explorative pharmacodynamics analysis if needed will be described in a separate plan.

#### 13 SCHEDULE OF ANALYSES

The final analysis will take place when all participants discontinue the study.

#### 14 REFERENCES

- 1. Ellis MJ, etc. Outcome Prediction for Estrogen Receptor–Positive Breast Cancer Based on Postneoadjuvant Endocrine Therapy Tumor Characteristics. J Natl Cancer Inst. 2008 Oct 1; 100(19): 1380–1388.
- 2. Hurvitz SA, Quiroga V, Park YH, et al. Neoadjuvant giredestrant (GDC-9545) + palbociclib versus anastrozole + palbociclib in postmenopausal women with estrogen receptor-positive, HER2-negative, untreated early breast cancer: Primary analysis of the randomized, open-label, phase II coopERA breast cancer study. San Antonio Breast Cancer Symposium 2021. Cancer Res 15 February 2022; 82 (4\_Supplement): PD13–06.
- 3. ICH Harmonised Tripartite Guideline E9, Statistical Principles for Clinical Trials, 1998
- 4. ICH Harmonised Tripartite Guideline E3, Structure and Content of Clinical Study Reports. 1995
- 5. ICH Harmonised Tripartite Guideline E6(R1), Guideline for Good Clinical Practice, 1996
- 6. ICH guideline E2F, Note for guidance on development safety update reports, EMA/CHMP/ICH/309348/2008, September 2010
- ICH E9 (R1) addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical 6 principles for clinical trials, Step 2b (Draft), EMA/CHMP/ICH/436221/2017, 2017
- 8. Sanati S. etc. Abstract P4-11-13: Validation of the preoperative endocrine prognostic index in the ACOSOG (Alliance) Z1031 neoadjuvant aromatase inhibitor trial. Cancer Research, POSTER SESSION ABSTRACTS, MAY 01, 2015.





An Open-Label, Randomized, Non-Comparative Phase 2 Study of ARV-471 or Anastrozole in Post-Menopausal Women With ER+/HER2- Breast Cancer in the Neoadjuvant Setting

# **Table and Figure Shells**

1

Author:

SAP Version: v3.0

Table and Listing Shell Version: v2.0

Protocol No.: ARV-471-BC-201

Version:v2

Version Date: 15Nov2024

TLF Shells

# **SIGNATURE PAGE**



Protocol No.: ARV-471-BC-201

Version:v2

Version Date: 15Nov2024

TLF Shells

# INTRODUCTION

The following are mock table and listing shells. These represent the format of the analysis tables that will be programmed for this project. These are based on the statistical analysis plan (SAP) for study ARV-471-BC-201.

Statistical results are represented with placeholders such as "xxx.x." These placeholders will be populated with results when the tables are programmed based on the data.

These shells are in Microsoft Word, whereas the programmed tables are developed with SAS. Very minor differences in appearance should be expected between these shells and the programmed tables, although the general layout and format of the programmed tables will be consistent with these shells.

# TABLE OF CONTENTS

| R | EVISIONS | 12 |
|---|---|---|
| G | LOBAL CONVENTIONS | 13 |
| | Table 14.1.1.1 Summary of Analysis Sets Analysis Set: Full Analysis Set. | 16 |
| | Table 14.1.1.2 Summary of Participants with Tumor Biospsy Analysis Set: Full Analysis Set | 17 |
| | Table 14.1.2.1 Summary of Disposition and Discontinuation Analysis Set: Enrolled Participants | 18 |
| | Table 14.1.2.2 Summary of Disposition and Discontinuation Analysis Set: Ki-67 Evaluable Set | 19 |
| | Table 14.1.3 Summary of Protocol Deviation Analysis Set: Full Analysis Set | 20 |
| | Table 14.1.4.1 Summary of Demographic Characteristics Analysis Set: Full Analysis Set | 21 |
| | Table 14.1.4.2 Summary of Demographic Characteristics Analysis Set: Ki-67 Evaluable Set | 22 |
| | Table 14.1.5 Summary of Medical History by System Organ Class and Preferred Term Analysis Set: Full Analysis Set | 23 |
| | Table 14.1.6.1 Summary of Disease Staging and Disease Characteristics Analysis Set: Full Analysis Set | 24 |
| | Table 14.1.6.2 Summary of Disease Staging and Disease Characteristics Analysis Set: Ki-67 Evaluable Set | 27 |
| | Table 14.1.7.1 Summary of Disease Molecular Biology at Baseline Analysis Set: Full Analysis Set | 28 |
| | Table 14.1.7.2 Summary of Disease Molecular Biology at Baseline Analysis Set: Ki-67 Evaluable Set | 30 |
| | Table 14.1.8 Summary of Prior Cancer Related Surgery/Biopsy Analysis Set: Full Analysis Set | 31 |
| | Table 14.1.9 Summary of Prior Medication Analysis Set: Full Analysis Set. | 32 |
| | Table 14.1.10 Summary of Concomitant Medication Analysis Set: Full Analysis Set. | 33 |
| | Table 14.1.11 Summary of ARV-471 and Anastrozole Compliance and Exposure Analysis Set: Safety Analysis Set | 34 |
| | Table 14.2.1.1.1 Summary of Ki-67 Percentage Change from Baseline at C1D15 with Central Ki-67 as a Covariate Analysis Set Ki-67 Evaluable Set | |
| | Table 14.2.1.1.2 Summary of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 Percentage Change from Baseline at C1D15 with Local Ki-67 as a Covariate Analysis Set: February of Ki-67 | |
| | Table 14.2.1.1.3 Summary of Ki-67 Percentage Change from Baseline at C1D15 without Covariate Analysis Set: Ki-67 Evalual Set | |

| Cable 14.2.1.2.1 Summary of Ki-67 Percentage Change from Baseline at C1D15– Subgroup Analysis by Tumor Size Analysis Set: Ki-67 Evaluable Set |
|---|
| Cable 14.2.1.2.2 Summary of Ki-67 Percentage Change from Baseline at C1D15 – Subgroup Analysis by Local Ki-67 Baseline Score Analysis Set: Ki-67 Evaluable Set |
| Cable 14.2.1.2.3 Summary of Ki-67 Percentage Change from Baseline at C1D15– Subgroup Analysis by Central Ki-67 Baseline Score of 20% Analysis Set: Ki-67 Evaluable Set |
| Cable 14.2.1.2.4 Summary of Ki-67 Percentage Change from Baseline at C1D15 – Subgroup Analysis by Central Ki-67 Baseline Score of 5% Analysis Set: Ki-67 Evaluable Set |
| Cable 14.2.1.3.1 Summary of Ki-67 Percentage Change from Baseline at Surgery with Central Ki-67 as a Covariate Analysis Set: Gull Analysis Set |
| Table 14.2.1.3.2 Summary of Ki-67 Percentage Change from Baseline at Surgery with Local Ki-67 as a Covariate Analysis Set: 47 |
| Cable 14.2.1.3.3 Summary of Ki-67 Percentage Change from Baseline at Surgery without Covariate Analysis Set: Full Analysis Set 48 |
| Fable 14.2.1.4.1 Summary of Ki-67 Percentage Change from Baseline at Surgery – Subgroup Analysis by Tumor Size Analysis Set: Full Analysis Set 49 |
| Cable 14.2.1.4.2 Summary of Ki-67 Percentage Change from Baseline at Surgery – Subgroup Analysis by Local Ki-67 Baseline Score Analysis Set: Full Analysis Set. 51 |
| Cable 14.2.1.4.3 Summary of Ki-67 Percentage Change from Baseline at Surgery – Subgroup Analysis by Central Ki-67 Baseline Score Analysis Set: Full Analysis Set. 53 |
| Cable 14.2.1.5.1 Summary of Concordance Ki-67 Baseline Score between Central and Local Laboratories Analysis Set: Ki-67 Evaluable Set 55 |
| Sable 14.2.1.5.2 Summary of Concordance Central/Local Ki-67 Baseline Score with Randomization Baseline Ki-67 Score Analysis Set: Ki-67 Evaluable Set |
| Cable 14.2.1.5.3 Summary of Concordance Acutal Primary Breast Tumor Size with Randomization Primary Breast Tumor Size Analysis Set: Ki-67 Evaluable Set 57 |
| Fable 14.2.2.1.1 Summary of Post-Surgery Pathological Response and pCR Rate - Determined by Site Pathologist Analysis Set: Full Analysis Set 58 |

| Table 14.2.2.1.2 Summary of Post-Surgery Pathological Response and pCR Rate – Calculated Analysis Set: Full Analysis Set | 59 |
|---|---|
| Table 14.2.2.1.3.1 Summary of Post-Surgery Disease Staging Analysis Set: Full Analysis Set | 60 |
| Table 14.2.2.1.3.2 Summary of Post-Surgery Disease Staging Analysis Set: Ki-67 Evaluable Set | 61 |
| Table 14.2.2.2 Summary of Modified Pre-operative Endocrine Prognostic Index (mPEPI) Score and mPEPI 0 Rate Analysis Set: Full Analysis Set. | |
| Table 14.2.2.3 Summary of Breast Conserving Surgery (BCS) and BCS Rate Analysis Set: Full Analysis Set | 63 |
| Table 14.2.2.4 Summary of Radiographic Response per mRECIST during Cycle 6 Analysis Set: Full Analysis Set | 64 |
| Table 14.2.2.5.1 Summary of Complete Cycle Cell Arrest (CCCA) and CCCA Rate Analysis Set: Full Analysis Set | 65 |
| Table 14.2.2.5.2 Summary of Complete Cycle Cell Arrest (CCCA) and CCCA Rate – Subgroup Analysis by Central Ki-67 Baseli Score Analysis Set: Full Analysis Set. | |
| Table 14.2.3.1.1 Summary of the Primary Breast Tumor Change - Caliper-based Analysis Set: Full Analysis Set | 69 |
| Table 14.2.3.1.2 Summary of the Primary Breast Tumor Change - Caliper-based by Baseline Tumor Size Analysis Set: Full Analysis Set | 70 |
| Table 14.2.3.2.1 Summary of Target Lesion Change Analysis Set: Full Analysis Set | 71 |
| Table 14.2.3.2.2 Summary of Target Lesion Change by Baseline Tumor Size Analysis Set: Full Analysis Set | 72 |
| Table 14.2.3.3.1 Summary of Target Lesion (Primary Tumor) Change Analysis Set: Full Analysis Set | 73 |
| Table 14.2.3.3.2 Summary of Target Lesion (Primary Tumor) Change by Baseline Tumor SizeAnalysis Set: Full Analysis Set | 74 |
| Table 14.2.4.1.1 Summary of ER AQUA Score Percentage Change at C1D15 from Baseline Value Analysis Set: Full Analysis Se | |
| Table 14.2.4.1.2 Summary of ER AQUA Score Percentage Change at C1D15 from Baseline Value without Covariate Analysis Set: Full Analysis Set. | 76 |
| Table 14.2.4.1.3 Summary of Log-Transformed ER AQUA Score Change at C1D15 from Baseline Value without Covariate Analysis Set: Full Analysis Set | 77 |
| Table 14.2.4.2.1 Summary of ER AQUA Score Percentage Change at Surgery from Baseline Value Analysis Set: Full Analysis Set | et |
| Table 14.2.4.2.2 Summary of ER AQUA Score Percentage Change at Surgery from Baseline Value without Covariate Analysis Set: Full Analysis Set. | |
| Analysis Set: Full Analysis Set. | |
|---|---|
| Table 14.2.5.1.1 Summary of PR H-score Percentage Change at C1D15 from Baseline Value without Covariate Analysis Set | 8 |
| Table 14.2.5.1.2 Summary of Log-Transformed PR H-score Change at C1D15 from Baseline Value without Covar Set: Full Analysis Set | |
| Table 14.2.5.2.1 Summary of PR H-score Percentage Change at Surgery from Baseline Value without Covariate Analysis Set | |
| Table 14.2.5.2.2 Summary of Log-Transformed PR H-score Change at Surgery from Baseline Value without Cova<br>Set: Full Analysis Set | |
| Table 14.3.1 Summary of Treatment Emergent Adverse Events Overview Analysis Set: Safety Analysis Set | 8 |
| Table 14.3.2.1 Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term A Safety Analysis Set | • |
| Table 14.3.2.2 Summary of Treatment Emergent Adverse Events Related to Study Drug by System Organ Class a Term Analysis Set: Safety Analysis Set | |
| Table 14.3.2.3 Summary of Treatment Emergent Adverse Events with Grade 3 or Higher by System Organ Class Term Analysis Set: Safety Analysis Set | |
| Table 14.3.2.4 Summary of Treatment Emergent Adverse Events with Grade 3 or Higher Related to Study Drug by Class and Preferred Term Analysis Set: Safety Analysis Set | |
| Table 14.3.2.5.1 Summary of Treatment Emergent Adverse Events Leading to Drug Withdrawn by System Organ Preferred Term Analysis Set: Safety Analysis Set | |
| Table 14.3.2.5.2 Summary of Treatment Emergent Adverse Events Related to Study Drug Leading to Drug Withdom Organ Class and Preferred Term Analysis Set: Safety Analysis Set | |
| Table 14.3.2.6.1 Summary of Treatment Emergent Adverse Events Leading to Drug Interrupted by System Organ Preferred Term Analysis Set: Safety Analysis Set | |
| Table 14.3.2.6.2 Summary of Treatment Emergent Adverse Events Related to Study Drug Leading to Drug Interru<br>Organ Class and Preferred Term Analysis Set: Safety Analysis Set | ipted by System |

| Table 14.3.2.7.1 Summary of Treatment Emergent Adverse Events Leading Term Analysis Set: Safety Analysis Set | |
|---|---|
| Table 14.3.2.7.2 Summary of Treatment Emergent Adverse Events Related to Organ Class and Preferred Term Analysis Set: Safety Analysis Set | |
| Table 14.3.2.8 Summary of Treatment Emergent Adverse Events by Preferre | ed Term Analysis Set: Safety Analysis Set 89 |
| Table 14.3.2.9 Summary of Treatment Emergent Adverse Events Related to Analysis Set | |
| Table 14.3.2.10 Summary of Treatment Emergent Adverse Events by System Grade Analysis Set: Safety Analysis Set | |
| Table 14.3.2.11 Summary of Treatment Emergent Adverse Events Related to and Maximum CTCAE Grade Analysis Set: Safety Analysis Set | |
| Table 14.3.2.12 Summary of MedDRA SMQ for Torsade de Pointes by Pref Set: Safety Analysis Set | · |
| Table 14.3.3.1 Summary of Serious Treatment Emergent Adverse Events by Set: Safety Analysis Set | , |
| Table 14.3.3.2 Summary of Serious Treatment Emergent Adverse Events Re<br>Preferred Term Analysis Set: Safety Analysis Set | |
| Table 14.3.3.3 Summary of Serious Treatment Emergent Adverse Events by | Preferred Term Analysis Set: Safety Analysis Set 92 |
| Table 14.3.3.4 Summary of Serious Treatment Emergent Adverse Events Re Safety Analysis Set | |
| Table 14.3.3.5 Summary of Serious Treatment Emergent Adverse Events by CTCAE Grade Analysis Set: Safety Analysis Set | |
| Table 14.3.3.6 Summary of Serious Treatment Emergent Adverse Events Re<br>Term and Maximum CTCAE Grade Analysis Set: Safety Analysis Set | |
| Table 14.3.3.7 Summary of Treatment Emergent Adverse Events Leading to Analysis Set: Safety Analysis Set | |
| Table 14.3.3.8 Summary of Subject Death Analysis Set: Safety Analysis Set | et |
| Table 14.3.7.1 Summary of Hematology Laboratory by Visit Analysis Set: | Safety Analysis Set |

| Table 14.3.7.3 Summary of Coagulation Laboratory by Visit Analysis Set: Safety Analysis Set | <del>9</del> 7 |
|---|---|
| Table 14.3.7.5 Summary of Serum Chemistry Laboratory by Visit Analysis Set: Safety Analysis Set | 97 |
| Table 14.3.7.2.1 Shift of Hematology CTCAE Grade from Baseline to Worst Post-baseline Analysis Set: Safety Analysis Set 9 | 98 |
| Table 14.3.7.2.2 Summary of Hematology CTCAE On-Treatment Worsening Analysis Set: Safety Analysis Set | 99 |
| Table 14.3.7.4 Shift of Coagulation CTCAE Grade from Baseline to Worst Post-baseline Analysis Set: Safety Analysis Set 10 | 00 |
| Fable 14.3.7.6 Shift of Serum Chemistry CTCAE Grade from Baseline to Worst Post-baseline Analysis Set: Safety Analysis Set 10 | 00 |
| Γable 14.3.8.1 Summary of 12-lead ECGs by Visit Analysis Set: Safety Analysis Set | 01 |
| Table 14.3.8.2 Summary of QTcF/QTcB Interval Clinically Significant Analysis Set: Safety Analysis Set | 02 |
| Fable 14.3.10 Summary of ARV-471 and ARV-473 Plasma Concentration (unit) by Visit Analysis Set: Pharmacokinetic Analysis Set | |
| Figure 14.2.1.1 Spider Plot for Individual Ki-67 Value Analysis Set: Full Analysis Set | 04 |
| Figure 14.2.1.2.1 Box Plot for Ki-67 Percentage Change from Baseline at Cycle 1 Day 15 Analysis Set: Ki-67 Evaluable Set 10 | 05 |
| Figure 14.2.1.2.2 Box Plot for Ki-67 Percentage Change from Baseline at Surgery Analysis Set: Full Analysis Set | 06 |
| Figure 14.2.3.1 Waterfall Plot for Best Percentage Change of Primary Tumor from Baseline (Caliper-based) Analysis Set: Full Analysis Set | 0 <b>7</b> |
| Figure 14.2.3.2.1 Waterfall Plot for Best Percentage Change of Target Lesion from Baseline Analysis Set: Full Analysis Set 10 | 08 |
| Figure 14.2.3.2.2 Spider Plot for the Percent Target Lesion Size Change from Baseline by Subject and Timepoint Analysis Set: Fu Analysis Set | |
| Figure 14.2.4.1 Spider Plot for Individual ER AQUA Score Analysis Set: Full Analysis Set | 10 |
| Figure 14.2.4.2.1 Box Plot for ER AQUA Score Percentage Change from Baseline at Cycle 1 Day 15 Analysis Set: Full Analysis Set | |
| Figure 14.2.4.2.2 Box Plot for ER AQUA Score Percentage Change from Baseline at Surgery Analysis Set: Full Analysis Set 11 | 12 |
| Figure 14.2.5.1 Spider Plot for Individual PR H-score Analysis Set: Full Analysis Set | 13 |
| Figure 14.2.5.2.1 Box Plot for PR H-score Percentage Change from Baseline at Cycle 1 Day 15 Analysis Set: Full Analysis Set | |

| Figure 14.2.5.2.2 Box Plot for PR H-score Percentage Change from Baseline at Surgery Analysis Set: Full Analysis Set | 115 |
|---|---|
| Figure 14.3.2.8 Tornado Plot for Treatment Emergent Adverse Events by Preferred Term Analysis Set: Safety Analysis Set | 116 |
| Listing 16.2.1.1 Subject Enrollment Analysis Set: Full Analysis Set | 117 |
| Listing 16.2.1.2 Subject Disposition Analysis Set: Enrolled Participants | 118 |
| Listing 16.2.2 Deviations from the Clinical Protocol Analysis Set: Full Analysis Set | 119 |
| Listing 16.2.4.1 Demographic Characteristics Analysis Set: Full Analysis Set. | 120 |
| Listing 16.2.4.2 Medical History Analysis Set: Full Analysis Set | 121 |
| Listing 16.2.4.3 Disease Staging - Initial Diagnosis Analysis Set: Full Analysis Set. | 122 |
| Listing 16.2.4.4 Disease Staging - Current Diagnosis Analysis Set: Full Analysis Set | 123 |
| Listing 16.2.4.5 Molecular Biology of Disease Analysis Set: Full Analysis Set | 124 |
| Listing 16.2.4.6 Prior and Concomitant Medications Analysis Set: Full Analysis Set | 125 |
| Listing 16.2.5.1 Study Drug Exposure and Compliance Analysis Set: Safety Analysis Set. | 126 |
| Listing 16.2.5.2 Study Drug Administration Analysis Set: Safety Analysis Set | 127 |
| Listing 16.2.5.3 PK Dosing - ARV-471 Analysis Set: Safety Analysis Set. | 128 |
| Listing 16.2.5.4 ARV-471 and ARV-473 Plasma Concentration Analysis Set: PK Analysis Set | 129 |
| Listing 16.2.6.1 Efficacy Parameters – Part 1 of 2 Analysis Set: Full Analysis Set | 130 |
| Listing 16.2.6.2 Efficacy Parameters – Part 2 of 2 Analysis Set: Full Analysis Set | 131 |
| Listing 16.2.6.3 Target Lesion (TL) Analysis Set: Full Analysis Set. | 132 |
| Listing 16.2.6.4 Primary Breast Tumor Change - Caliper-based Analysis Set: Full Analysis Set | 133 |
| Listing 16.2.6.5 Tumor Biopsy Analysis Set: Full Analysis Set | 134 |
| Listing 16.2.6.6 Imaging Response Assessment - mRECIST Analysis Set: Full Analysis Set. | 135 |
| Listing 16.2.6.7 Cytology Results Analysis Set: Full Analysis Set. | 136 |
| Listing 16.2.6.8 Disease Staging - Post-Surgery Analysis Set: Full Analysis Set. | 137 |
| Listing 16.2.7.1 Adverse Events by Subject Analysis Set: Safety Analysis Set | 138 |
| Listing 16.2.7.2 Serious Adverse Events by Subject Analysis Set: Safety Analysis Set | 138 |

| Listing 16.2.8.1 Hematology Tests with CTCAE Grade ≥ 3 Analysis Set: Safety Analysis Set | 140 |
|---|---|
| Listing 16.2.8.2 Clinical Chemistry Tests with CTCAE Grade ≥ 3 Analysis Set: Safety Analysis Set | 140 |
| Listing 16.2.8.3 Hematology Tests Analysis Set: Safety Analysis Set | 14 |
| Listing 16.2.8.4 Clinical Chemistry Tests Analysis Set: Safety Analysis Set | 14 |
| Listing 16.2.8.5 Coagulation Tests Analysis Set: Safety Analysis Set. | 14 |
| Listing 16.2.8.6 Urinalysis Analysis Set: Safety Analysis Set | 142 |
| Listing 16.2.9 Vital Signs Analysis Set: Safety Analysis Set | 143 |
| Listing 16.2.10 12-Lead ECG Analysis Set: Safety Analysis Set | 144 |
| Listing 16.2.11 ECOG Performance Status Analysis Set: Safety Analysis Set. | 145 |

# **REVISIONS**

| Date | Brief Description |
|---|---|
| 10March2023 | First draft 0.1 |
| 17April2023 | Updates based on Arvinas comments |
| 24April2023 | Accept updates in Version 0.2 and correct some typo |
| 15Jan2024 | Add more TFL shells based on Arvinas comments on dryrun TFLs |
| 24May2024 | Add additional TFL shells based on Arvinas comments and new requests |
| 03June2024 | Accept the updates in version 0.4 |
| 24June2024 | Update Baseline definition |
| 02October2024 | Update based on Arvinas' comments on dryrun #2 draft |
| 11October2024 | Update based on Arvinas' replies on the Caidya's updates and meeting discussion on 08OCT2024: |
| | * Update the definition of subgroups – derivation will be based on EDC and lab data instead of IRT |
| | * Add summary for participants with Tumor Biopsies at each visit, medical history, absolute dose intensity, |
| | relative dose intensity, subgroup analysis for change of tumor size by baseline tumor size category |
| | * Add additional plots for KI-67 at surgery, ER AQUA Score, PR H-score |
| | * Update Concomitant Medications and TEAE definition |
| 14November2024 | * Accept changes in version 1.2 |
| | * Update based on Arvinas' comments on dryrun #2 Final: add Grade 3 or higher panel in Figure 14.3.2.8; |
| | update footnotes or contents text for more details; Renumbering the listings |
| 15November2024 | Accept Changes in version 1.2 |

## GLOBAL CONVENTIONS

# **Format and Ordering of Groups**

Columns in summary tables will be ordered as follow:

| ARV-471 200 mg | Anastrozole 1 mg | Total |
|----------------|------------------|-------|
| N=XX | N=XX | N=XXX |
| n (%) | n (%) | n (%) |

<sup>&</sup>quot;Total" column in some efficacy tables will be removed if it is not necessary.

# **General Display Conventions**

Summary tables and subject data listings will be in landscape format. Table titles will be centered.

# **Sorting Conventions**

For MH summaries, Primary System Organ Classes (SOCs) will be ordered descending count for All Subjects and Preferred Terms (PTs) will be ordered by descending count for All Subjects or alphabetically for PTs with the same count for All Subjects.

For AE summaries, Primary SOCs will be ordered descending count for All Subjects and PTs will be ordered by descending count for all subjects

# **Display of Continuous Statistics**

Means and medians will be shown to one more decimal place and the standard deviation will be shown to two more decimal that the source data values. In cases where variables are derived and have floating point values (no fixed number of decimal places), an appropriate level of precision will be determined based on the context.

Statistics that cannot be derived will be shown as a dash ( "-") in summary tables.

Two-Sided confidence intervals are displayed with a format such as "(xx.x, xx.x)." If a confidence interval cannot be produced due to insufficient data, then a dash ("-") will be shown in place of the entire confidence interval.

# **Display of Percentages**

The following conventions apply for percentages:

- Percentages will be displayed to one decimal place unless otherwise specified
- No percentage will be shown if the corresponding count is 0
- Percentages that are exactly equal to 100% will be displayed as "100%"
- Percentages that round down to 0.0% will be displayed as "<0.1%"
- Percentages that round up to 100.0% will be displayed as ">99.9%"

Percentages are shown in parentheses after the corresponding count such as "25 (5.2)" where extra spaces are included after the left parenthesis to ensure that decimal places for all percentages align within the same column.

# **Display of P-Values**

Unless otherwise noted, p-values will be displayed as follows:

- P-values between 0.0001 and 0.9999 will be displayed in the format "0.xxxx"
- P-values that are exactly equal to 1 will be displayed as "1.0000"
- P-values < 0.0001 will be displayed as "< 0.0001"
- P-values >0.9999 and not exactly equal to 1 will be displayed as ">0.9999"

P-values that are descriptive and not associated with a formal test of hypothesis will not be flagged based on statistical significance. The following note will be shown in the table:

```
Note: P-values are for descriptive purposes and are not evaluated for statistical significance.
```

Unless otherwise noted, p-values that are statistically significant will be flagged with an asterisk. The table footnote is dependent on the setting, but the following example footnote is appropriate for many settings:

```
* Statistically significant at the 0.05 level.
```

# **Display of Dates in Subject Data Listings**

Dates will be shown as follows:

- DDMMMYYYY for complete dates
- MMMYYYY for dates with only a month and year
- YYYY for dates with only a year

Partial dates are not imputed for subject data listings even if such dates are imputed for statistical algorithms. Relative day (if shown) is only derived for complete dates.

# **Display of Time in Subject Data Listings**

Time will be shown as follows:

- HH:MM for complete time
- HH for time with only hours

Partial time is not imputed for subject data listings.

# **Display of Missing Values in Subject Data Listings**

For subject data listings, missing numeric values will be shown as a dash ( "-"). Missing character values will be shown as blanks.

Table 14.1.1.1 Summary of Analysis Sets Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Analysis Set | n (%) | n (%) | n (%) |
| Full Analysis Set [1] | XXX (XX.X) | XX (XX.X) | XXX(XX.X) |
| Safety Analysis Set [2] | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Ki-67 Evaluable Set [3] | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Pharmacodynamic/Biomarker Analysis Set [4] | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| PK Concentration Analysis Set [5] | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |

- [1] Full Analysis Set is defined as all enrolled participants who were randomized.
- [2] Safety Analysis Set is defined as all enrolled participants who receive at least 1 dose of study intervention.
- [3] Ki-67 Evaluable Set is defined as all enrolled participants who were randomized and received at least one dose of study treatment and had evaluable Ki-67 measurements other than '0' or '< 1' from baseline and evaluable Ki-67 measurements from C1D15 visits.
- [4] Pharmacodynamic/Biomarker Analysis Set is defined as all enrolled participants with at least 1 of the Pharmacodynamic/Biomarkers evaluated at pre and/or post dose.
- [5] PK Concentration Analysis Set includes all participants in the Safety Analysis Set who have at least one plasma concentration (including those below the limit of quantification) for ARV-471, or ARV-473.

Source: Listing 16.2.1.1.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY. (add this footnote in all TFLs)

Table 14.1.1.2 Summary of Participants with Tumor Biospsy Analysis Set: Full Analysis Set

Test: Ki-67

| | ARV-471 | Anastrozole | Total |
|------------------------|--------------|-------------|------------|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| At Screen, N' | XXX | XXX | XXX |
| With result, n (%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Uninterpretable, n (%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| At Cycle 1 Day 15, N' | XXX | XXX | XXX |
| With result, n (%) | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Uninterpretable, n (%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| At Cycle 6 Day 18, N' | XXX | XXX | XXX |
| With result, n (%) | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Uninterpretable, n (%) | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| At Unscheduled, N' | XXX | XXX | XXX |
| With result, n (%) | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Uninterpretable, n (%) | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |

Note: N' is the number of participants at the visit. It is the denominator of the visit.

Source: Listing 16.2.6.5.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY. (add this footnote in all TFLs)

## Programming Note:

Repeat the table for each test on a new page. "Test: Progesterone Receptor"

Table 14.1.2.1
Summary of Disposition and Discontinuation
Analysis Set: Enrolled Participants

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Total<br>N=XXX |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| Number of Enrolled Participants, N' | | | XXX |
| Number of Screen Failures, N' | | | XX |
| Number of Eligible Participants not Randomized, N' | | | XX |
| Number of Participants Randomized (Full Analysis Set), N | XXX | XX | XXX |
| Never Dosed | X(XX.X) | X(XX.X) | X(XX.X) |
| Completed Treatment per Protocol | XXX(XX.X) | XX (XX.X) | XXX (XX.X) |
| ARV-471/Anastrozole Early Discontinuation | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Reason for ARV-471/Anastrozole Early Discontinuation | | | |
| Disease Progression per Response Criteria | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Clinical Progression | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Withdrawal of Consent | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Significant non-compliance | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Pregnancy | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Death | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Adverse Event | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Study Terminated by Sponsor | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Lost to Follow-up | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Completed Study per Protocol | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Study Early Discontinuation | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Reason for Study Early Discontinuation | | | |
| Withdrawal of Consent | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Study Terminated by Sponsor | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Lost to Follow-up | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Death | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

Note: Enrolled Participants included all subjects who signed the Informed Consent.

Note: Column N and percentage are based on the number of subjects in Full Analysis Set.

Source: Listing 16.2.1.2.

## Repeat the following table with Table 14.1.2.1 shell

Table 14.1.2.2 Summary of Disposition and Discontinuation Analysis Set: Ki-67 Evaluable Set

Table 14.1.3 Summary of Protocol Deviation Analysis Set: Full Analysis Set

| | ARV-471<br>200 mg N=XX<br>n (%) | Anastrozole<br>1 mg N=XX<br>n (%) | Total<br>N=XXX |
|---|---|---|---|
| | | | n (%) |
| Number of Subjects with Any Protocol | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Deviation | | | |
| Informed Consent | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| IMP/NIMP | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Protocol Compliance | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Safety | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ICH/GCP | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| <insert></insert> | | | |
| Number of Subjects with Major or | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Critical Protocol Deviation | | | |
| Informed Consent | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| IMP/NIMP | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Protocol Compliance | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Safety | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ICH/GCP | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| <insert></insert> | | | |
| Number of Subjects with Minor Protocol | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Deviation | | | |
| Informed Consent | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| IMP/NIMP | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Protocol Compliance | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Safety | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| ICH/GCP | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| <insert></insert> | | | |

Source: Listing 16.2.2.

Table 14.1.4.1 Summary of Demographic Characteristics Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Sex, n(%) | | | |
| Female | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| remate | AAA (AA•A) | AA (AA.A) | ۸۸۸ (۸۸۰۸) |
| Age (years) | | | |
| n | XXX | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Age Group, n(%) | | | |
| ≥ 60 Years | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| < 60 Years | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| V 00 IGGIS | 71111 (1111 • 11) | 2121 (2121 + 21) | 212221 (2121 * 21) |
| Race [1], n(%) | | | |
| American Indian or Alaskan Native | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Asian | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Black or African American | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Native Hawaiian/Other Pacific Islander | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| White | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Unknown | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Ethnicity, n(%) | | | |
| Hispanic or Latino | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Not Hispanic or Latino | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Not Reported | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Weight (kg) at Baseline | | | |
| n | XXX | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX • X | XX.X | XX • X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Height (cm) at Baseline | | | |
| n | xxx | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | xx.x(xx.xx)<br>xx.x | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX) |
| Min, Max | | | |
| riii, rida | XX, XX | xx, xx | XX, XX |

| 0 | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
|---|---|---|---|
| 1 | XXX (XX.X) | XX (XX.X) | XXX (XX.X |
| ize of Primary Breast Tumor (T-stage), n(%) | | | |
| ≤ 2 cm | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| >2 to < 5 cm | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| ≥ 5 cm | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| ost-menopausal Reason, n(%) | | | |
| Prior bilateral oophorectomy | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Age >= 60 years | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Age < 60 years and amenorrhoeic for at least 12 months | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |

<sup>[1]</sup> Multiple race might be reported.

Source: Listing 16.2.4.1.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY.

## Repeat the following table with Table 14.1.4.1 shell

Table 14.1.4.2 Summary of Demographic Characteristics Analysis Set: Ki-67 Evaluable Set

Table 14.1.5

Summary of Medical History by System Organ Class and Preferred Term
Analysis Set: Full Analysis Set

| System Organ Class | ARV-471 | Anastrozole | Total |
|-------------------------------------|--------------|-------------|-----------|
| Preferred Term | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Patients with Medical History, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | | | |
| Preferred Term #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <insert></insert> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre><insert></insert></pre> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Medical history was coded with MedDRA version 27.0.

Note: Subjects are counted once per Preferred Term and once per System Organ Class.

Sources: Listing 16.2.4.2.

Table 14.1.6.1
Summary of Disease Staging and Disease Characteristics
Analysis Set: Full Analysis Set

| | ARV-471 | | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Time since Initial Diagnosis (months) | | | |
| n | xxx | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Time since Current Staging (months) | | | |
| n | xxx | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX • X | XX • X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Primary Diagnosis: ER+ HER2- Breast Cancer, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Disease Stage at Initial Diagnosis, n(%) | | | |
| Stage 0 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IA | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Stage IB | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Stage IIA | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIB | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIIA | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIIB | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIIC | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IV | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Unknown | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Disease Stage at Screening, n(%) | | | |
| Stage 0 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IA | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IB | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIA | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIB | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIIA | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIIB | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IIIC | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Stage IV | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Unknown | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

| Primary Tumor at Initial Diagnosis, n(%) | | | |
|---|---|---|---|
| TX | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| TO | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Tis | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T1mi | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Tla | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T1b | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Tlc | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T3 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T4a | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T4b | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T4c | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Primary Tumor at Screening, n(%) | | | |
| TX | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| TO | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Tis | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T1mi | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Tla | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T1b | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Tlc | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T3 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| T4a | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| T4b | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| T4c | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Imaging Modality for Primary Tumor at Screening, n(%) | | | |
| CT | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| MRI | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Ultrasound | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Mammogram | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Regional Lymph Node at Initial Diagnosis, n(%) | | | |
| CNX | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| cN0 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| cN1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| cN2a | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| cN2b | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| cN3a | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| cN3b | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| cN3c | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

| Regional Lymph Node at Screening, n(%) | | | |
|---|---|---|---|
| cNX | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| cN0 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| cN1 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| cN2a | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| cN2b | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| cN3a | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| cN3b | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| cN3c | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Distant Metastasis at Initial Diagnosis, n(%) | | | |
| MO | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| M1 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Unknown | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Distant Metastasis at Screening, n(%) | | | |
| MO | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| M1 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Unknown | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Olikilowii | AAA (AA•A) | AA (AA•A) | AAA (AA•A) |
| Histopathological Classification at Initial Diagnosis, n(%) | | | |
| In-Situ Carcinoma | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Invasive Ductal Carcinoma | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Invasive Lobular Carcinoma | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Invasive Mixed Ductal and Lobular Breast Carcinoma | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Invasive Carcinoma NOS | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Invasive Adenocarcinoma NOS | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Tubular Carcinoma | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Invasive Mucinous Adenocarcinoma | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Histopathological Classification at Screening, n(%) | | | |
| In-Situ Carcinoma | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Invasive Ductal Carcinoma | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Invasive Lobular Carcinoma | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Invasive Mixed Ductal and Lobular Breast Carcinoma | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Invasive Carcinoma NOS | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Invasive Adenocarcinoma NOS | XXX (XX.X) | XX (XX.X) | XXX(XX.X) |
| Tubular Carcinoma | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Invasive Mucinous Adenocarcinoma | XXX (XX.X) | XX (XX.X) | XXX(XX.X) |
| Other | XXX (XX.X) | XX (XX.X) | XXX(XX.X) |

| Grade 1 | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
|---|---|---|---|
| Grade 2 | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
| Grade 3 | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
| Grade X | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
| Histopathological Grade at Screening, n(%) | | | |
| Grade 1 | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
| Grade 2 | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
| Grade 3 | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
| Grade X | XXX(XX.X) | XX(XX.X) | XXX (XX.X |
| Planned Type of Breast Surgery, n(%) | | | |
| Planned Type of Breast Surgery, n(%) Breast conserving surgery | XXX (XX.X) | XX(XX.X) | XXX(XX.X |

Note: Time since initial diagnosis (months) is defined as time from the date of initial diagnosis to the date of first ARV-471/anastrozole dose. Time since current staging (months) is defined as time from the date of current staging to the date of first ARV-471/anastrozole dose.

Source: Listing 16.2.4.3 and Listing 16.2.4.4.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY.

## Programming Note:

#### Repeat the following table with Table 14.1.6.1 shell

Table 14.1.6.2 Summary of Disease Staging and Disease Characteristics Analysis Set: Ki-67 Evaluable Set

Table 14.1.7.1
Summary of Disease Molecular Biology at Baseline
Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| HER2 Status, Performed, n(%) | | | |
| Yes | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| No | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Sample Site of HER2 Status, n(%) | | | |
| Breast | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Lymph Node | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| HER2 Analytical Method, n(%) | | | |
| Immunohistochemistry (IHC) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| In Situ Hybridization (ISH) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| HER2 Analytical Result, n(%) | | | |
| 0 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 1+ | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 2+ | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 3+ | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Positive | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Negative | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Unknown | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Ki67, Performed, n(%) | | | |
| Yes | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| No | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Sample Site of Ki67, n(%) | | | |
| Breast | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Lymph Node | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| d of Tumor Cells with Ki67 (Local) | | | |
| n | XXX | XX | Xx |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

| \$ 20\$, n(\$) | < 20%, n(%) | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
|---|---|---|---|---|
| n xxx xx | ≥ 20%, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Mean (Standard Deviation) xx.x(xx.xx) xx.x xx.x(xx.xx) xx.x xx.x xx xx.x xx.x xx.x | % of Tumor Cells with Ki67 (Central) | | | |
| Median Max xx.x xx | n | XXX | xx | Xx |
| Min, Max xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) <t< td=""><td>Mean (Standard Deviation)</td><td>xx.x(xx.xx)</td><td>xx.x(xx.xx)</td><td>xx.x(xx.xx)</td></t<> | Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| < 20%, n(%) | Median | XX.X | XX.X | XX.X |
| ≥ 20%, n(%) XXX(XX.X) XXX(XX.X) XXX(XX.X) Estrogen Receptor, Performed, n(%) XXX(XX.X) XXX(XX.X) XXX(XX.X) Sample Site of Estrogen Receptor, n(%) XXX(XX.X) XXX(XX.X) XXX(XX.X) Breast XXX(XX.X) XXX(XX.X) XXX(XX.X) Lymph Node XXX(XX.X) XX(XX.X) XXX(XX.X) Other XXX(XX.X) XX(XX.X) XXX(XX.X) % of Tumor Cells with Estrogen Receptor (Local) XXX XX XX n XXX XX XX.X(XX.X) XX.X(XX.XX) XX.X(XX.XX) Median XXX.X XX.X XXX.X | Min, Max | xx, xx | XX, XX | XX, XX |
| Estrogen Receptor, Performed, n(%) Yes No XXX (XX.X) Sample Site of Estrogen Receptor, n(%) Breast XXX (XX.X) XXX (XX. | < 20%, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Yes XXX (XX.X) XX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) <td>≥ 20%, n(%)</td> <td>XXX (XX.X)</td> <td>XX(XX.X)</td> <td>XXX(XX.X)</td> | ≥ 20%, n(%) | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| No XXX (XX.X) XX (XX.X) XXX (XX.XX) XXX (XX.XX) | Estrogen Receptor, Performed, n(%) | | | |
| Sample Site of Estrogen Receptor, n(%) XXX (XX.X) XXX (XX.XX) XXX | Yes | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ## Breast | No | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| ## Breast | Sample Site of Estrogen Receptor, n(%) | | | |
| other XXX (XX.X) XXX (XX.X) XXX (XX.X) % of Tumor Cells with Estrogen Receptor (Local) xxx xxx xx Xx n xxx xx.x (xx.xx) xx.x (xx.xx | | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| <pre>% of Tumor Cells with Estrogen Receptor (Local)</pre> | Lymph Node | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| n xxx xx Xx Mean (Standard Deviation) xx.x(xx.xx) xx.x(xx.xx) xx.x(xx.xx) Median xx.x xx.x xx.x xx.x Min, Max xx < | Other | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Mean (Standard Deviation) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) xx.x x xx.x x xx.x x xx.x x xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx xx.x xx </td <td>% of Tumor Cells with Estrogen Receptor (Local)</td> <td></td> <td></td> <td></td> | % of Tumor Cells with Estrogen Receptor (Local) | | | |
| Median Max xx.x xx xx, xx xx.x xx, xx xxx xx, xx< | n | XXX | xx | Xx |
| Min, Max xx, xx xx, xx xx, xx xx, xx < 10%, n(%) | | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| <pre></pre> | Median | XX.X | XX.X | XX.X |
| ≥ 10%, n(%) Progesterone Receptor, Performed , n(%) Yes | Min, Max | xx, xx | XX, XX | XX, XX |
| Progesterone Receptor, Performed , n(%) XXX (XX.X) XX (XX.X) XXX (XX | < 10%, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Yes XXX (XX.X) XX (XX.X) XXX (XX.X) No XXX (XX.X) XX (XX.X) XXX (XX.X) Sample Site of Progesterone Receptor, n(%) XXX (XX.X) XX (XX.X) XXX (XX.X) Breast XXX (XX.X) XX (XX.X) XXX (XX.X) Lymph Node XXX (XX.X) XX (XX.X) XXX (XX.X) | ≥ 10%, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| No XXX (XX.X) XX (XX.X) XXX (XX.X) Sample Site of Progesterone Receptor, n(%) XXX (XX.X) XX (XX.X) XXX (XX.X) Breast XXX (XX.X) XX (XX.X) XXX (XX.X) Lymph Node XXX (XX.X) XX (XX.X) XXX (XX.X) | Progesterone Receptor, Performed , n(%) | | | |
| Sample Site of Progesterone Receptor, n(%) Breast XXX(XX.X) XX(XX.X) XXX(XX.X) Lymph Node XXX(XX.X) XX(XX.X) | Yes | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Breast XXX (XX.X) XX (XX.X) XXX (XX.X) Lymph Node XXX (XX.X) XX (XX.X) XXX (XX.X) | No | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Breast XXX (XX.X) XX (XX.X) XXX (XX.X) Lymph Node XXX (XX.X) XX (XX.X) XXX (XX.X) | Sample Site of Progesterone Receptor, n(%) | | | |
| | | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Other XXX(XX.X) XX(XX.X) XXX(XX.X) | Lymph Node | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| | Other | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

| n | XXX | XX | Xx |
|---------------------------|-------------|-------------|------------|
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| < 1%, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ≥ 1%, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

Note: All the data are from local laboratories unless otherwise indicated.

Source: Listing 16.2.4.5.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY.

## Programming Note:

Repeat the following table with Table 14.1.7.1 shell

Table 14.1.7.2

Summary of Disease Molecular Biology at Baseline
Analysis Set: Ki-67 Evaluable Set

Table 14.1.8

Summary of Prior Cancer Related Surgery/Biopsy
Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Any Prior Surgery/Biopsy Related to Trial Disease[1], n(%) | | | |
| Yes | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| 100 | 717171 (7171 • 71) | 7171 (7171 • 71) | 212121 (2121 • 21) |
| Procedure[1], n(%) | | | |
| Sentinel node biopsy | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Axillary sampling | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Fine needle aspiration, | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Core needle biopsy | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Procedure Location[1], n(%) | | | |
| Breast | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Lymph node | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Laterality[1], n(%) | | | |
| Left | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Right | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Bilateral | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Not applicable | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Time since Most Recent Surgery/Biopsy (months) | | | |
| n | xxx | XX | Xxx |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |

Note: Time since most recent surgery/biopsy is defined as time from the most recent date of surgery to the date of first ARV-471/Anastrozole dose.

<sup>[1]</sup> A subject might receive multiple Surgery/Biopsy.

Table 14.1.9
Summary of Prior Medication Analysis Set: Full Analysis Set

| ATC level 2 Preferred Name | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Total<br>N=XXX |
|---|---|---|---|
| Subjects with Any Prior Medication, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ATC level 2 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 2 | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| ATC level 2 2 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

Note: Prior medications are coded according to the World Health Organization drug dictionary (WHO-Drug B3 Global version September 2024).

Note: Prior medications include non-study drug medications that are ended before Day 1.

Source: Listing 16.2.4.6.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY.

Table 14.1.10 Summary of Concomitant Medication Analysis Set: Full Analysis Set

| ATC level 2 Preferred Name | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Total<br>N=XXX |
|---|---|---|---|
| Subjects with Any Concomitant Medication, n(%) | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| ATC level 2 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ATC level 2 2 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Name 2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

Note: Prior medications are coded according to the World Health Organization drug dictionary (WHO-Drug B3 Global version September 2024).

Note: Concomitant medications include non-study drug medications that are used/started on/after Day 1 and within 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Source: Listing 16.2.4.6.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY.

Table 14.1.11
Summary of ARV-471 and Anastrozole Compliance and Exposure
Analysis Set: Safety Analysis Set

| | ARV-471 | Anastrozole |
|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX |
| Duration of Treatment (week) | | |
| n | XXX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX • X |
| Min, Max | xx, xx | XX, XX |
| Cumulative Dose (mg) | | |
| n | XXX | XX |
| Mean (Standard Deviation) | XX.X(XX.XX) | xx.x(xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| Absolute Dose Intensity (mg/week) | | |
| n | XXX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX |
| Total Planned Dose (mg) | | |
| n | XXX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX |
| Compliance (%) | | |
| n | XXX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| <pre>Jumber (%) of Compliant Patients, n(%)</pre> | XXX (XX.X) | XX(XX.X) |
| Relative Dose Intensity (%) | | |
| n | XXX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx |

| Number of Subjects with at Least One Action Taken, n(%) | XXX (XX.X) | XX (XX.X) |
|---|---|---|
| Dose Interrupted | XXX(XX.X) | XX(XX.X) |
| Dose Discontinued | XXX(XX.X) | XX(XX.X) |
| Dose Reduced | XXX(XX.X) | XX(XX.X) |
| Dose Increased | XXX (XX.X) | XX(XX.X) |
| Reason for Dose Interrupted[1], n(%) | | |
| Adverse event | XXX (XX.X) | XX(XX.X) |
| Participant missed/Skipped dose | XXX(XX.X) | XX(XX.X) |
| Medication error | XXX(XX.X) | XX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) |
| Reason for Dose Reduced[1], n(%) | | |
| Adverse event | XXX(XX.X) | XX(XX.X) |
| Participant missed/Skipped dose | XXX (XX.X) | XX(XX.X) |
| Medication error | XXX (XX.X) | XX(XX.X) |
| Other | XXX(XX.X) | XX(XX.X) |
| Reason for Dose Discontinued[1], n(%) | | |
| Adverse event | XXX(XX.X) | XX(XX.X) |
| Participant missed/Skipped dose | XXX (XX.X) | XX (XX.X) |
| Medication error | XXX (XX.X) | XX(XX.X) |
| Other | XXX (XX.X) | XX (XX.X) |
| Reason for Dose Increased[1], n(%) | | |
| Adverse event | XXX (XX.X) | XX(XX.X) |
| Participant missed/Skipped dose | XXX (XX.X) | XX (XX.X) |
| Medication error | XXX (XX.X) | XX (XX.X) |
| 110410401011 01101 | 171717 / 1777 • 17 / | 2227 / 2222 • 22 / |

<sup>[1]</sup> Multiple reasons might be reported.

Note: Compliance is 100\* (Total cumulative dose/Total planned dose), accounting for planned dose modifications and interruptions. Compliant Patients are those with compliance >= 80% - <= 120%. Absolute Dose Intensity (mg/week) is (Cumulative Dose (mg))/(Duration of Treatment (week)). Relative Dose Intesity (%) is 100\* (Absolute Dose Intensity (mg/week))/(Initial Planned Weekly Dose (mg/week), 1400 mg/week for ARV-471 and 7 mg/week for Anastrozole)). Source: Listing 16.2.5.1, and Listing 16.2.5.2.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY.

Table 14.2.1.1.1

Summary of Ki-67 Percentage Change from Baseline at C1D15 with Central Ki-67 as a Covariate
Analysis Set: Ki-67 Evaluable Set

| | ARV-471<br>200 mg N=XXX | Anastrozole | Difference |
|---|---|---|---|
| | | 1 mg N=XX | |
| log(Ki-67 at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) - log(Ki-67 at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | xx.x | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between Ki-67 at C1D15 and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at C1D15}) - \log(Ki-67 \text{ at baseline}))$ .

Source: Listing 16.2.6.1.

<sup>[1]</sup> Analysis based on an analysis of covariance (ANCOVA) model with baseline Ki-67 score (assessed **centrally**: <20% vs  $\geq$ 20%), the tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm) as covariates for treatment. Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

<sup>[2]</sup> Back transformed values of [1].

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Difference |
|---|---|---|---|
| log(Ki-67 at baseline) | | | |
| n | xxx | xx | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | xx.x | xx.x | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) | | | |
| n | xxx | xx | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) - log(Ki-67 at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between Ki-67 at C1D15 and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | xx.xx, xx.xx |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at C1D15}) - \log(Ki-67 \text{ at baseline}))$ .

Source: Listing 16.2.6.1.

<sup>[1]</sup> Analysis based on an analysis of covariance (ANCOVA) model with baseline Ki-67 score (assessed **locally**: <20% vs  $\geq$ 20%), the tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm) as covariates for treatment. Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

<sup>[2]</sup> Back transformed values of [1].

Table 14.2.1.1.3

Summary of Ki-67 Percentage Change from Baseline at C1D15 without Covariate
Analysis Set: Ki-67 Evaluable Set

| | ARV-471<br>200 mg N=XXX | Anastrozole | |
|---|---|---|---|
| | | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) - log(Ki-67 at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between Ki-67 at C1D15 and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at C1D15}) - \log(Ki-67 \text{ at baseline}))$ .

Source: Listing 16.2.6.1.

<sup>[1]</sup> Analysis based on an analysis of variance (ANOVA) model.

<sup>[2]</sup> Back transformed values of [1].

 ${\it Table 14.2.1.2.1} \\ {\it Summary of Ki-67 Percentage Change from Baseline at C1D15- Subgroup Analysis by Tumor Size } \\ {\it Analysis Set: Ki-67 Evaluable Set}$ 

Tumor Size: ≤2 cm

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) | | | |
| n | xxx | xx | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | XX.XX, XX.XX | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between Ki-67 at C1D15 and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at C1D15}) - \log(Ki-67 \text{ at baseline}))$ .

Note: Baseline tumor size categories are derived based on data collected instead of data reported in IRT.

- [1] Analysis based on an analysis of variance (ANOVA) model.
- [2] Back transformed values of [1].

Source: Listing 16.2.6.1.

Repeat the table for 'Tumor Size: >2 to <5 cm', and 'Tumor Size: ≥5 cm' on new page.

Table 14.2.1.2.2

Summary of Ki-67 Percentage Change from Baseline at C1D15 - Subgroup Analysis by Local Ki-67 Baseline Score
Analysis Set: Ki-67 Evaluable Set

Local Ki-67 Baseline Score: < 20%

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) | | | |
| n | xxx | xx | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | XX.XX, XX.XX | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between Ki-67 at C1D15 and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at C1D15}) - \log(Ki-67 \text{ at baseline}))$ .

Note: Baseline Ki-67 score are derived based on data collected instead of data reported in IRT.

- [1] Analysis based on an analysis of variance (ANOVA) model.
- [2] Back transformed values of [1].

Source: Listing 16.2.6.1.

### Repeat the table for 'Local Ki-67 Baseline Score: ≥ 20%" on new page.

Table 14.2.1.2.3

Summary of Ki-67 Percentage Change from Baseline at C1D15- Subgroup Analysis by Central Ki-67 Baseline Score of 20% Analysis Set: Ki-67 Evaluable Set

Central Ki-67 Baseline Score: < 20%

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between Ki-67 at C1D15 and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | xx.xx, xx.xx |
| 95% Confidence Interval for Geometric Means Difference[2] | | | xx.xx, xx.xx |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\exp(\log(\text{Ki-67 at C1D15}) - \log(\text{Ki-67 at baseline}))$ .

Note: Baseline Ki-67 score are derived based on data collected instead of data reported in IRT.[1] Analysis based on an analysis of variance (ANOVA) model.

[2] Back transformed values of [1].

Source: Listing 16.2.6.1.
# Programming Note:

Repeat the table for 'Central Ki-67 Baseline Score:  $\geq 20\%$ '' on new page.

Table 14.2.1.2.4

Summary of Ki-67 Percentage Change from Baseline at C1D15 - Subgroup Analysis by Central Ki-67 Baseline Score of 5% Analysis Set: Ki-67 Evaluable Set

Central Ki-67 Baseline Score: < 5%

| | ARV-471 | Anastrozole | · |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at C1D15) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between Ki-67 at C1D15 and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at C1D15}) - \log(Ki-67 \text{ at baseline}))$ .

Note: Baseline Ki-67 score are derived based on data collected instead of data reported in IRT.

- [1] Analysis based on an analysis of variance (ANOVA) model.
- [2] Back transformed values of [1].

Source: Listing 16.2.6.1.

## Programming Note:

Repeat the table for 'Central Ki-67 Baseline Score: ≥ 5%" on new page.

Table 14.2.1.3.1

Summary of Ki-67 Percentage Change from Baseline at Surgery with Central Ki-67 as a Covariate Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | xx.x | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) - log(Ki-67 at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between Ki-67 at Surgery and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from Surgery visit and baseline, which will be derived as =  $\exp(\log(\text{Ki}-67 \text{ at Surgery}) - \log(\text{Ki}-67 \text{ at baseline}))$ .

<sup>[1]</sup> Analysis based on an analysis of covariance (ANCOVA) model with baseline Ki-67 score (assessed **centrally**: <20% vs  $\geq$ 20%), the tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm) as covariates for treatment. Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

<sup>[2]</sup> Back transformed values of [1].

## Programming Note:

Table 14.2.1.3.2

Summary of Ki-67 Percentage Change from Baseline at Surgery with Local Ki-67 as a Covariate Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | xx, xx | |
| log(Ki-67 at Surgery) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| log(Ki-67 at Surgery) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between Ki-67 at Surgery and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from Surgery visit and baseline, which will be derived as =  $\exp(\log(\text{Ki-67 at Surgery}) - \log(\text{Ki-67 at baseline}))$ .

<sup>[1]</sup> Analysis based on an analysis of covariance (ANCOVA) model with baseline Ki-67 score (assessed **locally**: <20% vs  $\geq$ 20%), the tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm) as covariates for treatment. Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

<sup>[2]</sup> Back transformed values of [1].

## Programming Note:

Table 14.2.1.3.3

Summary of Ki-67 Percentage Change from Baseline at Surgery without Covariate

Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | XX.XX, XX.XX | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between Ki-67 at Surgery and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from Surgery visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at Surgery}) - \log(Ki-67 \text{ at baseline}))$ .

<sup>[1]</sup> Analysis based on an analysis of variance (ANOVA) model.

<sup>[2]</sup> Back transformed values of [1].

Source: Listing 16.2.6.1.

Table 14.2.1.4.1

Summary of Ki-67 Percentage Change from Baseline at Surgery - Subgroup Analysis by Tumor Size

Analysis Set: Full Analysis Set

Tumor Size: ≤2 cm

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery | | | |
| n) | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between Ki-67 at Surgery and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from Surgery visit and baseline, which will be derived as =  $\exp(\log(Ki-67 \text{ at Surgery}) - \log(Ki-67 \text{ at baseline}))$ .

Note: Baseline tumor size categories are derived based on data collected instead of data reported in IRT.

- [1] Analysis based on an analysis of variance (ANOVA) model.
- [2] Back transformed values of [1].

Source: Listing 16.2.6.1.

## Programming Note:

Repeat the table for 'Tumor Size: >2 to <5 cm', and 'Tumor Size: ≥5 cm' on new page.

Table 14.2.1.4.2

Summary of Ki-67 Percentage Change from Baseline at Surgery - Subgroup Analysis by Local Ki-67 Baseline Score
Analysis Set: Full Analysis Set

Local Ki-67 Baseline Score: < 20%

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| log(Ki-67 at Surgery | | | |
| n) | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | XX.XX, XX.XX | |
| 95% Confidence Interval for LSM[1] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between Ki-67 at Surgery and Ki-67 at baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 95% Confidence Interval for Geometric Means[2] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.X |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from Surgery visit and baseline, which will be derived as =  $\exp(\log(\text{Ki}-67 \text{ at Surgery}) - \log(\text{Ki}-67 \text{ at baseline}))$ .

Note: Baseline Ki-67 score are derived based on data collected instead of data reported in IRT.

- [1] Analysis based on an analysis of variance (ANOVA) model.
- [2] Back transformed values of [1].

Source: Listing 16.2.6.1.

## Programming Note:

Repeat the table for 'Local Ki-67 Baseline Score: ≥ 20%" on new page.

Table 14.2.1.4.3

Summary of Ki-67 Percentage Change from Baseline at Surgery - Subgroup Analysis by Central Ki-67 Baseline Score
Analysis Set: Full Analysis Set

Central Ki-67 Baseline Score: < 20%

| | ARV-471 | Anastrozole | <u> </u> |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(Ki-67 at Surgery) - log(Ki-67 at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between Ki-67 at Surgery and Ki-67 at baseline | | | |
| Geometric Means[2] | xx.x | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: The endpoint is the ratio between the Ki-67 measurements obtained from Surgery visit and baseline, which will be derived as =  $\exp(\log(\text{Ki}-67 \text{ at Surgery}) - \log(\text{Ki}-67 \text{ at baseline}))$ .

Note: Baseline Ki-67 score are derived based on data collected instead of data reported in IRT.

- [1] Analysis based on an analysis of variance (ANOVA) model.
- [2] Back transformed values of [1].

Source: Listing 16.2.6.1.

## Programming Note:

Repeat the table for 'Central Ki-67 Baseline Score: ≥ 20%" on new page.

Table 14.2.1.5.1
Summary of Concordance Ki-67 Baseline Score between Central and Local Laboratories
Analysis Set: Ki-67 Evaluable Set

| | Local Ki-67 Baseline | Local Ki-67 Baseline | |
|---|---|---|---|
| | Score <20% | Score ≥20% | Total |
| ARV-471 200 mg (N=XXX), n(%) | | | |
| Central Ki-67 Baseline Score <20% | XXX(XX.X) | XXX (XX.X) | XXX(XX.X) |
| Central Ki-67 Baseline Score ≥20% | XXX(XX.X) | XXX (XX.X) | XXX(XX.X) |
| Total | XXX (XX.X) | XXX(XX.X) | XXX(XX.X) |
| Anastrozole 1 mg (N=XX), n(%) | | | |
| Central Ki-67 Baseline Score <20% | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Central Ki-67 Baseline Score ≥20% | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Total | XX(XX.X) | XX(XX.X) | XX(XX.X) |

Note: The percentage is based on N.

Table 14.2.1.5.2

Summary of Concordance Central/Local Ki-67 Baseline Score with Randomization Baseline Ki-67 Score

Analysis Set: Ki-67 Evaluable Set

| Randomization Baseline<br>Ki-67 Score <20% | Randomization Baseline<br>Ki-67 Score ≥20% | Total |
|---|---|---|
| XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| XXX (XX.X) | XXX(XX.X) | XXX(XX.X) |
| XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XX(XX.X) | XX(XX.X) | XX(XX.X) |
| XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XX (XX.X) | Ki-67 Score <20% Ki-67 Score ≥20% XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XXX (XX.X) XX (XX.X) XX (XX.X) |

Note: The percentage is based on N.

Table 14.2.1.5.3

Summary of Concordance Acutal Primary Breast Tumor Size with Randomization Primary Breast Tumor Size

Analysis Set: Ki-67 Evaluable Set

| | Randomization Primary Breast Tumor Size <=2 cm | Randomization Primary Breast Tumor Size >2-<5 cm | Randomization Primary Breast Tumor Size >2-<5 cm | Total |
|---|---|---|---|---|
| ARV-471200 mg (N=XXX), n(%) | | | | |
| Acutal Primary Breast Tumor Size <=2 cm | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| Acutal Primary Breast Tumor Size >2-<5 cm | XXX (XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| Acutal Primary Breast Tumor Size >2-<5 cm | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| Total | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| ARV-471200 mg (N=XXX), n(%) | | | | |
| Acutal Primary Breast Tumor Size <=2 cm | XXX (XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| Acutal Primary Breast Tumor Size >2-<5 cm | XXX (XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| Acutal Primary Breast Tumor Size >2-<5 cm | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |
| Total | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) | XXX(XX.X) |

Note: The percentage is based on N.

Table 14.2.2.1.1

Summary of Post-Surgery Pathological Response and pCR Rate - Determined by Site Pathologist
Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | D: 66 |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| Participants Not Receiving Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| Participants Receiving Unscheduled Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| Post-Surgery Pathological Response in Participants | | | |
| Receiving Surgery at C6D18, n(%) | | | |
| Pathological Complete Response (pCR) | XXX(XX.X) | XX(XX.X) | |
| Pathological Partial Response (pPR) | XXX(XX.X) | XX(XX.X) | |
| No Response (NR) | XXX(XX.X) | XX(XX.X) | |
| pCR Rate in Participants Receiving Surgery at C6D18, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |

Note: pCR rate is the proportion of participants with pCR.

Table 14.2.2.1.2

Summary of Post-Surgery Pathological Response and pCR Rate - Calculated Analysis Set: Full Analysis Set

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Difference |
|---|---|---|---|
| Participants Not Receiving Surgery, n(%) | XXX (XX.X) | XX(XX.X) | |
| Participants Receiving Unscheduled Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| Post-Surgery Pathological Response in Participants Receiving Surgery at C6D18, $n(%)$ | | | |
| Calculated Pathological Complete Response (pCR) | XXX(XX.X) | XX(XX.X) | |
| Non pCR | XXX(XX.X) | XX(XX.X) | |
| pCR Rate in Participants Receiving Surgery at C6D18, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |

Note: pCR is programmatically derived according to the definition in the protocol using Disease Staging - Post-Surgery data: pCR is defined as no invasive cancer in the breast and sampled axillary lymph nodes following completion of neoadjuvant systemic therapy (Pathologic Tumor - ypT = ypT0 or ypTis, and Pathologic Lymph Nodes - ypN = ypN0).pCR rate is the proportion of participants with pCR.

Source: Listing 16.2.6.2.

Table 14.2.2.1.3.1
Summary of Post-Surgery Disease Staging
Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Participants Not Receiving Surgery, n(%) | XXX (XX.X) | XX (XX.X) | XX(XX.X) |
| Participants Receiving Unscheduled Surgery, n(%) | XXX(XX.X) | XX(XX.X) | XX(XX.X) |
| Pathologic Tumor - ypT in Participants Receiving Surgery at | t | | |
| C6D18, n(%) | | | |
| ypTx | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT0 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypTis | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT1mi | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT1a | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT1b | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT1c | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| урТ2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| урТЗ | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT4a | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT4b | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypT4c | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| No No | XXX (XX.X)<br>XXX (XX.X) | XX (XX.X)<br>XX (XX.X) | XXX (XX.X) |
| Yes | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Pathologic Lymph Nodes - ypN in Participants Receiving | | | |
| Surgery at C6D18, n(%) | | | |
| ypNX | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| ypN0 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypNO(i+) | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypN0 (mol+) | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypN1 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypN1mi | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypN1a | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypN1b | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypN1c | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| ypN2 | | XX (XX.X) | |
| ypN2<br>ypN2a | XXX (XX.X) | | XXX (XX.X) |
| ypN2b | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| уриз | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| уриз<br>уриЗа | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| уриза<br>ури3b | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| уризс | XXX (XX.X)<br>XXX (XX.X) | XX (XX.X)<br>XX (XX.X) | XXX (XX.X)<br>XXX (XX.X) |

<date> / <time> / / cogram name>

| C6D18, n(%) | | | |
|---|---|---|---|
| M0 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| pM1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Unknown | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Lymphatic Vascular Invasion Classification in P | articipants | | |

Source: Listing 16.2.6.8.

Date of data extraction: DDMMMYYYY; Date of Creation: DDMMMYYYY.

## Repeat the following table with Table 14.2.2.1.3.1 shell

Table 14.2.2.1.3.2
Summary of Post-Surgery Disease Staging
Analysis Set: Ki-67 Evaluable Set

Table 14.2.2.2 Summary of Modified Pre-operative Endocrine Prognostic Index (mPEPI) Score and mPEPI 0 Rate Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| Participants Not Assessed at C6D18, n(%) | XXX (XX.X) | XX (XX.X) | |
| mPEPI) Score at at C6D18, n(%) | | | |
| 0 | XXX(XX.X) | XX(XX.X) | |
| 1~2 | XXX(XX.X) | XX(XX.X) | |
| 3 | XXX(XX.X) | XX(XX.X) | |
| >3 | XXX(XX.X) | XX(XX.X) | |
| PEPI 0 Rate, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| dds Ratio of mPEPIO Rate [1] | XX.XX | | |
| 80% confidence interval [1] | XX.XX,XX.XX | | |
| 95% confidence interval [1] | XX.XX,XX.XX | | |
| odds Ratio of mPEPIO Rate [2] | XX.XX | | |
| 80% confidence interval [2] | XX.XX,XX.XX | | |
| 95% confidence interval [2] | XX.XX,XX.XX | | |

Note: mPEPIO rate is the proportion of participants achieving O for total mPEPI after treatment (before surgery).

<sup>[1]</sup> Analysis based on Cochran-Mantel-Haenszel method adjusted for the stratification factors, including baseline Ki-67 score (assessed centrally: <20% vs  $\geq$ 20%) and tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm). Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

<sup>[2]</sup> Analysis based on Cochran-Mantel-Haenszel method adjusted for the stratification factors, including baseline Ki-67 score (assessed locally: <20% vs  $\ge20\%$ ) and tumor size ( $\le2$  cm, >2 to <5 cm, or  $\ge5$  cm). Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT. Source: Listing 16.2.6.1.

Table 14.2.2.3

Summary of Breast Conserving Surgery (BCS) and BCS Rate
Analysis Set: Full Analysis Set

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Difference |
|---|---|---|---|
| Participants Not Receiving Surgery, n(%) | XXX (XX.X) | XX(XX.X) | |
| Participants Receiving Unscheduled Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| Participants Receiving Mastectomy at C6D18, n(%) | XXX(XX.X) | XX(XX.X) | |
| Participants Receiving Breast Conserving Surgery at C6D18, n(%) | XXX(XX.X) | XX(XX.X) | |
| BCS Rate in Participants Receiving Breast Conserving Surgery at C6D18, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |

Note: Breast conserving surgery (BCS) Rate is the proportion of participants receiving breast conserving surgery. Source: Listing 16.2.6.2.

Table 14.2.2.4

Summary of Radiographic Response per mRECIST during Cycle 6

Analysis Set: Full Analysis Set

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX |
|---|---|---|
| Radiographic Response per mRECIST during Cycle 6, n(%) | | |
| Complete response (CR) | XXX(XX.X) | XX(XX.X) |
| Partial response (PR) | XXX(XX.X) | XX(XX.X) |
| Stable disease (SD) | XXX(XX.X) | XX(XX.X) |
| Progressive disease (PD) | XXX(XX.X) | XX(XX.X) |
| Not evaluable (NE) | XXX(XX.X) | XX(XX.X) |

Note: Participants without disease assessment is categorized as Not evaluable.

Table 14.2.2.5.1

Summary of Complete Cycle Cell Arrest (CCCA) and CCCA Rate
Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| Complete Cycle Cell Arrest at Week 2, n(%) | | | |
| No | XXX(XX.X) | XX(XX.X) | |
| Yes | XXX(XX.X) | XX(XX.X) | |
| CCCA Rate, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| Odds Ratio of CCCA Rate [1] | XX.XX | | |
| 80% confidence interval [1] | XX.XX,XX.XX | | |
| 95% confidence interval [1] | XX.XX,XX.XX | | |
| Odds Ratio of CCCA Rate [2] | XX.XX | | |
| 80% confidence interval [2] | XX.XX,XX.XX | | |
| 95% confidence interval [2] | XX.XX,XX.XX | | |
| Participants Not Receiving Surgery, n(%) | XXX (XX.X) | XX(XX.X) | |
| Participants Receiving Unscheduled Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| Complete Cycle Cell Arrest at C6D18 Surgery, n(%)<br>No | VVV (VV V) | VV (VV V) | |
| | XXX (XX.X) | XX (XX.X) | |
| Yes | XXX (XX.X) | XX(XX.X) | |
| CCCA Rate, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| Odds Ratio of CCCA Rate [1] | XX.XX | | |
| 80% confidence interval [1] | XX.XX,XX.XX | | |
| 95% confidence interval [1] | XX.XX,XX.XX | | |
| Odds Ratio of CCCA Rate [2] | XX.XX | | |
| 80% confidence interval [2] | XX.XX,XX.XX | | |
| 95% confidence interval [2] | XX.XX,XX.XX | | |

Note: Complete cycle cell arrest (CCCA) at Week 2/surgery is defined as Ki67 score ≤ 2.7%. CCCA rate is the proportion of participants achieving CCCA) at Week 2 (or C1D15)/surgery.

<sup>[1]</sup> Analysis based on Cochran-Mantel-Haenszel method adjusted for the stratification factors, including baseline Ki-67 score (assessed centrally: <20% vs  $\ge20\%$ ) and tumor size ( $\le2$  cm, >2 to <5 cm, or  $\ge5$  cm). Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

<sup>[2]</sup> Analysis based on Cochran-Mantel-Haenszel method adjusted for the stratification factors, including baseline Ki-67 score (assessed locally: <20% vs  $\ge20\%$ ) and tumor size ( $\le2$  cm, >2 to <5 cm, or  $\ge5$  cm). Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

Table 14.2.2.5.2

Summary of Complete Cycle Cell Arrest (CCCA) and CCCA Rate - Subgroup Analysis by Central Ki-67 Baseline Score
Analysis Set: Full Analysis Set

Central Ki-67 Baseline Score: < 5%

| | ARV-471 | Anastrozole | · |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| Complete Cycle Cell Arrest at Week 2, n(%) | XXX (XX.X) | XX(XX.X) | |
| No | XXX(XX.X) | XX(XX.X) | |
| Yes | XXX(XX.X) | XX(XX.X) | |
| CCCA Rate, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| Odds Ratio of CCCA Rate [1] | XX.XX | | |
| 80% confidence interval [1] | XX.XX,XX.XX | | |
| 95% confidence interval [1] | XX.XX,XX.XX | | |
| Odds Ratio of CCCA Rate [2] | XX.XX | | |
| 80% confidence interval [2] | XX.XX,XX.XX | | |
| 95% confidence interval [2] | XX.XX,XX.XX | | |
| Participants Not Receiving Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| Participants Receiving Unscheduled Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| Complete Cycle Cell Arrest at C6D18 Surgery, n(%) | XXX(XX.X) | XX(XX.X) | |
| No | XXX(XX.X) | XX(XX.X) | |
| Yes | XXX(XX.X) | XX(XX.X) | |
| CCCA Rate, n(%) | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| 80% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% Wilson confidence interval | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| Odds Ratio of CCCA Rate [1] | XX.XX | | |
| 80% confidence interval [1] | XX.XX,XX.XX | | |
| 95% confidence interval [1] | XX.XX,XX.XX | | |
| Odds Ratio of CCCA Rate [2] | XX.XX | | |
| 80% confidence interval [2] | XX.XX,XX.XX | | |
| 95% confidence interval [2] | XX.XX,XX.XX | | |

Note: Complete cycle cell arrest (CCCA) at Week 2/surgery is defined as Ki67 score ≤ 2.7%. CCCA rate is the proportion of participants achieving CCCA at Week 2 (or C1D15)/surgery.

<sup>[1]</sup> Analysis based on Cochran-Mantel-Haenszel method adjusted for the stratification factors, including baseline Ki-67 score (assessed centrally: <20% vs  $\geq$ 20%) and tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm). Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

<sup>[2]</sup> Analysis based on Cochran-Mantel-Haenszel method adjusted for the stratification factors, including baseline Ki-67 score (assessed locally: <20% vs  $\ge20\%$ ) and tumor size ( $\le2$  cm, >2 to <5 cm, or  $\ge5$  cm). Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT.

Source: Listing 16.2.6.2.

## Programming Note:

Repeat the table for 'Central Ki-67 Baseline Score: ≥ 5%" on new page.

Table 14.2.3.1.1 Summary of the Primary Breast Tumor Change - Caliper-based Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Baseline (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Best Percentage Change from Baseline (%) | | | |
| n | XXX | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| <cycle day="" x="" y=""></cycle> | | | |
| Tumor Assessment (mm) | | | |
| n | XXX | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |

Note: The best percentage change from baseline is maximum percentage decrease or minimum percentage increase if there is no decrease per participant.

 ${\it Table~14.2.3.1.2}$  Summary of the Primary Breast Tumor Change - Caliper-based by Baseline Tumor Size Analysis Set: Full Analysis Set

Baseline Tumor Size: ≤2 cm

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Baseline (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Best Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | xx.x | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| <cycle day="" x="" y=""></cycle> | | | |
| Tumor Assessment (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |

#### <insert Visit>

Note: The best percentage change from baseline is maximum percentage decrease or minimum percentage increase if there is no decrease per participant.

Note: Baseline tumor size categories are derived based on data collected instead of data reported in IRT. Source: Listing 16.2.6.4.

## Programming Note:

Repeated >2 to <5 cm, and  $\ge 5$  cm on separated pages

Table 14.2.3.2.1 Summary of Target Lesion Change Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Baseline (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Best Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| <cycle day="" x="" y=""></cycle> | | | |
| Tumor Assessment (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |

Note: The percentage change is based on the sum of all target lesions per participant.

Note: The best percentage change from baseline is maximum percentage decrease or minimum percentage increase if there is no decrease per participant.

Table 14.2.3.2.2

Summary of Target Lesion Change by Baseline Tumor Size
Analysis Set: Full Analysis Set

Baseline Tumor Size: ≤2 cm

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Baseline (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Best Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| <cycle day="" x="" y=""></cycle> | | | |
| Tumor Assessment (mm) | | | |
| n | XXX | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |

#### <insert Visit>

Note: The percentage change is based on the sum of all target lesions per participant.

Note: The best percentage change from baseline is maximum percentage decrease or minimum percentage increase if there is no decrease per participant.

Note: Baseline tumor size categories are derived based on data collected instead of data reported in IRT.

Source: Listing 16.2.6.3.

## Programming Note:

Repeated >2 to <5 cm, and  $\ge5$  cm on separated pages

Table 14.2.3.3.1 Summary of Target Lesion (Primary Tumor) Change Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Baseline (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Best Percentage Change from Baseline (%) | | | |
| n | XXX | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| <pre><cycle day="" x="" y=""></cycle></pre> | | | |
| Tumor Assessment (mm) | | | |
| n | XXX | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | xx.x | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |

Note: The percentage change is based on the target lesions being marked as the primary tumor per participant.

Note: The best percentage change from baseline is maximum percentage decrease or minimum percentage increase if there is no decrease per participant.

Table 14.2.3.3.2 Summary of Target Lesion (Primary Tumor) Change by Baseline Tumor SizeAnalysis Set: Full Analysis Set

Baseline Tumor Size: ≤2 cm

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Total<br>N=XXX |
|---|---|---|---|
| Baseline (mm) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Best Percentage Change from Baseline (%) | | | |
| n | xxx | xx | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | xx.x | xx.x | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Cycle x Day Y> | | | |
| Tumor Assessment (mm) | | | |
| n | XXX | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| Median | xx.x | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Percentage Change from Baseline (%) | | | |
| n | XXX | XX | XX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| | XX.X | XX.X | XX.X |
| Median | | | |

Note: The percentage change is based on the target lesions being marked as the primary tumor per participant.

Note: The best percentage change from baseline is maximum percentage decrease or minimum percentage increase if there is no decrease per participant.

Note: Baseline tumor size categories are derived based on data collected instead of data reported in IRT.

Source: Listing 16.2.6.3.

## Programming Note:

Repeated >2 to <5 cm, and  $\ge 5$  cm on separated pages

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Difference |
|---|---|---|---|
| ER AQUA score at baseline | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| ER AQUA score at C1D15 | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| ER AQUA score percentage change at C1D15 | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 95% Confidence Interval for LSM[1] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |

Note: AQUA = absolute quantification score in arbitrary units.

## Programming Note:

<sup>[1]</sup> Analysis based on an analysis of covariance (ANCOVA) model with baseline Ki-67 score (assessed <u>centrally</u>: <20% vs  $\geq$ 20%), the tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm) as covariates for treatment. Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT. Source: Listing 16.2.6.2.

| | ARV-471<br>200 mg N=XXX | Anastrozole | Difference |
|---|---|---|---|
| | | 1 mg N=XX | |
| ER AQUA score at baseline | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| ER AQUA score at C1D15 | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| ER AQUA score percentage change at C1D15 | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |

Note: AQUA = absolute quantification score in arbitrary units. [1] Analysis based on an analysis of variance (ANOVA) model. Source: Listing 16.2.6.2.

#### Programming Note:

Table 14.2.4.1.3

Summary of Log-Transformed ER AQUA Score Change at C1D15 from Baseline Value without Covariate Analysis Set: Full Analysis Set

| | ARV-471<br>200 mg N=XXX | Anastrozole | |
|---|---|---|---|
| | | 1 mg N=XX | Difference |
| log(ER AQUA score at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(ER AQUA score at C1D15) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(ER AQUA score at C1D15) - log(ER AQUA score at baseline | ) | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between ER AQUA score at C1D15 and baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2 | ] | | xx.xx, xx.xx |
| 95% Confidence Interval for Geometric Means Difference[2 | 1 | | xx.xx, xx.xx |

Note: AQUA = absolute quantification score in arbitrary units.

<sup>[1]</sup> Analysis based on an analysis of variance (ANOVA) model.

<sup>[2]</sup> Back transformed values of [1].

Table 14.2.4.2.1

Summary of ER AQUA Score Percentage Change at Surgery from Baseline Value
Analysis Set: Full Analysis Set

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Difference |
|---|---|---|---|
| ER AQUA score at baseline | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| ER AQUA score at surgery | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| IR AQUA score percentage change at surgery | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | XX.XX, XX.XX | XX.XX, XX.XX | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |

Note: AQUA = absolute quantification score in arbitrary units.

<sup>[1]</sup> Analysis based on an analysis of covariance (ANCOVA) model with baseline Ki-67 score (assessed <u>centrally</u>: <20% vs  $\geq$ 20%), the tumor size ( $\leq$ 2 cm, >2 to <5 cm, or  $\geq$ 5 cm) as covariates for treatment. Baseline Ki-67 score and/or the tumor size categories are derived based on data collected instead of data reported in IRT. Source: Listing 16.2.6.2.
Table 14.2.4.2.2 Summary of ER AQUA Score Percentage Change at Surgery from Baseline Value without Covariate Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| ER AQUA score at baseline | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| ER AQUA score at surgery | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| ER AQUA score percentage change at surgery | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |

Note: AQUA = absolute quantification score in arbitrary units. [1] Analysis based on an analysis of variance (ANOVA) model. Source: Listing 16.2.6.2.

Table 14.2.4.2.3

Summary of Log-Transformed ER AQUA Score Change at Surgery from Baseline Value without Covariate Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(ER AQUA score at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(ER AQUA score at surgery) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(ER AQUA score at surgery) - log(ER AQUA score at baselir | ne) | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| Ratio between ER AQUA score at Surgery and baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | xx.xx, xx.xx |

Note: AQUA = absolute quantification score in arbitrary units.

Source: Listing 16.2.6.2.

<sup>[1]</sup> Analysis based on an analysis of variance (ANOVA) model.

<sup>[2]</sup> Back transformed values of [1].

Table 14.2.5.1.1

Summary of PR H-score Percentage Change at C1D15 from Baseline Value without Covariate Analysis Set: Full Analysis Set

| | ARV-471<br>200 mg N=XXX | Anastrozole | |
|---|---|---|---|
| | | 1 mg N=XX | Difference |
| PR H-score at baseline | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| PR H-score at C1D15 | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| PR H-score percentage change at C1D15 | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | XX.XX, XX.XX | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |

Note: PR (progesterone receptor) H-score = (SCORE\_1)\*1 + (SCORE\_2)\*2 + (SCORE\_3)\*3 from PgR636 assessment. [1] Analysis based on an analysis of variance (ANOVA) model. Source: Listing 16.2.6.1.

Table 14.2.5.1.2

Summary of Log-Transformed PR H-score Change at C1D15 from Baseline Value without Covariate Analysis Set: Full Analysis Set

| | ARV-471 Anastrozole | | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(PR H-score at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | xx.x | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| log(PR H-score at C1D15) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(PR H-score at C1D15) - log(PR H-score at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between PR H-score at C1D15 and baseline | | | |
| Geometric Means[2] | xx.x | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: PR (progesterone receptor) H-score = (SCORE 1)\*1 + (SCORE 2)\*2 + (SCORE 3)\*3 from PgR636 assessment.

Source: Listing 16.2.6.1.

<sup>[1]</sup> Analysis based on an analysis of variance (ANOVA) model.

<sup>[2]</sup> Back transformed values of [1].

Table 14.2.5.2.1

Summary of PR H-score Percentage Change at Surgery from Baseline Value without Covariate
Analysis Set: Full Analysis Set

| | ARV-471 | Anastrozole | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| PR H-score at baseline | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| PR H-score at surgery | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| PR H-score percentage change at surgery | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | xx, xx | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx |
| 80% Confidence Interval for LSM[1] | XX.XX, XX.XX | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | XX.XX, XX.XX | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |
| 95% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.X |

Note: PR (progesterone receptor) H-score = (SCORE\_1)\*1 + (SCORE\_2)\*2 + (SCORE\_3)\*3 from PgR636 assessment. [1] Analysis based on an analysis of variance (ANOVA) model. Source: Listing 16.2.6.1.

 ${\it Table 14.2.5.2.2} \\ {\it Summary of Log-Transformed PR H-score Change at Surgery from Baseline Value without Covariate } \\ {\it Analysis Set: Full Analysis Set} \\$ 

| | ARV-471 Anastrozole | | |
|---|---|---|---|
| | 200 mg N=XXX | 1 mg N=XX | Difference |
| log(PR H-score at baseline) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(PR H-score at surgery) | | | |
| n | XXX | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | XX, XX | XX, XX | |
| log(PR H-score at surgery) - log(PR H-score at baseline) | | | |
| n | xxx | XX | |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | |
| Median | XX.X | XX.X | |
| Min, Max | xx, xx | XX, XX | |
| LSM (Standard Error)[1] | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| 80% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for LSM[1] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for LSM Difference[1] | | | XX.XX, XX.XX |
| 95% Confidence Interval for LSM Difference[1] | | | xx.xx, xx.xx |
| Ratio between PR H-score at surgery and baseline | | | |
| Geometric Means[2] | XX.X | XX.X | XX.X |
| 80% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 95% Confidence Interval for Geometric Means[2] | xx.xx, xx.xx | xx.xx, xx.xx | |
| 80% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |
| 95% Confidence Interval for Geometric Means Difference[2] | | | XX.XX, XX.XX |

Note: PR (progesterone receptor) H-score = (SCORE\_1)\*1 + (SCORE\_2)\*2 + (SCORE\_3)\*3 from PgR636 assessment.

Source: Listing 16.2.6.1.

<sup>[1]</sup> Analysis based on an analysis of variance (ANOVA) model.

<sup>[2]</sup> Back transformed values of [1].

Table 14.3.1
Summary of Treatment Emergent Adverse Events Overview
Analysis Set: Safety Analysis Set

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| Number of subjects with any of, n(%) | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| TEAEs | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| TEAEs related to study drug | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| TEAEs with grade 3 or higher | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| TEAEs with grade 3 or higher related to study drug | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| erious TEAEs | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| erious TEAEs related to study drug | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| EAEs leading to drug withdrawn | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| EAEs related to study drug leading to drug withdrawn | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| EAEs leading to drug interruption | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| EAEs related to study drug leading to drug interruption | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| EAEs leading to dose reduction | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| EAEs related to study drug leading to dose reduction | XXX(XX.X) | XX (XX.X) | XXX(XX.X) |
| EAEs with outcome of death | XXX(XX.X) | XX (XX.X) | XXX(XX.X) |

Note: A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV-471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Source: Listing 16.2.7.1.

Table 14.3.2.1

Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term
Analysis Set: Safety Analysis Set

| System organ class | ARV-471 | Anastrozole | Total |
|------------------------------|--------------|-------------|----------|
| Preferred Term | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Subjects with any TEAE, n(%) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| System organ class 1 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term 1 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term 2 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| System organ class 2 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term 1 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term 2 | XX (XX.X) | XX (XX.X) | XX(XX.X) |

Note: Adverse events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version 27.0.

Note: A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Source: Listings 16.2.7.1.

Repeat the following tables with Table 14.3.2.1 shell

Table 14.3.2.2

Summary of Treatment Emergent Adverse Events Related to Study Drug by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

Programming Note: update "Subjects with any TEAE" to "Subjects with any TEAE Related to Study Drug"

Table 14.3.2.3

Summary of Treatment Emergent Adverse Events with Grade 3 or Higher by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

Programming Note: update "Subjects with any TEAE" to "Subjects with any Grade 3 or higher TEAE"

Table 14.3.2.4

Summary of Treatment Emergent Adverse Events with Grade 3 or Higher Related to Study Drug by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

Programming Note: update "Subjects with any TEAE" to "Subjects with any Grade 3 or higher TEAE Related to Study Drug"

Table 14.3.2.5.1

Summary of Treatment Emergent Adverse Events Leading to Drug Withdrawn by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

Programming Note:

update "Subjects with any TEAE" to "Subjects with any TEAE Leading to Drug Withdrawn"

Table 14.3.2.5.2

Summary of Treatment Emergent Adverse Events Related to Study Drug Leading to Drug Withdrawn by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

# Programming Note:

update "Subjects with any TEAE" to "Subjects with any TEAE Related to Study Drug Leading to Drug Withdrawn"

Table 14.3.2.6.1

Summary of Treatment Emergent Adverse Events Leading to Drug Interrupted by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

# Programming Note:

update "Subjects with any TEAE" to "Subjects with any TEAE Leading to Drug Interrupted"

Table 14.3.2.6.2

Summary of Treatment Emergent Adverse Events Related to Study Drug Leading to Drug Interrupted by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

#### Programming Note:

update "Subjects with any TEAE" to "Subjects with any TEAE Related to Study Drug Leading to Drug Interrupted"

Table 14.3.2.7.1

Summary of Treatment Emergent Adverse Events Leading to Dose Reduced by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

# Programming Note:

update "Subjects with any TEAE" to "Subjects with any TEAE Leading to Dose Reduced"

Table 14.3.2.7.2

Summary of Treatment Emergent Adverse Events Related to Study Drug Leading to Dose Reduced by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

# Programming Note:

update "Subjects with any TEAE" to "Subjects with any TEAE Related to Study Drug Leading to Dose Reduced"

Table 14.3.2.8

Summary of Treatment Emergent Adverse Events by Preferred Term
Analysis Set: Safety Analysis Set

| Preferred Term | ARV-471<br>200 mg N=XX | Anastrozole<br>1 mg N=XX | Total<br>N=XXX |
|---|---|---|---|
| Subjects with any TEAE, n(%) | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Term 1 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Preferred Term 2 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Term 3 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Term 4 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |

Note: Adverse events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version 27.0.

Note: A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Source: Listings 16.2.7.1.

# Programming Note:

Repeat the following tables with Table 14.3.2.8 shell

Table 14.3.2.9

Summary of Treatment Emergent Adverse Events Related to Study Drug by Preferred Term

Analysis Set: Safety Analysis Set

Programming Note: update "Subjects with any TEAE" to "Subjects with any TEAE Related to Study Drug"

Table 14.3.2.10

Summary of Treatment Emergent Adverse Events by System Organ Class,
Preferred Term and Maximum CTCAE Grade
Analysis Set: Safety Analysis Set

| System organ class | ARV-471 | Anastrozole | Total |
|------------------------------|--------------|-------------|------------|
| Preferred Term | | | |
| CTCAE Grade | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Subjects with any TEAE, n(%) | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 3 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 4 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 5 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| System organ class 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 3 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 4 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 5 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Preferred Term 1 | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 1 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 2 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 3 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 4 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 5 | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

Note: Adverse events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version 27.0, and graded according to the NCI-CTCAE version 5.0.

Note: A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV-471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Source: Listings 16.2.7.1.

# Repeat the following tables with Table 14.3.2.10 shell

# ${\tt Table~14.3.2.11}\\ {\tt Summary~of~Treatment~Emergent~Adverse~Events~Related~to~Study~Drug~by~System~Organ~Class,}$

ummary of Treatment Emergent Adverse Events Related to Study Drug by System Organ Class Preferred Term and Maximum CTCAE Grade Analysis Set: Safety Analysis Set

Programming Note: update "Subjects with any TEAE" to "Subjects with any TEAE Related to Study Drug"

Table 14.3.2.12

Summary of MedDRA SMQ for Torsade de Pointes by Preferred Term and Maximum CTCAE Grade
Analysis Set: Safety Analysis Set

| Preferred Term | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| CTCAE Grade | 200 mg N=XX | 1 mg N=XX | N=XXX |
| Subjects with any SMQ for Torsade de Pointes, n(%) | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Grade 1 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Grade 2 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Grade 3 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Grade 4 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Grade 5 | XXX (XX.X) | XX (XX.X) | XXX (XX.X) |
| Preferred Term 1 | XXX (XX.X) | XX (XX.X) | XXX(XX.X) |
| Grade 1 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 2 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 3 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 4 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 5 | XXX(XX.X) | XX(XX.X) | XXX (XX.X) |
| Preferred Term 2 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 1 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 2 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 3 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |
| Grade 4 | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Grade 5 | XXX (XX.X) | XX(XX.X) | XXX (XX.X) |

Note: Adverse events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version 27.0, and graded according to the NCI-CTCAE version 5.0.

Source: Listings 16.2.7.1.

# Programming Note:

PTs include Electrocardiogram QT interval abnormal, Electrocardiogram QT prolonged, Long QT syndrome, Long QT syndrome congenital, Torsade de pointes, Ventricular tachycardia, Arrhythmic storm, Cardiac arrest, Cardiac death, Cardiac fibrillation, Cardiorespiratory arrest, Electrocardiogram repolarisation abnormality, Electrocardiogram U wave inversion, Electrocardiogram U wave present, Electrocardiogram U-wave abnormality, Loss of consciousness, Seizure, Sudden cardiac death, Sudden death, Syncope, Ventricular arrhythmia, Ventricular fibrillation, Ventricular flutter, Ventricular tachyarrhythmia.

#### Repeat the following tables with Table 14.3.2.1 shell

Table 14.3.3.1

Programming Note:

update "Subjects with any TEAE" to "Subjects with any Serious TEAE" update "Source: Listings 16.2.7.1." to "Source: Listings 16.2.7.2."

Table 14.3.3.2

Summary of Serious Treatment Emergent Adverse Events Related to Study Drug by System Organ Class and Preferred Term

Analysis Set: Safety Analysis Set

Programming Note:

update "Subjects with any TEAE" to "Subjects with any Serious TEAE Related to Study Drug" update "Source: Listings 16.2.7.1." to "Source: Listings 16.2.7.2."

Repeat the following tables with Table 14.3.2.8 shell

Table 14.3.3.3

Summary of Serious Treatment Emergent Adverse Events by Preferred Term Analysis Set: Safety Analysis Set

Programming Note:

update "Subjects with any TEAE" to "Subjects with any Serious TEAE" update "Source: Listings 16.2.7.1." to "Source: Listings 16.2.7.2."

#### Table 14.3.3.4

Summary of Serious Treatment Emergent Adverse Events Related to Study Drug by Preferred Term Analysis Set: Safety Analysis Set

# Programming Note:

update "Subjects with any TEAE" to "Subjects with any Serious TEAE Related to Study Drug" update "Source: Listings 16.2.7.1." to "Source: Listings 16.2.7.2."

Repeat the following tables with Table 14.3.2.10 shell

Table 14.3.3.5

Summary of Serious Treatment Emergent Adverse Events by System Organ Class,

Preferred Term and Maximum CTCAE Grade

Analysis Set: Safety Analysis Set

#### Programming Note:

update "Subjects with any TEAE" to "Subjects with any Serious TEAE" update "Source: Listings 16.2.7.1." to "Source: Listings 16.2.7.2."

Table 14.3.3.6

Summary of Serious Treatment Emergent Adverse Events Related to Study Drug by System Organ Class,
Preferred Term and Maximum CTCAE Grade
Analysis Set: Safety Analysis Set

# Programming Note:

update "Subjects with any TEAE" to "Subjects with any Serious TEAE Related to Study Drug" update "Source: Listings 16.2.7.1." to "Source: Listings 16.2.7.2."

Repeat the following tables with Table 14.3.2.1 shell

Table 14.3.3.7

Summary of Treatment Emergent Adverse Events Leading to Death by System Organ Class

and Preferred Term Analysis Set: Safety Analysis Set

# Programming Note:

update "Subjects with any TEAE" to "Subjects with any TEAE Leading to Death"

Table 14.3.3.8 Summary of Subject Death Analysis Set: Safety Analysis Set

| | ARV-471<br>200 mg N=XXX | Anastrozole<br>1 mg N=XX | Total<br>N=XXX |
|---|---|---|---|
| Number of Subject Death, n(%) | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |
| Reason of Subject Death, n(%) | | | |
| Disease progression | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Adverse Event | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Unknown | XXX(XX.X) | XX (XX.X) | XXX(XX.X) |
| Other | XXX (XX.X) | XX(XX.X) | XXX(XX.X) |

Source: Listing 16.2.1.1.

Table 14.3.7.1 Summary of Hematology Laboratory by Visit Analysis Set: Safety Analysis Set

Test (SI unit): Hemoglobin (g/L)

| | ARV-471 | Anastrozole | Total |
|---------------------------|--------------|-------------|-------------|
| Time point | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Baseline | | | |
| n | XXX | xx | XXX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Cycle 1 Day x | | | |
| Absolute Value | | | |
| n | XXX | xx | XXX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| Change from Baseline | | | |
| n | XXX | xx | XXX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |

Note: The baseline value is defined to be the last non-missing assessment on/before the date of the first ARV-

471/anastrozole dose. Source: Listing 16.2.8.3.

Programming Note:

Each Test starts from a new page.

# Repeat the following tables with Table 14.3.7.1 shell

Table 14.3.7.3

Summary of Coagulation Laboratory by Visit
Analysis Set: Safety Analysis Set

Replace 'Source: Listing 16.2.8.3' with 'Source: Listing 16.2.8.5'

Table 14.3.7.5

Summary of Serum Chemistry Laboratory by Visit

Analysis Set: Safety Analysis Set

Replace 'Source: Listing 16.2.8.3' with 'Source: Listing 16.2.8.4'

Table 14.3.7.2.1
Shift of Hematology CTCAE Grade from Baseline to Worst Post-baseline
Analysis Set: Safety Analysis Set

Test: Anemia

| | | Worst Post-baseline CTCAE Grade, n(%) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Baseline<br>CTCAE Grade | | | | | | | |
| | | Missing | 0 | 1 | 2 | 3 | 4 | Total |
| ARV-471200 mg (N=XXX) | Missing | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| - | 0 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 1 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 2 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 3 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 4 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | Total | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(100) |
| Anastrozole 1 mg (N=XX) | Missing | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 0 | XX(XX.X) | XX(XX,X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) |
| | 1 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 2 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 3 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 4 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | Total | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(100) |
| Total (N=XXX) | Missing | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) |
| | 0 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 1 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 2 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 3 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | 4 | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XXX (100) |

Note: The baseline value is defined to be the last non-missing assessment on/before the date of the first ARV-

471/anastrozole dose.

Note: Grade is derived using CTCAE 5.0.

Source: Listing 16.2.8.3.

# Programming Note:

Each Test starts from a new page

Table 14.3.7.2.2

Summary of Hematology CTCAE On-Treatment Worsening
Analysis Set: Safety Analysis Set

| | AR | V-471 200 mg N=XXX | Ar | Anastrozole 1 mg N=XX |
|---|---|---|---|---|
| | N' | Worsened from Baseline, n(%) | N' | Worsten from Baseline, n(%) |
| Neutrophil count decreased | XXX | XX (XX.X) | XXX | XX (XX.X) |
| White blood cell count decrease | XXX | XX(XX.X) | XXX | XX(XX.X) |
| Anemia | XXX | XX(XX.X) | XXX | XX(XX.X) |
| Platelat count decreased | XXX | XX(XX.X) | XXX | XX(XX.X) |

Note: The baseline value is defined to be the last non-missing assessment on/before the date of the first ARV-471/anastrozole dose.

Note: Include lab data up to 28 days after the last dose of study intervention, which is grade using CTCAE 5.0. Note: N' is the number of participants with baseline and at least on on-treatment assessment for the parameter of interest. It is the denominator of the percentage. n is the number of participants with CTCAE grade of on-treatment lab results worsten than baseline CTCAE grade.

Note: Treatment-worsening shift includes grade 0 baseline to grade 1/2/3/4 postbaseline, grade 1 at baseline to grade 2/3/4 postbaseline, grade 2 at baseline to grade 3/4 postbaseline, or grade 3 at baseline to grade 4 postbaseline. Source: Listing 16.2.8.3

# Repeat the following tables with Table 14.3.7.2.1 shell

Table 14.3.7.4

Shift of Coagulation CTCAE Grade from Baseline to Worst Post-baseline Analysis Set: Safety Analysis Set

Replace 'Source: Listing 16.2.8.3' with 'Source: Listing 16.2.8.5'

Table 14.3.7.6
Shift of Serum Chemistry CTCAE Grade from Baseline to Worst Post-baseline
Analysis Set: Safety Analysis Set

Replace 'Source: Listing 16.2.8.3' with 'Source: Listing 16.2.8.4'

Table 14.3.8.1 Summary of 12-lead ECGs by Visit Analysis Set: Safety Analysis Set

Test (SI unit): Heart rate (beats/min)

| | ARV-471 | Anastrozole | Total |
|---------------------------|--------------|-------------|-------------|
| Time point | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| Baseline | | | |
| n | xxx | xx | XXX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Cycle 1 Day x | | | |
| Absolute Value | | | |
| n | XXX | xx | XXX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| Change from Baseline | | | |
| n | XXX | xx | XXX |
| Mean (Standard Deviation) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |

Note: The baseline value is defined to be the last non-missing assessment on/before the date of the first ARV-471/anastrozole dose.

Source: Listing 16.2.10.

# Programming Note:

Each test starts on a new page.

Table 14.3.8.2 Summary of QTcF/QTcB Interval Clinically Significant Analysis Set: Safety Analysis Set

Test: QTcF

| | ARV-471 | Anastrozole | Total |
|---|---|---|---|
| Time point | 200 mg N=XXX | 1 mg N=XX | N=XXX |
| QTcF at Baseline, n(%) | | | |
| QTcF >450 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| QTcF >480 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| QTcF >500 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| QTcF Worst Post-Baseline, n(%) | | | |
| QTcF >450 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| QTcF >480 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| QTcF >500 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| TcF Worst Change from Baseline, n(%) | | | |
| >30 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| >60 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Cycle X Day Y, n(%) | | | |
| Value QTcF >450 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Value QTcF >480 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Value QTcF >500 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Change from baseline >30 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |
| Change from baseline >60 msec | XXX(XX.X) | XX(XX.X) | XXX(XX.X) |

<insert Visit>

Note: The baseline value is defined to be the last non-missing assessment on/before the date of the first ARV-471/anastrozole dose.

Source: Listing 16.2.10.

# Programming Note:

Repeat Table for QTcB and Change QTcF to QTcB in the Table

Table 14.3.10

Summary of ARV-471 and ARV-473 Plasma Concentration (unit) by Visit

Analysis Set: Pharmacokinetic Analysis Set

| | | | | Min, Max | Geometric Mean | Geometric |
|---|---|---|---|---|---|---|
| | n | Mean (SD) | Median | | | CV <del>%</del> |
| ARV-471 Plasm Concentration (unit) | | | | | | |
| Pre-biopsy | XXX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| CxDy Pre-dose | XXX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| CxDy 1 hour (± 15 min) post-dose | XXX | xx.x(xx.xx) | XX.X | XX,XX | xx.x | XX.XX |
| CxDy 2 hours (± 15 min) post-dose | XXX | xx.x(xx.xx) | XX.X | XX,XX | xx.x | XX.XX |
| CxDy 4 hours (± 30 min) post-dose | XXX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| Pre-surgery | XXX | xx.x(xx.xx) | xx.x | xx,xx | XX.X | xx.xx |
| ARV-473 Plasm Concentration (unit) | | | | | | |
| Pre-biopsy | XXX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| CxDy Pre-dose | XXX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| CxDy 1 hour (± 15 min) post-dose | XXX | xx.x(xx.xx) | XX.X | XX,XX | xx.x | XX.XX |
| CxDy 2 hours (± 15 min) post-dose | XXX | xx.x(xx.xx) | XX.X | XX,XX | xx.x | XX.XX |
| CxDy 4 hours (± 30 min) post-dose | XXX | xx.x(xx.xx) | XX.X | xx, xx | XX.X | XX.XX |
| Pre-surgery | XXX | xx.x(xx.xx) | XX.X | xx,xx | XX.X | XX.XX |

Note: SD = Standard deviation; CV = Coefficient of variation.

Source: Listing 16.2.5.4.

Figure 14.2.1.1 Spider Plot for Individual Ki-67 Value Analysis Set: Full Analysis Set



Note: N is the number of participants in the Full Analysis Set. n is the number of participants with Ki-67 assessment at each visit.

Note: Week 2 Visit occurs on Cycle 1 Day 15 (C1D15).Note: Missing data is not included in the ARV-471 and anastrozole plots. Subjects treated with ARV-471 with missing data at baseline include XXX, XXXX, XXXX; with missing at week 2 include XXXX, XXXXX, XXXXX; with missing at C6D18 include 015-002, 015-005, xxxx. Subjects treated with Anastrozle with missing data at baseline include XXXX, XXXXX, XXXX, with missing at week 2 include XXXX, XXXXX, with missing at C6D18 include xxx, xxxx, xxxx.

Source: Listing 16.2.6.1.

Figure 14.2.1.2.1

Box Plot for Ki-67 Percentage Change from Baseline at Cycle 1 Day 15

Analysis Set: Ki-67 Evaluable Set



Note: Ki-67 Percentage Change from Baseline at C1D15 = 100 × (Ki-67 at C1D15 - Ki-67 at baseline)/Ki-67 at baseline.

Note: N is the number of participants in the Ki-67 Evaluable Set. n is the number of participants with Ki-67 assessment at baseline and C1D15.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot.

Source: Table 14.2.1.1.3 and Listing 16.2.6.1.

# Programming Note:

Add panel on separated page for Surgery

Figure 14.2.1.2.2

Box Plot for Ki-67 Percentage Change from Baseline at Surgery

Analysis Set: Full Analysis Set



Note: Ki-67 Percentage Change from Baseline at surgery = 100 ×(Ki-67 at surgery - Ki-67 at baseline)/Ki-67 at baseline. Note: N is the number of participants in the Full Analysis Set. n is the number of participants with Ki-67 assessment at baseline and Surgery (C6D18).

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot. Source: Table 14.2.1.3.3 and Listing 16.2.6.1.

Figure 14.2.3.1

Waterfall Plot for Best Percentage Change of Primary Tumor from Baseline (Caliper-based)

Analysis Set: Full Analysis Set



Note: Best percentage change of primary tumor from baseline is maximum decrease or minimum increase if no decrease being observed.

Note: N is the number of participants in the Full Analysis Set. n is the number of participants with Primary Tumor assessment at baseline and post-baseline.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot. Source: Listing 16.2.6.2.

# Programming Note:

• ARV- 471 uses blue color and Anastrozle uses red color as Figure 14.2.1.1.Add subject ID at the bottom.

Figure 14.2.3.2.1

Waterfall Plot for Best Percentage Change of Target Lesion from Baseline
Analysis Set: Full Analysis Set



Note: Best percentage change of all targte lesions from baseline is maximum decrease or minimum increase if no decrease being observed.

Note: N is the number of participants in the Full Analysis Set. n is the number of participants with Target Lesion assessment at baseline and post-baseline.

Note: Select Best Overall Response(BOR) based on the order: CR, PR, SD, PD, NE.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot.Source: Table 14.2.3.2 and 16.2.6.3.

- ARV- 471 uses blue color and Anastrozle uses red color as Figure 14.2.1.1.
- Add subject ID at the bottom. add BOR on the top or bottom of each bar.Please use imgsu. IMGSRES and imgun. IMGRESP for Figure 14.2.3.2.1 (select the best response based on the sequency of CR>PR>SD>PD>NE)

Figure 14.2.3.2.2

Spider Plot for the Percent Target Lesion Size Change from Baseline by Subject and Timepoint Analysis Set: Full Analysis Set





Note: The percentage change is based on the sum of all target lesions per participant.

Note: N is the number of participants in the Full Analysis Set. n is the number of participants with Target Lesion assessment at baseline and post-baseline.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot.Source: Table 14.2.3.2 and 16.2.6.3.

- ARV- 471 uses blue color and Anastrozle uses red color as Figure 14.2.1.1.
- Timepoint use Screen, Cycle 1, Cycle 2, Cycle 3 ..... instead of Time (week)

Figure 14.2.4.1

Spider Plot for Individual ER AQUA Score
Analysis Set: Full Analysis Set



Note: N is the number of participants in the Full Analysis Set. n is the number of participants with ER AQUA Score at each visit.

Note: Missing data is not included in the ARV-471 and anastrozole plots. Subjects treated with ARV-471 with missing data at baseline include XXX, XXXX, XXXX, with missing at week 2 include XXXX, XXXXX, XXXXX; with missing at C6D18 include 015-002, 015-005, xxxx. Subjects treated with Anastrozle do not have ER AQUA score assessment. Source: Table 14.2.1.1.3 and Listing 16.2.6.2.

Note: Week 2 Visit occurs on Cycle 1 Day 15 (C1D15).

Figure 14.2.4.2.1

Box Plot for ER AQUA Score Percentage Change from Baseline at Cycle 1 Day 15

Analysis Set: Full Analysis Set



Note: ER AQUA Score Percentage Change from Baseline at C1D15 = 100 × (ER AQUA Score at C1D15 - ER AQUA Score at baseline)/ER AQUA Score at baseline.

Note: N is the number of participants in the Full Analysis Set. n is the number of participants with ER AQUA Score at baseline and C1D15.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot. Source: Table 14.2.4.1.2 and Listing 16.2.6.2.

# Programming Note:

See Figure 14.2.1.2.1 for reference as well.

Figure 14.2.4.2.2

Box Plot for ER AQUA Score Percentage Change from Baseline at Surgery

Analysis Set: Full Analysis Set



Note: ER AQUA Score Percentage Change from Baseline at surgery = 100 × (ER AQUA Score at surgery - ER AQUA Score at baseline) / ER AQUA Score at baseline.

Note: N is the number of participants in the Full Analysis Set. n is the number of participants with ER AQUA Score at baseline and Surgery (C6D18).

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot. Source: Table 14.2.4.2.2 and Listing 16.2.6.2.

# Programming Note:

See Figure 14.2.1.2.1 for reference as well.

Figure 14.2.5.1 Spider Plot for Individual PR H-score Analysis Set: Full Analysis Set



Note: N is the number of participants in the Full Analysis Set. n is the number of participants with PR H-score at each visit.

Note: Missing data is not included in the ARV-471 and anastrozole plots. Subjects treated with ARV-471 with missing data at baseline include XXX, XXXX, XXXX; with missing at week 2 include XXXX, XXXXX, WITH missing at C6D18 include 015-002, 015-005, xxxx. Subjects treated with Anastrozle with missing data at baseline include XXXX, XXXXX, with missing at week 2 include XXXX, XXXXX, with missing at C6D18 include xxx, xxxx, xxxxx. Source: Listing 16.2.6.1.

Note: Week 2 Visit occurs on Cycle 1 Day 15 (C1D15).

Figure 14.2.5.2.1

Box Plot for PR H-score Percentage Change from Baseline at Cycle 1 Day 15

Analysis Set: Full Analysis Set



Note: PR H-score Percentage Change from Baseline at C1D15 = 100 × ( PR H-score at C1D15 - PR H-score at baseline)/PR H-score at baseline.

Note: N is the number of participants in the Full Analysis Set. n is the number of participants with PR H-score at baseline and C1D15.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot. Source: Listing 16.2.6.1.
Figure 14.2.5.2.2

Box Plot for PR H-score Percentage Change from Baseline at Surgery

Analysis Set: Full Analysis Set



Note: PR H-score Percentage Change from Baseline at surgery = 100 × (PR H-score at surgery - PR H-score at baseline)/PR H-score at baseline.

Note: N is the number of participants in the Full Analysis Set. n is the number of participants with PR H-score at baseline and Surgery (C6D18).

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the ARV-471 plot.

Note: Subjects without baseline and/or postbaseline assessment (XXXX, XXX, and XXX), or with different number of tumor at baseline/postbaseline (XXX, XXX, and XXXX) are not included in the Anastrozle plot.

Source: Listing 16.2.6.1.

Figure 14.3.2.8

Tornado Plot for Treatment Emergent Adverse Events by Preferred Term
Analysis Set: Safety Analysis Set



Note: Adverse events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version 27.0.

Note: A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Source: Table 14.3.2.8, Table 14.3.2.3 and Listings 16.2.7.1.

# Programming Note:

• Add figure legend to indicate Arm A and Arm B color.

Listing 16.2.1.1 Subject Enrollment Analysis Set: Full Analysis Set

| Subject<br>ID | Informed<br>Consent Date | Date of First<br>ARV-471/<br>Anastrozole<br>Dose | Date of Last<br>ARV-<br>471/Anastrozole<br>Dose (Study Day) | Safety Analysis Set/<br>Ki-67 Evaluable Set/<br>Pharmacodynamic Analysis Set/<br>Pharmacokinetic Analysis set | Date of Death<br>(Study Day) | Primary Cause of Death |
|---|---|---|---|---|---|---|
| XXXX-XXX | DDMMMYYY | DDMMMYYY | DDMMMYYY (xx) | Yes/Yes/Yes | | |
| XXXX-XXX | DD <b>MMM</b> YYY | DDMMMYYY | DDMMMYYY (xx) | Yes/Yes/Yes | DDMMMYYY (xx) | Disease Progression |
| XXXX-XXX | DD <b>MMM</b> YYY | DDMMMYYY | DDMMMYYY (xx) | No/No/No | | |
| XXXX-XXX | DD <b>MMM</b> YYY | DDMMMYYY | DDMMMYYY (xx) | Yes/No/Yes/Yes | DDMMMYYY (xx) | Other: XXXXX |
| XXXX-XXX | DD <b>MMM</b> YYY | DDMMMYYY | DDMMMYYY (xx) | Yes/Yes/No/Yes | | |
| XXXX-XXX | DD <b>MMM</b> YYY | DDMMMYYY | DDMMMYYY (xx) | Yes/Yes/Yes/No | DDMMMYYY (xx) | Adverse Event |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: Full Analysis Set is defined as all enrolled participants who were randomized. Safety Analysis Set is defined as all enrolled participants who receive at least 1 dose of study intervention. Ki-67 Evaluable Set is defined as all enrolled participants who were randomized and received at least one dose of study treatment and had evaluable Ki-67 measurements other than '0' or '< 1' from baseline and evaluable Ki-67 measurements from C1D15 visits. Pharmacodynamic/Biomarker Analysis Set is defined as all enrolled participants with at least 1 of the Pharmacodynamic/Biomarkers evaluated at pre and/or post dose. PK Concentration Analysis Set includes all participants in the Safety Analysis Set who have at least one plasma concentration (including those below the limit of quantification) for ARV-471, or ARV-473.

#### **Programming Note:**

• Sorting order is by Subject ID.

# Listing 16.2.1.2 Subject Disposition Analysis Set: Enrolled Participants

Randomized Treatment: ARV-471 200 mg

| | Date of Last | | | |
|---|---|---|---|---|
| | ARV-471/Anastrozole | | Date of Study | |
| Subject | Dose (Study Day) | Reason for Treatment | Discontinuation | Reason for Study |
| ID | Dose (Study Day) | Discontinuation | (Study Day) | Discontinuation |
| XXXX-XXX | DDMMMYYY (XX) | Never Dosed | DDMMMYYY (XX) | Withdrawal of Consent: DDMMMYYY |
| XXXX-XXX | DDMMMYYY (XX) | Disease Progression per Response Criteria | DDMMMYYY (XX) | Study Terminated by Sponsor |
| XXXX-XXX | DDMMMYYY (XX) | Clinical Progression: XXXXXXXXXXXXX | DDMMMYYY (XX) | Completed study per protocol |
| XXXX-XXX | DDMMMYYY (XX) | Withdrawal of Consent: Other - XXXXXXXXXX | DDMMMYYY (XX) | Lost to Follow-up |
| XXXX-XXX | DDMMMYYY (XX) | Completed Treatment per protocol | | Death |
| XXXX-XXX | DDMMMYYY (XX) | Significant non-compliance | DDMMMYYY (XX) | Other: XXXXXXXXXXXXXXXXX |
| XXX-XXX | DDMMMYYY (XX) | Pregnancy | DDMMMYYY (XX) | Withdrawal of Consent: DDMMMYYY |
| XXX-XXX | DDMMMYYY (XX) | Death | DDMMMYYY (XX) | Study Terminated by Sponsor |
| XXX-XXX | DDMMMYYY (XX) | Adverse Event: XX, XX, XX | DDMMMYYY (XX) | Completed study per protocol |
| XXX-XXX | DDMMMYYY (XX) | Study Terminated by Sponsor | DDMMMYYY (XX) | Lost to Follow-up: DDMMMYYY |
| XXXX-XXX | DDMMMYYY (XX) | Lost to Follow-up | | Death |
| XXXX-XXX | DDMMMYYY (XX) | Other: XXXXXXXXXXXX | DDMMMYYY (XX) | Other: XXXXXXXXXXXXXXXXX |
| XXXX-XXX | DDMMMYYY (XX) | Withdrawal of Consent: Participant refused | DDMMMYYY (XX) | Withdrawal of Consent: DDMMMYYY |
| | | further study treatment/intervention, but | | |
| | | will continue to be followed | | |
| XXXX-XXX | DDMMMYYY (XX) | Withdrawal of Consent: Participant withdrawal | DDMMMYYY (XX) | Study Terminated by Sponsor |
| | | from study | | 1 1 |

Note: Enrolled Participants included all subjects who signed the Informed Consent.

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

#### **Programming Note:**

- Sorting order is by Subject ID.
- Include Screen Failure in a separated page.
- Date after Lost to Follow-up is for the date of last Know to be Alive.

Listing 16.2.2 Deviations from the Clinical Protocol Analysis Set: Full Analysis Set

| Subject<br>ID | Date of Protocol<br>Deviation (Study<br>Day) | Protocol Deviation Description | Protocol Deviation Category | Protocol<br>Deviation<br>Severity |
|---|---|---|---|---|
| XXX-XXX | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXX | Minor |
| | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor |
| | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXX | Minor |
| XXX-XXX | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor |
| XXX-XXX | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

### **Programming Note:**

• Sorting order is by Subject ID, Date of Protocol Deviation.

Listing 16.2.4.1
Demographic Characteristics
Analysis Set: Full Analysis Set

| | | | | | | | ECOG |
|---|---|---|---|---|---|---|---|
| | Year of | | | | | | Performance |
| Subject | Birth/Age | | | | Weight (kg) H | Height (cm) | Status at |
| ID | (years) | Sex/ | Ethnicity | Race | at Baseline a | at Baseline | Baseline |
| XXXX-XXX | YYYY/XX | Female | Hispanic or Latino | American Indian or Alaskan Native | XXX.X | XXX.X | 0 |
| XXXX-XXX | YYYY/XX | Female | Not Hispanic or Latino | Asian | XXX.X | XXX.X | 0 |
| XXXX-XXX | YYYY/XX | Female | Not Reported | Black or African American | XXX.X | XXX.X | 1 |
| XXXX-XXX | YYYY/XX | Female | Not Reported | Native Hawaiian or Other Pacific Islander | XXX.X | XXX.X | 1 |
| XXXX-XXX | YYYY/XX | Female | Not Hispanic or Latino | White | XXX.X | XXX.X | 1 |
| XXXX-XXX | YYYY/XX | Female | Not Hispanic or Latino | Not Reported | XXX.X | XXX.X | 1 |
| XXXX-XXX | YYYY/XX | Female | Not Hispanic or Latino | White | XXX.X | XXX.X | 0 |
| XXXX-XXX | YYYY/XX | Female | Not Reported | Other: XXXXXX | XXX.X | XXX.X | 1 |

# **Programming Note:**

• Sorting order is by Subject ID.

#### Listing 16.2.4.2 Medical History Analysis Set: Full Analysis Set

Randomized Treatment: ARV-471 200 mg

| | | | Start Date | | |
|---|---|---|---|---|---|
| | | System Organ Class/ | (Study Day)/ | | Taking |
| Subject | | Preferred Term/ | Stop Date | | Medication for |
| ID | Category | Medical Condition or Past Surgery Term | (Study Day) | CTCAE Grade | Condition? |
| XXXX-XXX | Medical Condition | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/ | Grade 1 | No |
| | | XXXXXXXXXXXXXXXXX/ | Ongoing | | |
| | | XXXXXXXXXXXXXXXXXXXX | 3 3 | | |
| | Medical Condition | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/ | Grade 2 | Yes |
| | | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx) | | |
| | | XXXXXXXXXXXXXXXXXXXX | | | |
| | Surgery | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/ | Grade 3 | Yes |
| | | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx) | | |
| | | XXXXXXXXXXXXXXXXXXX | | | |
| XXXX-XXX | Medical Condition | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/ | Grade 4 | Yes |
| | | XXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx) | | |
| | | XXXXXXXXXXXXXXXXXXX | | | |
| | Medical Condition | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | Grade 1 | No |
| | | XXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx) | | |
| | | XXXXXXXXXXXXXXXXXXX | | | |
| | Medical Condition | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | Grade 2 | Yes |
| | | XXXXXXXXXXXXXXXXX/ | Ongoing | | |
| | | XXXXXXXXXXXXXXXXXXX | | | |
| | Medical Condition | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | Grade 1 | Yes |
| | | XXXXXXXXXXXXXXXXXXX/ | Ongoing | | |
| | | XXXXXXXXXXXXXXXXXXX | | | |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: Medical Condition/Past Surgery was coded with MedDRA version 24.1.

#### **Programming Note:**

Sorting order is by Subject ID, System Organ Class, Preferred Term.

Listing 16.2.4.3
Disease Staging - Initial Diagnosis
Analysis Set: Full Analysis Set

| Subject<br>ID | Date of Initial<br>Diagnosis<br>(Study Day) | Primary<br>Diagnosis | Disease Stage<br>at Initial<br>Diagnosis | Primary Tumor/<br>Regional Lymph Node/<br>Distant Metastasis | Histopathological<br>Classification | Histopathological<br>Grade |
|---|---|---|---|---|---|---|
| XXXX-XXX | DDMMMYYY (xx) | ER+ HER2- BC | Stage 0 | TX/cNX/Unknown | In-Situ Carcinoma | Grade 1 |
| XXXX-XXX | DDMMMYYY (xx) | ER+ HER2- BC | Stage IA | T0/cN0/M0 | Invasive Ductal Carcinoma | Grade 3 |
| XXXX-XXX | DDMMMYYY (xx) | ER+ HER2- BC | Stage IB | Tis/cN1/M1 | Invasive Lobular Carcinoma | Grade 1 |
| XXXX-XXX | DDMMMYYY (xx) | ER+ HER2- BC | Stage IIA | T1mi/cN2a/M0 | Invasive Carcinoma NOS | Grade x |
| XXXX-XXX | DDMMMYYY (xx) | ER+ HER2- BC | Stage IIB | Tla/cN2b/M0 | Invasive Mucinous | Grade 1 |
| XXXX-XXX | DDMMMYYY (xx) | ER+ HER2- BC | Stage IIIA | T1b/cN2c/M0 | Adenocarcinoma | Grade 2 |
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Unknown | T1c/cN3c/M1 | Other: XXXXXXX | Grade 1 |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: BC = Breast Cancer.

#### **Programming Note:**

• Sorting order is by Subject ID

Listing 16.2.4.4
Disease Staging - Current Diagnosis
Analysis Set: Full Analysis Set

| Subject<br>ID | Date of Current<br>Staging<br>(Study Day) | Primary<br>Diagnosis | Disease Stage<br>at Initial<br>Diagnosis | Primary Tumor/<br>Regional Lymph Node/<br>Distant Metastasis | Histopathological<br>Classification/<br>Histopathological Grade | Imaging<br>Modality/<br>Planned Type<br>of Surgery |
|---|---|---|---|---|---|---|
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Stage 0 | TX/cNX/Unknown | In-Situ Carcinoma/1 | CT/Mastectomy |
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Stage IA | T0/cN0/M0 | Invasive Ductal Carcinoma/3 | MRI/Mastectomy |
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Stage IB | Tis/cN1/M1 | Invasive Lobular Carcinoma/2 | Ultrasound/BCS |
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Stage IIA | T1mi/cN2a/M0 | Invasive Carcinoma NOS/2 | Mammogram/BCS |
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Stage IIB | T1a/cN2b/M0 | Invasive Mucinous/1 | PET-CT/BCS |
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Stage IIIA | T1b/cN2c/M0 | Adenocarcinoma/1 | PET-MRI/BCS |
| XXXX-XXX | DDMMMYYY(xx) | ER+ HER2- BC | Unknown | T1c/cN3c/M1 | Other: XXXXXXX/X | CT/BCS |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: BC = Breast Cancer; BCS = Breast conserving surgery.

#### **Programming Note:**

• Sorting order is by Subject ID

Listing 16.2.4.5 Molecular Biology of Disease Analysis Set: Full Analysis Set

| Subject<br>ID | Analyte/<br>Biomarker | Date of<br>Collection<br>(Study Day) | Specimen<br>Type | Sample Site | Analytical<br>Method/Result | Quantitative<br>Parameter | Quantitative<br>Result (%) |
|---|---|---|---|---|---|---|---|
| XXXX-XXX | HER2 | DDMMMYYY (xx) | Tumor tissue | Breast | IHC/1+ | | |
| | KI67 | DDMMMYYY (xx) | Tumor tissue | Lymph Node | | Tumor cells | XX.X |
| | Estrogen receptor | DDMMMYYY (xx) | Tumor tissue | Other: XXXXX | | Tumor cells | XX.X |
| | Progesterone receptor | DDMMMYYY (xx) | Tumor tissue | Breast | | Tumor cells | XX.X |
| XXXX-XXX | HER2 | DDMMMYYY (xx) | Tumor tissue | Breast | ISH/Negative | | |
| | KI67 | DDMMMYYY (xx) | Tumor tissue | Breast | | Tumor cells | XX.X |
| | Estrogen receptor | DDMMMYYY (xx) | Tumor tissue | Other: XXXXX | | Tumor cells | XX.X |
| | Progesterone receptor | DDMMMYYY (xx) | Tumor tissue | Other: XXXXX | | Tumor cells | XX.X |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. \* indicates the baseline value.

#### **Programming Note:**

Sorting order is by Subject ID, Analyte/Biomarker, Date of Collection.

Include data in 'Molecular Biology of Disease - HER2 Status' and 'Molecular Biology of Disease - Hormone Receptor/KI67 Status'

Listing 16.2.4.6
Prior and Concomitant Medications
Analysis Set: Full Analysis Set

| | | ATC Category II/ | Start Date (Study Day)/ | | | |
|---|---|---|---|---|---|---|
| | Prior or | Preferred Name/ | | Dose/ | Frequency/ | |
| Subject | Concomitant | Medication Name | Stop Date (Study Day) | | Route | |
| ID | | | | Unit | | Use |
| XXX-XXX | Prior | XXXXXXXXXXXXX/ | DDMMMYYY (XX)/ | XX/ | TID/ AE:#1, # | |
| | | XXXXXXXXXXXX/ | Ongoing | Capsule | Oral | |
| | | XXXXXXXXXXXXXX | | | | |
| | Concomitant | XXXXXXXXXXXXX/ | DDMMMYYY (XX)/ | XX/ | QIS/ | MH |
| | | XXXXXXXXXXXX/ | DDMMMYYY (XX) | Gram | Intramuscular | |
| | | XXXXXXXXXXXXXX | | | | |
| | Concomitant | XXXXXXXXXXXXX/ | DDMMMYYY (XX)/ | XX/ | BID/ | MH |
| | | XXXXXXXXXXXX/ | DDMMMYYY (XX) | Microgram | Subcutaneous | |
| | | XXXXXXXXXXXXXX | | | | |
| XXX-XXX | Concomitant | XXXXXXXXXXXXX/ | DDMMMYYY (XX)/ | XX/ | UNKNOWN / | AE:#1 |
| | | XXXXXXXXXXXX/ | DDMMMYYY (XX) | Spray | Topical | |
| | | XXXXXXXXXXXXXX | | | | |
| | Concomitant | XXXXXXXXXXXXX/ | DDMMMYYY (XX)/ | XX/ | Other: XXX/ | Prophylaxis |
| | | XXXXXXXXXXXX/ | DDMMMYYY (XX) | Other: XXXX | Unknown | |
| | | XXXXXXXXXXXXXX | | | | |
| XXX-XXX | Prior | XXXXXXXXXXXXX/ | DDMMMYYY (XX)/ | XX/ | QAM/ | Other: XXXXX |
| | | XXXXXXXXXXXX/ | DDMMMYYY (XX) | Tablet | Other: XXXX | |
| | | XXXXXXXXXXXXXX | | | | |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

Note: Prior and Concomitant Medications are coded with WHODRUG Global B3 Sep 2022.

Note: Prior medications include non-study drug medications that are ended before Day 1. Concomitant medications include non-study drug medications that are used/started on/after Day 1 and within 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

#### **Programming Note:**

• Sorting order is by Subject ID, Prior or Concomitant, ATC Category II, Preferred Name

Listing 16.2.5.1 Study Drug Exposure and Compliance Analysis Set: Safety Analysis Set

Treatment: ARV-471 200 mg

| | Duration of<br>Treatment | | Absolute Dose<br>Intensity | Intensity | | | Number | Number |
|---|---|---|---|---|---|---|---|---|
| Subject | (week) | Cumulative | (mg/week) | (%) | Total Planned | Compliance | of Doses | of Doses |
| ID | | Dose (mg) | | | Dose (mg) | (응) | Interrupted | Reduced |
| XXX-XXX | XX.X | XX | XX.X | XX.X | XX | XX.X | XXX | XXX |
| XXXX-XXX | XX.X | XX | XX.X | XX.X | XX | XX.X | XXX | XXX |
| XXX-XXX | XX.X | XX | XX.X | XX.X | XX | XX.X | XXX | XXX |

Note: Duration of treatment (week) is defined as the time from the date of first dose to the date of last dose. Cumulative dose (mg) is the sum of 'Actual total daily dose' × (End date- Start date+1) per record. Total planned dose (mg) is the sum of 'Planned total daily dose' × (End date- Start date+1) per record. Compliance is 100\*(Cumulative dose/Total planned dose), accounting for planned dose modifications and interruptions. Absolute dose intensity (mg/week) is (Cumulative Dose (mg))/(Duration of Treatment (week)). Relative dose intesity (%) is (Absolute Dose Intensity (mg/week))/(Initial Planned Weekly Dose (mg/week), 1400 for ARV-471 and 7 for Anastrozole)).

## **Programming Note:**

• Sorting order is by Subject ID.

#### Listing 16.2.5.2 Study Drug Administration Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| | | | | | Actual | Action Taken | |
|---|---|---|---|---|---|---|---|
| | | | Start Date | End Date | Total Daily | Regarding Dose | |
| Subject | Planned Total | Route/ | (Study Day) | (Study Day) | Dose/Unit | Administration? | Reason for Dose |
| ID | Daily Dose/Unit | Frequency | | | | | Adjustment |
| XXXX-XXX | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | No action taken | |
| | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | Interrupted | Other: XXXX |
| | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | Discontinued | AE: #x |
| | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | Reduced | Missed dose |
| | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | No action taken | |
| XXXX-XXX | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | Interrupted | Medication error |
| | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | No action taken | |
| | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | No action taken | |
| | xx/XXXX | Oral/QD | DDMMMYYY (XX) | DDMMMYYY (XX) | xx/XXXX | Increased | |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: AE = Adverse Event; Missed dose = Participant missed/Skipped dose.

#### **Programming Note:**

• Sorting order is by Subject ID, Start date.

Listing 16.2.5.3
PK Dosing - ARV-471
Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| | | | | | | | Vomit within | |
|---|---|---|---|---|---|---|---|---|
| | | Reference Time | | Start Date Time | Actual<br>Dose | Dose Taken | 6 Hours<br>After | Post Dose<br>Vomiting Start |
| Subject | Visit | Point | Route/ | (Study Day) | (mg) | with Food? | Dosing? | Date Time |
| ID | | | Frequency | 7 | | | | |
| XXXX-XXX | C1D15 | Prior dose | Oral/QD | DDMMMYYY HH:MM(XX) | XXX | No | No | |
| | C2D1 | Prior dose | Oral/QD | DDMMMYYY HH:MM(XX) | XXX | No | Yes/AE#XXX | DDMMMYYY HH:MM |
| | C6D18 | Prior dose | Oral/QD | DDMMMYYY HH:MM(XX) | XXX | No | No | |
| XXXX-XXX | C1D15 | In clinic dose | Oral/QD | DDMMMYYY HH:MM(XX) | XXX | Yes | No | |
| | C2D1 | In clinic dose | Oral/QD | DDMMMYYY HH:MM(XX) | XXX | No | Yes/AE#XXXX | DDMMMYYY HH:MM |
| | C6D18 | In clinic dose | Oral/QD | DDMMMYYY HH:MM(XX) | XXX | Yes | No | |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

#### **Programming Note:**

• Sorting order is by Subject ID, Start Date.

Listing 16.2.5.4

ARV-471 and ARV-473 Plasma Concentration

Analysis Set: PK Analysis Set

| Subject | | | Collection Date Tir | ne | | | |
|---|---|---|---|---|---|---|---|
| ID | Test (unit) | Visit | (Study Day) | Time Point | Result | Comments | Flag[1] |
| XXXX-XXX | ARV-471 (unit) | C1D15 | DDMMMYYYY HH:MM (XX | () Pre-biopsy | XXX.X | | |
| | | C2D1 | DDMMMYYYY HH:MM (XX | () Pre-dose | XXX.X | | a |
| | | | DDMMMYYYY HH:MM (XX | () 1 hour (± 15 min) post-dose | XXX.X | | |
| | | | DDMMMYYYY HH:MM (XX | () 2 hours (± 15 min) post-dose | XXX.X | XXXXXX | |
| | | | DDMMMYYYY HH:MM (XX | (4 hours (± 30 min) post-dose | XXX.X | | |
| | | C6D18 | DDMMMYYYY HH:MM (XX | () pre-surgery | XXX.X | | С |

ARV-473 (unit)

XXXX-XXX

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.
[1] a: Pre-dose samples are collected after dosing time. b: Post-dose samples are collected out of time window on Cycle 2 Day 1. c: When ARV-471 dose is different from planned dose.

# **Programming Note:**

• Sorting order is by Subject ID, Test, Visit.

Listing 16.2.6.1
Efficacy Parameters - Part 1 of 2
Analysis Set: Full Analysis Set

| | | Actual/Random | % of Tumor | | | | | Percentage |
|---|---|---|---|---|---|---|---|---|
| | Ki-67 | iztion Size | cells with Ki67 | Ki-67 Expression | Ratio of Ki-67 | Percentage Change | mPEPI Score | Change (%) of |
| | Evaluable | of Primary | Local/Central/R | (%) at Baseline/ | between | (%) of Ki-67 at | at Baseline/ | PR H-score at |
| Subject | Analysis | Breast Tumor | andomization | C1D15/Surgery | C1D15/Surgery | C1D15/Surgery | after | C1D15/Surgery |
| ID | Set | (cm) | | | and Baseline | from Baseline | Treatment | from Baseline |
| XXXX-XXX | Yes | ≤2/≤2 | <20%/≥20%/<20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | >3/0 | XX.X/XX.X |
| XXXX-XXX | Yes | >2to<5/>2to<5 | ≥20%/<20%/<20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | 1~2/0 | XX.X/XX.X |
| XXXX-XXX | Yes | ≥5/≥5 | <20%/<20%/<20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | 3/1~2 | XX.X/XX.X |
| XXXX-XXX | Yes | ≤2/≤2 | ≥20%/≥20%/≥20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | >3/1~2 | XX.X/XX.X |
| XXXX-XXX | Yes | >2to<5 | ≥20%/≥20%/≥20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | 0/0 | XX.X/XX.X |
| XXXX-XXX | Yes | ≥5/>2to<5 | ≥20%/≥20%/≥20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | 1~2/0 | XX.X/XX.X |
| XXXX-XXX | Yes | ≤2/≤2 | <20%/<20%/<20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | 3/0 | XX.X/XX.X |
| XXXX-XXX | No | >2to<5/≥5 | ≥20%/≥20%/≥20% | XX.X/XX.X/XX.X | XX.X/XX.X | XX.X/XX.X | >3/1~2 | XX.X/XX.X |

Note: mPEPI = Modified Pre-operative Endocrine Prognostic Index.

Note: Ratio of Ki-67 between C1D15/Surgery and baseline =  $\log(\text{Ki-67 at C1D15/Surgery}) - \log(\text{Ki-67 at baseline})$ , the variable for the primary endpoint.

Note: Ki-67 Percentage Change from Baseline at C1D15/Surgery =  $100 \times (\text{Ki-}67 \text{ at C1D15/Surgery} - \text{Ki-}67 \text{ at baseline}) / \text{Ki-}67 \text{ at baseline}$ 

## **Programming Note:**

• Sorting order is by Subject ID.

Listing 16.2.6.2
Efficacy Parameters - Part 2 of 2
Analysis Set: Full Analysis Set

| | | | | | | Caliper | Complete | Percentage |
|---|---|---|---|---|---|---|---|---|
| | Ki-67 | Actual/Random | % of Tumor cells | Post-Surgery | | Based Best | Cycle Cell | Change (%) of ER |
| | Evaluable | iztion Size | with Ki67 | Pathological | Breast | Percentage | Arrest at | AQUA score at |
| Subject | Analysis | of Primary | Local/Central/RaF | Response/Derived | d Conserving | Change from | Week | C1D15/Surgery |
| ID | Set | Breast Tumor | ndomization | Response | Surger | Baseline (%) | 2/Surgery | from Baseline |
| XXXX-XXX | Yes | ≤2/≤2 | <20%/≥20%/<20% | pCR/pCR | Yes | XX.X | Yes/Yes | XX.X/XX.X |
| XXXX-XXX | Yes | >2to<5/>2to<5 | ≥20%/<20%/<20% | pPR/non-pCR | No | XX.X | Yes/Yes | XX.X/XX.X |
| XXXX-XXX | Yes | ≥5/≥5 | <20%/<20%/<20% | pPR/pCR | Yes | XX.X | No/Yes | XX.X/XX.X |
| XXXX-XXX | Yes | ≤2/≤2 | ≥20%/≥20%/≥20% | pCR/pCR | Yes | XX.X | Yes/No | XX.X/XX.X |
| XXXX-XXX | Yes | >2to<5 | ≥20%/≥20%/≥20% | pPR/non-pCR | Yes | XX.X | Yes/Yes | XX.X/XX.X |
| XXXX-XXX | Yes | ≥5/>2to<5 | ≥20%/≥20%/≥20% | pPR/non-pCR | Yes | XX.X | No/Yes | XX.X/XX.X |
| XXXX-XXX | Yes | ≤2/≤2 | <20%/<20%/<20% | pCR/non-pCR | No | XX.X | Yes/Yes | XX.X/XX.X |
| XXXX-XXX | No | >2to<5/≥5 | ≥20%/≥20%/≥20% | NR/non-pCR | Yes | XX.X | Yes/Yes | XX.X/XX.X |

Note: pCR = Pathological Complete Response.

Note: Complete cycle cell arrest at Week 2/Surgery is defined as Ki67 score ≤ 2.7%.

Note: Percentage Change (%) of ER at C1D15/Surgery from Baseline 100 × (ER AQUA at C1D15/surgery - ER AQUA at

baseline)/ER AQUA at baseline.

# **Programming Note:**

• Sorting order is by Subject ID.

Listing 16.2.6.3 Target Lesion (TL) Analysis Set: Full Analysis Set

| | | | Date of | | | Sum of Primary | % Change from |
|---|---|---|---|---|---|---|---|
| Subject | Baseline | Assessment | Assessment | Sum of TL | % Change from | Tumor TL | Baseline of |
| ID | Tumor Size | Timepoint | (Study Day) | (mm) | Baseline of TL | (mm) | Primary Tunor TL |
| XXXX-XXX | ≤2 cm | Screen | DDMMMYYY (XX) | XXX | | XXX | |
| | | Cycle 1 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X |
| | | Cycle 2 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X* |
| | | Cycle 3 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X |
| | | Cycle 4 | DDMMMYYY (XX) | XXX | XX.X* | XXX | XX.X |
| | | Cycle 5 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X |
| | | Cycle 6 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X |
| XXXX-XXX | ≤2 cm | Screen | DDMMMYYY (XX) | XXX | | XXX | |
| | | Cycle 1 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X |
| | | Cycle 2 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X |
| | | Cycle 3 | DDMMMYYY (XX) | XXX | XX.X | XXX | XX.X* |
| | | Cycle 4 | DDMMMYYY (XX) | XXX | XX.X* | XXX | XX.X |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: Best percentage change of TL from baseline (indicated with \*) is maximum decrease or minimum increase if no decrease being observed.

#### **Programming Note:**

• Sorting order is by Subject ID, Date of Assessment

Listing 16.2.6.4 Primary Breast Tumor Change - Caliper-based
Analysis Set: Full Analysis Set

| Subject | Baseline | | Date of Assessment (Study Day) | Primary Breast<br>Tumor (mm) | % Change | Best % Change from Baseline ? |
|---|---|---|---|---|---|---|
| ID | Tumor Size | Assessment Timepoint | (Beddy Ddy) | ramor (mm) | from Baseline | TIOM DUSCIING . |
| XXXX-XXX | ≤2 cm | Screen | DDMMMYYY (XX) | XXX | | |
| | | Cycle 1 | DDMMMYYY (XX) | XXX | XX.X | |
| | | Cycle 2 | DDMMMYYY (XX) | XXX | XX.X | |
| | | Cycle 3 | DDMMMYYY (XX) | XXX | XX.X | |
| | | Cycle 4 | DDMMMYYY (XX) | XXX | XX.X | Yes |
| | | Cycle 5 | DDMMMYYY (XX) | XXX | XX.X | |
| | | Cycle 6 | DDMMMYYY (XX) | XXX | XX.X | |
| XXXX-XXX | ≤2 cm | Screen | DDMMMYYY (XX) | XXX | | |
| | | Cycle 1 | DDMMMYYY (XX) | XXX | XX.X | |
| | | Cycle 2 | DDMMMYYY (XX) | XXX | XX.X | |
| | | Cycle 3 | DDMMMYYY (XX) | XXX | XX.X | |
| | | Cycle 4 | DDMMMYYY (XX) | XXX | XX.X | Yes |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: Best percentage change from baseline is maximum decrease or minimum increase if no decrease being observed.

#### **Programming Note:**

• Sorting order is by Subject ID, Date of Assessment

Listing 16.2.6.5 Tumor Biopsy Analysis Set: Full Analysis Set

| Subject | | | Collection Date | Result/<br>% Change from | | Location/ |
|---|---|---|---|---|---|---|
| ID | Test (SI unit) | Visit | (Study Day) | Baseline | Interpretation | Method |
| XXXX-XXX | Ki-67 (%) | Screening | DDMMMYYYY (XX) | XX.X* | Positive | Breast/IHC |
| | | C1D15 | DDMMMYYYY (XX) | XX.X/XX.X | Intermediate Proliferation Rate | Breast/IHC |
| | | C6D18 | DDMMMYYYY (XX) | XX.X/XX.X | High Proliferation Rate | Unknown/IHC |
| | <insert (xxx)=""></insert> | Screening | DDMMMYYYY (XX) | XX.X* | High Proliferation Rate | Breast/IHC |
| | | C1D15 | DDMMMYYYY (XX) | XX.X/XX.X | Intermediate Proliferation Rate | Breast/IHC |
| | | C6D18 | DDMMMYYYY (XX) | XX.X/XX.X | Positive | Breast/IHC |
| | | Unscheduled | DDMMMYYYY (XX) | XX.X/XX.X | Positive | Breast/IHC |
| XXXX-XXX | Ki-67 (%) | Screening | DDMMMYYYY (XX) | XX.X* | High Proliferation Rate | Other:XX/IHC |
| | | C1D15 | DDMMMYYYY (XX) | Uninterpretable | Uninterpretable | Breast/IHC |
| | | C6D18 | DDMMMYYYY (XX) | XX.X/XX.X | Positive | Breast/IHC |
| | | Unscheduled | DDMMMYYYY (XX) | XX.X/XX.X | Positive | Breast/IHC |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

Note: IHC = Immunohistochemistry. Note: \* indicates baseline value.

#### **Programming Note:**

• Sorting order is by Subject ID, Test, Collection date

Listing 16.2.6.6 Imaging Response Assessment - mRECIST Analysis Set: Full Analysis Set

| Subject | Assessment | Date of Assessment | Target Lesion | Non-Target Lesion | Any New | Response at this |
|---|---|---|---|---|---|---|
| ID | Timepoint | (Study Day) | Response | Response | Lesions? | Timepoint |
| XXXX-XXX | Cycle 1 | DDMMMYYY (XX) | Partial Response | Non-CR/Non-PD | No | Partial Response |
| | Cycle 2 | DDMMMYYY (XX) | Partial Response | Non-CR/Non-PD | No | Partial Response |
| | Cycle 3 | DDMMMYYY (XX) | Partial Response | Non-CR/Non-PD | No | Partial Response |
| | Cycle 4 | DDMMMYYY (XX) | Partial Response | Non-CR/Non-PD | Yes | Progressive Disease |
| | Cycle 5 | DDMMMYYY (XX) | Progressive Disease | Not Evaluable | Yes | Progressive Disease |
| | Pre-Surgery | DDMMMYYY (XX) | | | | |
| XXXX-XXX | Cycle 1 | DDMMMYYY (XX) | Stable Disease | Not Evaluable | No | Stable Disease |
| | Cycle 2 | DDMMMYYY (XX) | Stable Disease | Not Evaluable | No | Stable Disease |
| | Cycle 3 | DDMMMYYY (XX) | Not Evaluable | Complete Response | No | Not Evaluable |
| | Cycle 4 | DDMMMYYY (XX) | Complete Response | Complete Response | No | Complete Response |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

#### **Programming Note:**

• Sorting order is by Subject ID, Date of Procedure

Listing 16.2.6.7 Cytology Results Analysis Set: Full Analysis Set

| Subject<br>D | Date Sample<br>Collected (Study Day) | Specimen Type | Findings |
|---|---|---|---|
| XXX-XXX | DDMMMYYY (XX) | Pleural Effusion | Benign |
| | DDMMMYYY (XX) | Abdominal/Pelvic Ascites | Atypical |
| XXX-XXX | DDMMMYYY (XX) | Other: XXXXXXXXX | Suspicious |
| | DDMMMYYY (XX) | DDMMMYYY (XX) | Malignant |
| XXX-XXX | DDMMMYYY (XX) | DDMMMYYY (XX) | Other: XXXXXXX |
| | DDMMMYYY (XX) | DDMMMYYY (XX) | Benign |
| | DDMMMYYY (XX) | DDMMMYYY (XX) | Atypical |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

#### **Programming Note:**

• Sorting order is by Subject ID, Date Sample Collected

Listing 16.2.6.8 Disease Staging - Post-Surgery Analysis Set: Full Analysis Set

| | Ki-67 | Date of Tumor | | Multiple Foci | _ | | Lymphatic<br>Vascular Invasion |
|---|---|---|---|---|---|---|---|
| Subject | Evaluable | Tissue Collected | Pathologic | of Residual | Lymph Nodes - | Distant | Classification |
| ID | Analysis Set | (Study Day) | Tumor - ypT | Tumor? | урN | Metastasis ypT | |
| XXXX-XXX | Yes | DDMMMYYY (XX) | урТх | No | УрИХ | MO | Present |
| XXXX-XXX | Yes | DDMMMYYY (XX) | ypT0 | No | ypN0 | pM1 | Not Present |
| XXXX-XXX | Yes | DDMMMYYY (XX) | ypTis | No | ypN0(i+) | Unknown | Unknown |
| XXXX-XXX | Yes | DDMMMYYY (XX) | ypT1mi | Yes | <pre>ypN0 (mol+)</pre> | MO | Not Present |
| XXXX-XXX | Yes | DDMMMYYY (XX) | ypT1a | Yes | ypN1 | MO | Not Present |
| XXXX-XXX | Yes | DDMMMYYY (XX) | ypT1b | Yes | ypN1mi | MO | Not Present |
| XXXX-XXX | Yes | DDMMMYYY (XX) | ypT1c | No | ypN1a | MO | Not Present |
| XXXX-XXX | No | DDMMMYYY (XX) | урТ2 | No | ypN1b | Unknown | Not Present |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

#### **Programming Note:**

• Sorting order is by Subject ID, Date of Procedure

Listing 16.2.7.1

Adverse Events by Subject

Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| | | Start Date | Serious?/ | | Related to | Outcome/ |
|---|---|---|---|---|---|---|
| | | (StudyDay)/ | Toxicity | Relation to | Concomitant | Concomitant |
| | System Organ Class/ | Stop Date | Grade/ | Study Drug/ | Medication? | Medication Given/ |
| Subject | Preferred Term/ | (StudyDay)/ | Lead to Study | Action Taken | / | Non-drug |
| ID | Verbatim | TEAE? | Discontinued | with Study Drug | Specify | Treatment Given? |
| XXXX-XXX | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/ | Not Related/ | No | RED/ |
| | XXXXXXXXXXXXXXXXX/ | Ongoing/ | 2/ | Dose Not Change | ed | No/ |
| | XXXXXXXXXXXXXXXXXXXXXX | No | No | | | Yes |
| | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | Yes/ | Related/ | | NRED/ |
| | XXXXXXXXXXXXXXXXX/ | Ongoing/ | 4/ | Dose Reduced | | Yes/ |
| | XXXXXXXXXXXXXXXXXXXXXX | Yes | No | | | No |
| XXXX-XXX | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | Yes/ | Not Related / | Yes/ | REDWSEQ/ |
| | XXXXXXXXXXXXXXXXX/ | DDMMMYYY(xx)/ | 1/ | Drug Withdrawn | n XXXX, XXXX | X No/ |
| | XXXXXXXXXXXXXXXXXXXXXX | Yes | No | | | No |
| | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | No/ | Not Related / | No | Fatal/ |
| | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | 5/ | Not Applicable | 9 | Yes/ |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes | Yes | | | Yes |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: Adverse events (AE) were evaluated based on NCI-CTCAE (version 5.0), and coded with MedDRA Version 24.1. Note: A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV-471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Note: RED=Recovered/Resolved; NRED=Not Recovered/Not Resolved; REDWSEQ=Recovered/Resolved with Sequelae; REING=Recovering/Resolving.

#### **Programming Note:**

• Sorting order is by Subject ID, Start Date, System Organ Class and Preferred Term.

Listing 16.2.7.2 Serious Adverse Events by Subject Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| Subject ID Age/Race/ Sex | System Organ Class/<br>Preferred Term/<br>Verbatim | Start Date<br>(StudyDay)/<br>Stop Date<br>(StudyDay)/<br>TEAE? | Serious?/ Toxicity Grade/ Lead to Study Discontinued | Relation to<br>Study Drug/<br>Action Taken<br>with Study Drug | Related to<br>Concomitant<br>Medication?/<br>Specify | Outcome/<br>Concomitant<br>Medication Given/<br>Non-drug<br>Treatment Given? |
|---|---|---|---|---|---|---|
| XXXX-XXX/<br>XX/W/F | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYY (xx)/<br>Ongoing/<br>No | Yes/<br>2/<br>No | Not Related/<br>Dose Not Changed | No | RED/<br>No/<br>Yes |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>Ongoing/<br>Yes | Yes/<br>4/<br>No | Related/<br>Dose Reduced | | NRED/<br>Yes/<br>No |
| XXXX-XXX/<br>XX/B/M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY(xx)/<br>Yes | Yes/<br>1/<br>No | Not Related /<br>Drug Withdrawn | Yes/<br>XXXX,XXXXX | REDWSEQ/<br>No/<br>No |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY (xx)/<br>Yes | Yes/<br>5/<br>Yes | Not Related /<br>Not Applicable | No | Fatal/<br>Yes/<br>Yes |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: Adverse events (AE) were evaluated based on NCI-CTCAE (version 5.0), and coded with MedDRA Version 24.1. Note: A TEAE is an AE that emerges or worsens (ie increase in CTCAE grade) on/after the first dose of ARV-471/Anastrozole to 30 days from the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).

Note: RED=Recovered/Resolved; NRED=Not Recovered/Not Resolved; REDWSEQ=Recovered/Resolved with Sequelae; REING=Recovering/Resolving.

Note: N = American Indian or Alaskan Native; A = Asian; B = Black or African American; H = Native Hawaiian or Other Pacific Islander; W= White; NR = Not Reported; O= Other; M = Male; F = Female.

#### **Programming Note:**

• Sorting order is by Subject ID, Start Date, System Organ Class and Preferred Term.

Subject ID/Age/Race/Sex, Preferred Term, Treatment Arm, Onset Day, Grade, Investigator-Assessed Relatedness

Display order by treatment arm ARV-471 200mg first, then follow by Anastrozole 1mg

#### Listing 16.2.8.1 Hematology Tests with CTCAE Grade ≥ 3 Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| | | | | | Reference | | |
|---|---|---|---|---|---|---|---|
| | | | | Result/ | Reference | Range | CTCAE |
| Subject | | | Collection Date Time | Change from Baseline/ | Range | Indicator | Grade |
| ID | Test (SI unit) | Visit | (Study Day) | % Change from Baseline | | | |
| XXXX-XXX | Hemoglobin (g/L) | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XXX,XXX | Low | 1 |
| | | C1D1 | DDMMMYYYY HH:MM (XX) | XX.X* | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X/XX.X | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | |
| | <insert></insert> | | | | | | |

XXXX-XXX

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

#### **Programming Note:**

- Sorting order is by Subject ID, Test, Collection date
- if a subject has a test with CTCAE grade>=3, all visits of the test will be listed.

**Programming note**: Repeat Listing 16.2.8.1 for the following listings

Listing 16.2.8.2 Clinical Chemistry Tests with CTCAE Grade ≥ 3
Analysis Set: Safety Analysis Set

Listing 16.2.8.3
Hematology Tests
Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| | | | | | | Reference | |
|---|---|---|---|---|---|---|---|
| Subject | | | Collection | Result/ | Reference | Range | CTCAE |
| ID | Test (SI unit) | Visit | Date(Study Day) | Change from Baselin/ | Range | Indicator | Grade |
| XXXX-XXX | Hemoglobin (g/L) | Screening | DDMMMYYYY (XX) | XX.X | XXX,XXX | Low | 1 |
| | | C1D1 | DDMMMYYYY (XX) | XX.X* | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY (XX) | XX.X/XX.X | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | |

<insert>

XXXX-XXX

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

#### **Programming Note:**

• Sorting order is by Subject ID, Test, Collection date

**Programming note**: Repeat Listing 16.2.8.3 for the following listings

Listing 16.2.8.4 Clinical Chemistry Tests Analysis Set: Safety Analysis Set

Listing 16.2.8.5 Coagulation Tests Analysis Set: Safety Analysis Set Listing 16.2.8.6
Urinalysis
Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| Subject | | | Collection Date | Result |
|---|---|---|---|---|
| ID | Test | Visit | (Study Day) | (unit, if applicable) |
| XXXX-XXX | Clarity | Screening | DDMMMYYYY (XX) | Trace |
| | | C1D1 | DDMMMYYYY (XX) | 1+* |
| | | C1D8 | DDMMMYYYY (XX) | 2+ |
| | | <insert></insert> | | |
| | <insert></insert> | | | |

XXXX-XXX

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: \* indicates baseline value.

#### Programming Note:

• Sorting order is by Subject ID, Test, Visit.

Listing 16.2.9
Vital Signs
Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| Subject | | | Vital Signs Date | Result/ |
|---|---|---|---|---|
| ID | Test (SI unit) | Visit | (Study Day) | Change from Baseline |
| XXXX-XXX | Diastolic Blood Pressure (mmHg) | Screening | DDMMMYYYY (XX) | XX.X |
| | | C1D1 | DDMMMYYYY (XX) | XX.X* |
| | | C1D8 | DDMMMYYYY (XX) | XX.X/XX.X |
| | | <insert></insert> | | |
| | <insert></insert> | | | |

XXXX-XXX

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: \* indicates baseline value.

#### **Programming Note:**

- Sorting order is by Subject ID, Test, Visit.
- If Clinical provides a list of any parameter deemed significant, list the parameter of all visits of the patient

Listing 16.2.10
12-Lead ECG
Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| | | | ECG Date Time | | Test | |
|---|---|---|---|---|---|---|
| Subject<br>ID | Test (unit) | Visit | (Study Day) | Time Point | Number | Result |
| XXXX-XXX | Heart Rate (beats per minute) | Screening | DDMMMYYYY HH:MM (XX) | Screening | | XXX.X |
| | | C1D1 | DDMMMYYYY HH:MM (XX) | Predose | 1 | XXX.X |
| | | | DDMMMYYYY HH:MM (XX) | Predose | 2 | XXX.X |
| | | | DDMMMYYYY HH:MM (XX) | Predose | 3 | XXX.X |
| | | | DDMMMYYYY HH:MM (XX) | 4hr post dose | 1 | XXX.X |
| | | | DDMMMYYYY HH:MM (XX) | 4hr post dose | 2 | XXX.X |
| | | | DDMMMYYYY HH:MM (XX) | 4hr post dose | 3 | XXX.X |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | Predose | 1 | XXX.X |
| | | | DDMMMYYYY HH:MM (XX) | Predose | 2 | XXX.X |
| | | <insert></insert> | | | | |

XXXX-XXX

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1.

# **Programming Note:**

• Sorting order is by Subject ID, Test, Visit.

#### Listing 16.2.11 ECOG Performance Status Analysis Set: Safety Analysis Set

Actual Treatment: ARV-471 200 mg

| | ECOG Performance Status | | | |
|---|---|---|---|---|
| Subject | performed? | | ECOG Assessment Date | ECOG Performance |
| ID | | Visit | (Study Day) | Status |
| XXXX-XXX | Yes | Screening | DDMMMYYYY (XX) | 0 |
| | Yes | C1D1* | DDMMMYYYY (XX) | 0 |
| | Yes | C1D8 | | |
| | Yes | <insert></insert> | | |
| XXXX-XXX | No | | | |

Note: Day 1 is the date of first ARV-471/anastrozole dose. Study Day = Assessment Date - Date of Day 1 + 1 for assessment dates on or after date of Day 1. Study Day = Assessment Date - Date of Day 1 for assessment prior to Day 1. Note: \* indicates baseline value.

#### **Programming Note:**

• Sorting order is by Subject ID, Visit.

# DocuSign<sup>®</sup>

#### **Certificate Of Completion**

Envelope Id: E933EC7AAB2A4B90A40BC8D8FC42EFC6

Subject: Complete with Docusign: ARV-471-BC-201 Statistical Analysis Plan 3.pdf, ARV-471-BC-201 TLF\_shel...

Source Envelope:

Document Pages: 175 Certificate Pages: 5 AutoNav: Enabled

Envelopeld Stamping: Disabled Time Zone: (UTC) Monrovia, Reykjavik

Signatures: 4 Initials: 0

**Envelope Originator:** 

Status: Completed

Inc 2700 Wycliff Road, Suite 340

Raleigh, NC 27607

IP Address:

Sent: 15-Nov-2024 | 15:11 Viewed: 15-Nov-2024 | 15:16

Signed: 15-Nov-2024 | 15:20

#### **Record Tracking**

Status: Original

15-Nov-2024 | 15:07

Holder:

Timestamp

Location: DocuSign

#### Signer Events

Security Level: Email, Account Authentication (Required)

Signature

Signature Adoption: Pre-selected Style

Signature ID:

778A4A1E-6353-4D54-A315-A8F10F2EF4FE

Using IP Address:

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

Electronic Record and Signature Disclosure:

Accepted: 15-Nov-2024 | 15:16 ID: 8670a8fb-1231-4053-8add-9fe48a86c804



Sent: 15-Nov-2024 | 15:11 Viewed: 15-Nov-2024 | 15:12 Signed: 15-Nov-2024 | 15:12

Caidya

Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style

Signature ID:

3F1277AD-321D-4048-BF56-4AE5BED08E47

Using IP Address:

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I am the author of this document
I am the author of this document

Electronic Record and Signature Disclosure:

Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |

| Certified Delivery Events | Status | Timestamp |
|---|---|---|
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Summary Events Envelope Sent | Status Hashed/Encrypted | <b>Timestamps</b><br>15-Nov-2024 15:11 |
| Envelope Sent | Hashed/Encrypted | 15-Nov-2024 15:11 |
| Envelope Sent<br>Certified Delivered | Hashed/Encrypted<br>Security Checked | 15-Nov-2024 15:11<br>15-Nov-2024 15:12 |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted Security Checked Security Checked | 15-Nov-2024 15:11<br>15-Nov-2024 15:12<br>15-Nov-2024 15:12 |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Caidya (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Caidya:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to:

#### To advise Caidya of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Caidya

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Caidya

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: https://support.docusign.com/guides/signer-guide-signing-system-requirements.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send
  this Electronic Record and Disclosure to a location where you can print it, for future
  reference and access; and
- Until or unless you notify Caidya as described above, you consent to receive exclusively
  through electronic means all notices, disclosures, authorizations, acknowledgements, and
  other documents that are required to be provided or made available to you by Caidya
  during the course of your relationship with Caidya.